# STATISTICAL ANALYSIS PLAN (SAP)

RANDOMIZED, PLACEBO-CONTROLLED,
DOUBLE-BLIND PHASE 2 STUDY OF
PATRITUMAB (U3-1287) IN COMBINATION WITH
CETUXIMAB PLUS PLATINUM-BASED THERAPY
IN FIRST LINE SETTING IN SUBJECTS WITH
RECURRENT OR METASTATIC SQUAMOUS
CELL CARCINOMA OF THE HEAD AND NECK

**PROTOCOL U31287-A-U203** 

**VERSION 1.0, 29 NOVEMBER 2016** 

Daiichi Sankyo, Inc. 399 Thornall Street Edison, NJ 08837 United States

#### **CONFIDENTIALITY STATEMENT**

Information contained in this document is proprietary to Daiichi Sankyo Development Limited. The information is provided to you in confidence to enable you to perform the work, which is requested under an agreed upon and signed confidentiality statement. Do not give this document or any copy of it or reveal any proprietary information contained in it to any third party (other than those in your organization who are assisting you in this work and are bound by the confidentiality statement) without the prior written permission of an authorized representative of Daiichi Sankyo Development Limited.

### SAP APPROVAL FORM

**Document Title:** 

Statistical Analysis Plan (SAP)

**Protocol Number:** 

U31287-A-U203

Study Title:

RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND

PHASE 2 STUDY OF PATRITUMAB (U3-1287) IN

COMBINATION WITH CETUXIMAB PLUS PLATINUM-BASED

THERAPY IN FIRST LINE SETTING IN SUBJECTS WITH RECURRENT OR METASTATIC SQUAMOUS CELL

CARCINOMA OF THE HEAD AND NECK

**Document Date:** 

**29 NOVEMBER 2016** 

**Document Version:** 

Version 1.0

| Prepared By: | |
|--------------|---------------------------------|
| Print Name | Signature |
| Title | 30 Nar 2016 Date (DD MMM YYYY) |
| 7,000 | Day (DD NATHELLE) |
| Print Name | Signature |
| | 29 NOV2016 |
| Title | Date (DD MMM YYYY) |
| Reviewed By: | 7 |
| Print Name | Signature |
| Title | Date (DD MMM YYYY) |
| Print Name | Signature |
| Title | Date (DD NOMA WENG) |
| A IAIG | Date (DD MMM YYYY) |

### SAP APPROVAL FORM

**Document Title:** Statistical Analysis Plan (SAP)

Protocol Number: U31287-A-U203

Study Title: RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND

PHASE 2 STUDY OF PATRITUMAB (U3-1287) IN

COMBINATION WITH CETUXIMAB PLUS PLATINUM-BASED

THERAPY IN FIRST LINE SETTING IN SUBJECTS WITH

RECURRENT OR METASTATIC SQUAMOUS CELL

CARCINOMA OF THE HEAD AND NECK

**Document Date:** 29 NOVEMBER 2016

**Document Version:** Version 1.0

| Prepared By: | |
|-----------------------------------------|---------------------------------|
| Print Name | Signature |
| Title | Date (DD MMM YYYY) |
| Print Name | Signature |
| Biostatistics, DSPD Title | Date (DD MMM YYYY) |
| Reviewed By: | |
| Print Name | Sygnature |
| Title | 12 Date (DD MMM YYYY) |
| *************************************** | Date (DD MAIN 1111) |
| Print Name | Signature |
| Title | 12 Dec 2016. Date (DD MMM YYYY) |

### SAP APPROVAL FORM

Document Title:

Statistical Analysis Plan (SAP)

Protocol Number:

U31287-A-U203

Study Title:

RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND

PHASE 2 STUDY OF PATRITUMAB (U3-1287) IN

COMBINATION WITH CETUXIMAB PLUS PLATINUM-BASED THERAPY IN FIRST LINE SETTING IN SUBJECTS WITH

RECURRENT OR METASTATIC SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK

Document Date:

29 NOVEMBER 2016

Document Version:

Version 1.0

| Print Name | | Signature |
|---------------------|----------------|--------------------|
| | | 12 DEC 2016 |
| Title | | Date (DD MMM YYYY) |
| CRO Approved By: | | |
| Print Name | | Signature |
| | | 02 pec 2016 |
| Title | | Date (DD MMM YXXX) |
| Sponsor Approval By | 7: | |
| | YY | |
| Print Name | | Signature |
| | _ | |
| Title | | Date (DD MMM YYYY) |
| | | 1 |
| DOCUMENT REVISI | ON HISTORY | |
| Document Version | Document Date | Revisions |
| Version 1.0 | 29NOV2016 | Original SAP |
| | - Arraiginania | |

Statistical Analysis Plan (SAP)

**Document Title:** 

Title

### SAP APPROVAL FORM

| Protocol Number: | U31287-A-U203 |
|---|---|
| Study Title: | RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND PHASE 2 STUDY OF PATRITUMAB (U3-1287) IN COMBINATION WITH CETUXIMAB PLUS PLATINUM-BASED THERAPY IN FIRST LINE SETTING IN SUBJECTS WITH RECURRENT OR METASTATIC SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK |
| <b>Document Date:</b> | 29 NOVEMBER 2016 |
| Document Version: | Version 1.0 |
| Print Name | Signature |
| Title | Date (DD MMM YYYY) |
| CRO Approved By: | |
| Print Name | Signature |

| Sponsor Appro | val By: | |
|---------------|---------|-------------|
| Print Name | | Signature |
| | | 13 Pec 2016 |

| | Revisions | | Document Date | <b>Document Version</b> |
|---|-----------|--------------|---------------|-------------------------|
| | | Original SAP | 29NOV2016 | Version 1.0 |
| - | | | | |

Date (DD MMM YYYY)

Date (DD MMM YYYY)

### STATISTICAL ANALYSIS PLAN SYNOPSIS

| Protocol Number: | U31287-A-U203 |
|---|---|
| Protocol Version and Date: | VERSION 4.0 13 JUN 2016 |
| Name of Investigational<br>Product: | Patritumab (U3-1287) |
| Study Title: | Randomized, Placebo-Controlled, Double-Blind Phase 2<br>Study of Patritumab (U3-1287) in Combination with<br>Cetuximab plus Platinum-Based Therapy in First Line<br>Setting in Subjects with Recurrent or Metastatic Squamous<br>Cell Carcinoma of the Head and Neck |
| Study Phase: | Phase 2 |
| Study Objectives: | <ul> <li>To evaluate progression-free survival (PFS) in the heregulin (HRG) high expression population from subjects treated with patritumab + cetuximab + platinum-based therapy compared to placebo + cetuximab + platinum-based therapy.</li> <li>Secondary Objectives</li> <li>Evaluate overall survival (OS)</li> <li>Evaluate overall response rate (ORR)</li> <li>Refine the cutoff between heregulin high and low expression based on clinical data from this study</li> <li>Assess the population PK of patritumab in subjects with Squamous cell carcinoma of the head and neck (SCCHN)</li> <li>Assess the PK parameters of serum cetuximab and platinum concentrations when cetuximab and cisplatin or carboplatin (platinum-based therapy) are coadministered with patritumab in a sub group (n = 30) of subjects</li> <li>Evaluate the incidence of human antihuman antibody (HAHA) formation (anti-patritumab antibodies)</li> <li>Evaluate the safety and tolerability of the combination of patritumab + cetuximab + platinum-based therapy in first-line treatment of subjects with</li> </ul> |

#### Study Design:

This is a multicenter, randomized, placebo-controlled, double blind Phase 2 study to evaluate the PFS and safety in recurrent/metastatic first-line SCCHN in subjects treated with patritumab plus cetuximab plus platinum-based therapy compared with subjects randomized to the control arm consisting of placebo plus cetuximab plus platinum-based therapy.

There will be two treatment arms stratified by HRG status (high and low):

- 1. Patritumab + cetuximab + platinum-based therapy with HRG high and HRG low subjects
- 2. Placebo + cetuximab + platinum-based therapy with HRG high and HRG low subjects

Approximately 105 subje ts will be randomized to the patritumab and the control arms in a 2:1 stratification fashion between HRG high versus low strata (approximately 70 HRG-high and approximately 35 HRG-low subjects). When one HRG stratum is filled with the required sample size, the enrollment in that HRG stratum will cease. The randomized subjects will also be further stratified 1:1 by HPV status (positive vs negative). The cut-off for HRG high versus low before randomization will be set using the median HRG value of commercial tissue samples.

Number of Planned Study Centers:

Approximately 35 sites in Europe.

#### Planned Sample Size:

The primary efficacy endpoint is PFS. The sample size for this study is based on the number of required PFS events in the HRG-high stratum. For PFS, a clinically meaningful improvement is defined as 79% increase from median PFS of 4.2 months in the control arm to median PFS of 7.5 months in the patritumab arm (that is a HR of 0.56). A total of 70 HRG-high subjects will be randomized to observe 53 PFS events in the HRG high stratum assuming a one-sided alpha of 0.10, 80% power, and a 1:1 randomization ratio between 2 arms, a 12-month enrollment and 10-month follow-up, and 10% dropouts.

Under 2:1 (HRG high vs. low) stratification, a total of approximately 105 subjects (70 HRG high subjects and 35 HRG low subjects) will be r ndomized in both strata to observe at least 75 PFS events. The sample size from both strata combined will provide approximately 81% power to detect a HR=0.56 in PFS assuming one-sided alpha of 0.05 and other same assumptions above.

The sample size computation is performed using the test based on Survival Superiority Trials: Two Sample Test – Logrank Test: Given Accrual Duration and Study Duration in the EAST software (version 5.3, Cytel Inc.).

### Study Duration:

For the purpose of collecting survival data, the duration of the study will be until all subjects have died or a minimum of 13 months after the last subject is randomized whichever comes first, approximately 22 months for PFS and 25 months for OS.

Subjects receiving clinical benefit from treatment will be offered the opportunity to continue therapy with patritumab and cetuximab (platinum-based therapy administered for no more than 6 cycles) in the extension phase of this protocol.

## Summary of Eligibility Criteria:

#### **Key Inclusion Criteria**

- 1. Adult subjects ≥18 years old
- 2. Histologically confirmed recurrent disease or metastatic SCCHN tumor and/or from its lymph nodal metastases originating from the oral cavity, oropharynx, hypopharynx, and larynx
- 3. Heregulin expression level is required
- Samples must be taken from subjects who have recurrent or metastatic disease. These samples can be from either rec/met archived or fresh biopsy samples
- No cancer treatment between time of biopsy and submission of sample
- Surgical or core needle biopsy is acceptable
- Fine-needle aspiration or cytology is not acceptable for biopsies
- 4. Human papilloma virus (HPV) status or p16 (surrogate for HPV) is required. These results must come from tumor tissue. These results may be obtained from either a local lab or samples sent to the central lab
- HPV or p16 status can be from any tumor biopsy material from initial diagnosis
- 5. Measurable disease per Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1
- 6. Eastern Cooperative Oncology Group performance status 0 or 1
- 7. Hematological function, as follows:
- Absolute neutrophil count ≥  $1.5 \times 10^9$ /L
- Platelet count  $\geq 100 \times 10^9 / L$
- Hemoglobin  $\ge 10 \text{ g/dL}$
- 8. Renal function, as follows:
- Estimated serum creatinine clearance (mL/min) or glomerular filtration rate (GFR) ≥ 60 mL/min for cisplatin and ≥ 30 mL/min for carboplatin

- 9. Hepatic function, as follows:
- Aspartate aminotransferase ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, < 5 x ULN)
- Alanine aminotransferase ≤ 2.5 x ULN (if liver metastases are present, < 5 x ULN)</li>
- Alkaline phosphatase  $\leq 2.0 \text{ x ULN}$  (if bone or liver metastases are present,  $\leq 5 \text{ x ULN}$ )
- Bilirubin < 1.5 x ULN
- 10. Prothrombin time or partial thromboplastin time  $\leq$  1.5 x ULN
- 11. Women of childbearing potential must have a negative serum pregnancy test performed within 14 days prior to enrollment (where demanded by local regulations, test may be required within 72 hours prior to enrollment)
- 12. Adult subjects of child-bearing potential must agree to use double barrier contraceptive measures. Two of the following precautions must be used: bilateral vasec omy, bilateral tubal ligation, intrauterine device (IUD), combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine hormonereleasing system (IUS), condom with spermicide, abstinence. These contraception measures must be used for the entire duration of the study and for 6 months after the last study dose is received
- 13. Subjects must be willing and able to comply with schedule visits, treatment plan, laboratory tests, and other study procedures
- 14. Provided written informed consent(s)

**Key Exclusion Criteria** 

- 1. Left ventricular ejection fraction <50%
- 2. Prior epidermal growth factor receptor targeted regimen
- 3. No HRG expression result
- 4. No HPV or p16 status

- 5. Prior anti-HER3 therapy
- 6. Prior chemotherapy for recurrent/metastatic disease
- 7. Anti-cancer therapy between biopsy and submission of sample
- 8. Presence of squamous cell tumors of the nasopharynx
- 9. History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 2 years
- 10. Known history of brain metastases or currently active brain metastases
- 11. Uncontrolled hyperten ion (systolic > 160 mm Hg or diastolic > 100 mm Hg)
- 12. Clinically significant electrocardiogram (ECG) changes
- 13. Myocardial infarction within 1 year before enrollment, symptomatic congestive heart failure (New York Heart Association >Class II), unstable angina, or unstable cardiac arrhythmia requiring medication
- 14. Platinum-containing drug therapy with radiotherapy less than 6 months before study drug treatment
- 15 Therapeutic or palliative radiation therapy or major surgery within 4 weeks before study drug treatment. Radiation treatment to all sites of measureable disease unless progression is documented after radiation
- 16. Participated in clinical drug trials within 4 weeks before study drug treatment. Current participation in other investigational procedures
- 17. Uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals, known HIV infection, or active hepatitis B or C infection or undergoing medical treatment for infection
- 18. Uncontrolled type 1 or 2 diabetes mellitus
- 19. Known hypersensitivity or allergic reaction against any of the components of the trial treatment
- 20. Pregnant, breastfeeding, or unwilling/unable to use acceptable contraception
- 21. Residual toxicities ≥ Grade 1 from previous therapies that the Investigator determines would exclude

### participation

- 22. Psychological, social, familial, or geographical factors that would interfere with study participation or follow-up
- 23. Committed to an institution by virtue of an order issued either by judicial or administrative authorities
- 24. Employee or immediate relative of an employee of the sponsor, CRO, the study center, or their affiliates or partners
- 25. Receiving yellow fever vaccine or live attenuated vaccines (for subjects receiving carboplatin)
- 26. Presence of hemorrhagic tumors (for subjects receiving carboplatin)
- 27. Prophylactic use of phenytoin or fosphenytoin (for subjects receiving cisplatin or carboplatin)

#### Primary Endpoint:

The primary efficacy endpoint is PFS, defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1 as assessed by investigator) or death due to any cause.

#### Secondary Endpoint:

- OS
  - Date of randomization to death due to any cause
  - Subjects alive at time of data cut off for OS analysis will be censored at the last contact date at which subject is known to be alive
- ORR (CR and PR)
  - Proportion of subjects with the best ORR of complete response (CR) or partial response (PR) regardless of whether it is confirmed or unconfirmed
- Pharmacokinetic parameters: AUC<sub>0-21d</sub> and C<sub>max</sub> at end of infusion (EOI) for serum patritumab, cetuximab, and platinum concentrations in a subgroup (approximately 30 subjects).
  - Population PK methods will be used to assess the sparse data for serum patritumab concentrations

#### Safety

- Treatment-emergent Adverse events
- ≥ Grade 3 National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
- Clinical lab evaluations
- Myocardial function status (assessed by echocardiograms or multigated acquisition scan)
- ECGs
- Vital signs
- Physical exams
- Human anti-humanized antibody formation

### Stopping Criteria:

#### NA

#### Statistical Considerations:

This is a multicenter randomized Phase 2 study designed to evaluate the safety and efficacy of patritumab in combination with cetuximab and platinum-based therapy in recurrent/metastatic first-line SCCHN. The primary analyses for this study will occur when at least 53 PFS events have been observed in the HRG high stratum.

At the point of primary analysis for PFS, the treatment assignment for all randomized subjects will be unblinded to designated study personnel for the analysis after data are reconciled and cleaned and a snapshot of the clean database is created. To minimize potential bias, subjects and Investigators will not be informed about individual treatment assignment until study closure.

Final analyses will occur after study closure with mature OS data for the main study phase. At the time of study closure, subjects who are demonstrating clinical benefit [stable disease (SD) or better] from study treatment may be offered an opportunity to continue study treatment on the extension phase.

Assessments of change from baseline to post baseline or the ratio of post baseline to baseline will include only those subjects with both baseline and post baseline measurements. The last nonmissing value of a variable taken before the first dose of study drug will be used as the baseline value, unless otherwise specified. In general,

missing or dropout data will not be imputed for the purpose of data analysis. Descriptive summary statistics (n, mean, median, standard deviation, and range) will be calculated for continuous variables, and for categorical variables, the number and percentage in each category will be displayed by treatment group.

# Statistical Analysis for the Primary Endpoint:

The primary analysis is PFS comparison between the patritumab arm and the control arm in HRG-high stratum of the FAS. The testing hypotheses to compare PFS between the patritumab arm versus the control arm will be performed in two steps. In step 1, the null hypothesis that PFS is the same for both arms in the HRG high stratum of FAS is tested at the one sided 0.10 significance level. If this test in step 1 does not reject the null hypothesis, then in step 2A, the null hypothesis that PFS is the same for both arms in the FAS will be tested at the one-sided 0.05 significance level. If the test in step 1 is rejected, then in step 2B, the two-sided 80% confidence interval (CI) for hazard ratio (HR) of PFS in the HRG low stratum of the FAS will be estimated.

The comparison of PFS between the patritumab arm and the control rm will be performed using a log-rank test stratified by the stratification factors in both the FAS and the HRG high stratum of FAS. The stratification factors include HPV (positive vs other) and HRG (high vs. low, only for the FAS) at randomization. Kaplan-Meier methods will be used to calculate median PFS and CIs and generate Kaplan-Meier curves for PFS. Estimates of HR between 2 arms along with their two-sided 80% and 95% CIs will be calculated using stratified Cox's proportional hazards regression model. The model will include the treatment group as a covariate and the stratification factors used at randomization as strata.

The above analysis for PFS will also be performed in the per-protocol analysis set.

Statistical Analysis for the Secondary Endpoints:

Secondary efficacy variables include OS and ORR (CR and PR). Overall survival is defined from the date of randomization to death due to any cause and will be analyzed in the same manner as PFS. Subjects who are alive at the time of data cut off for overall survival analysis will be censored at the last contact date at which the subject is known to be alive. ORR is defined as the proportion of subjects with the best overall response of CR or PR regardless of whether it is confirmed or unconfirmed. The differences in the ORR between the control arm and patritumab arm will be presented along with two-sided 80% and 95% CIs based on the Wilson's score method with continuity correction. These analyses will be done using the FAS for HRG high and low strata.

Safety data will be analyzed descriptively.

Serum concentrations for patritumab, cetuximab, and cisplatin/carboplatin will be displayed in tables of individual values and aggregated by treatment group in summary tables with descriptive statistics. To explore possible drug-drug interactions between patritumab plus cetuximab or cisplatin/carboplatin, the PK of serum cetuximab and platinum concentrations will be compared with and without patritumab. For all subjects, sparse samples for serum patritumab concentrations will be assessed using population PK methods. The relationship between exposure and response will be explored using population PK modeling.

### **GENERAL INFORMATION**

| Name and Address of Sponsor: | Daiichi Sankyo, Inc.<br>399 Thornall Street<br>Edison, NJ 08837<br>United States |
|---|---|
| Name and Address of the SAP Author: | Princeton, NJ 08540 |
| Name and Address of the Sponsor Study Biostatistician: | PhD Daiichi Sankyo, Inc. 399 Thornall Street Edison NJ 08837 |

### TABLE OF CONTENTS

| STATIS | TICAL ANALYSIS PLAN SYNOPSIS | 4 |
|----------|------------------------------------------|----|
| GENER. | AL INFORMATION | 14 |
| TABLE | OF CONTENTS | 15 |
| LIST OF | F TABLES | 19 |
| LIST OF | F FIGURES | 22 |
| LIST OF | F DATA LISTINGS | 23 |
| LIST OF | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 25 |
| 1. | SCOPE | 27 |
| 2. | STUDY OBJECTIVES | 28 |
| 2.1. | Primary Objectives | 28 |
| 2.2. | Secondary Objectives | 28 |
| 2.3. | Exploratory Objectives | 28 |
| 3. | STUDY DESIGN | |
| 3.1. | General Study Design and Plan | 30 |
| 3.2. | Study Population | 37 |
| 3.3. | Randomization and Blinding | |
| 3.3.1. | Randomization | 37 |
| 3.3.2. | Blinding | 37 |
| 3.3.2.1. | Unblinding at Primary Analysis | 37 |
| 3.3.2.2. | Unblinding at Study Closure | 38 |
| 3.3.2.3. | Emergency Unblinding | 38 |
| 3.4. | Study Assessments | 38 |
| 4. | SAMPLE SIZE DETERMINATION | 39 |
| 5. | STUDY VARIABLES | 40 |
| 5.1. | Efficacy Variables | 40 |
| 5.1.1. | Primary Efficacy Variable | 40 |
| 5.1.2. | Secondary Efficacy Variables | 41 |
| 5.1.2.1. | Overall Survival (OS) | 41 |
| 5.1.2.2. | Object Response Rate (ORR) | 42 |
| 5.1.3. | Exploratory Efficacy Variables | 42 |

| 5.1.3.1. | Duration of Response | 42 |
|----------|-------------------------------------------------------|----|
| 5.1.3.2. | Time to Response | 43 |
| 5.1.3.3. | Time to Disease Progression (TTP) | 43 |
| 5.1.3.4. | Duration of Stable Disease (SD) | 43 |
| 5.2. | Safety Variables | 43 |
| 5.2.1. | Adverse Events | 43 |
| 5.2.2. | Clinical Laboratory Evaluations | 44 |
| 5.2.3. | Vital Signs | 44 |
| 5.2.4. | ECG | 44 |
| 5.2.5. | Physical Examinations | |
| 5.2.6. | Other Safety Variables | 44 |
| 5.3. | Pharmacokinetic Variables | 45 |
| 5.3.1. | Concentration Data | 45 |
| 5.3.2. | Pharmacokinetic (PK) Parameters. | |
| 5.4. | Pharmacodynamic (PD) Variables | |
| 5.5. | Biomarkers | 45 |
| 5.6. | Other Variables | 46 |
| 5.6.1. | Eastern Cooperative Oncology Group Performance Status | 46 |
| 5.6.2. | Patient Reported Outcomes . | 46 |
| 6. | ANALYSIS SETS | 49 |
| 6.1. | Analysis Sets Definitions | 49 |
| 6.1.1. | Full Analysis Set | 49 |
| 6.1.2. | Safety Analysis Set | 49 |
| 6.1.3. | Per-Protocol Analysis Set | 49 |
| 6.1.4. | Pharmacokinetic Analysis Set | 49 |
| 6.1.5. | Patient Reported Outcome Analysis Set | 49 |
| 6.2. | Protocol Deviations | 49 |
| 6.3. | Treatment Misallocations | 49 |
| 7. | GENERAL STATISTICAL CONSIDERATIONS | 51 |
| 7.1. | Adjustment for Covariates | 51 |
| 7.2. | Handling of Dropouts or Missing Data | 51 |
| 7.3. | Interim Analyses and Data Monitoring | 51 |

| 7.4. | Multicenter Studies | 52 |
|----------|--------------------------------------------|----|
| 7.5. | Multiple Comparisons/Multiplicity | 52 |
| 7.6. | Examination of Subgroups | 52 |
| 8. | STATISTICAL ANALYSIS | 53 |
| 8.1. | Study Population Data | 53 |
| 8.1.1. | Subject Disposition | 53 |
| 8.1.2. | Protocol Deviations | 53 |
| 8.1.3. | Demographic and Baseline Characteristics | 53 |
| 8.2. | Efficacy Analyses | 54 |
| 8.2.1. | Analysis of Primary Efficacy Variables | 54 |
| 8.2.2. | Analysis of Secondary Efficacy Variables | 55 |
| 8.2.2.1. | Overall Survival | 55 |
| 8.2.2.2. | Overall Survival Objective Response Rate | 55 |
| 8.2.2.3. | Cutoff for HRG Expression | |
| 8.2.3. | Analysis of Exploratory Efficacy Variables | 56 |
| 8.2.3.1. | Duration of Response | 56 |
| 8.2.3.2. | Time to Response | 56 |
| 8.2.3.3. | Time to Disease Progression | 56 |
| 8.2.3.4. | Duration of Stable Disease | 56 |
| 8.2.4. | Sensitivity and Subgroup Analysis | 56 |
| 8.2.4.1. | Sensitivity Analysis | 56 |
| 8.2.4.2. | Subgroup Analysis | 57 |
| 8.3. | Safety Analyses | 58 |
| 8.3.1. | Adverse Events | |
| 8.3.2. | Clinical Laboratory Evaluations | 59 |
| 8.3.4. | Vital Signs | 60 |
| 8.3.5. | ECG | 60 |
| 8.3.6. | Dosing and Extent of Exposure | 61 |
| 8.3.7. | Prior and Concomitant Medications | 62 |
| 8.3.9. | Analysis of Other Safety Variables | 62 |
| 8.4. | Pharmacokinetic Analyses | |
| 8.4.1. | Concentration Data | 63 |

| 8.4.1.1. | Sparse Patritumab PK | 63 |
|----------|-----------------------------------------------------------|----|
| 8.4.1.2. | Intensive PK | 63 |
| 8.4.2. | Analysis of Pharmacokinetic (PK) Parameters | 63 |
| 8.4.3. | Population Pharmacokinetic (PK) and Exposure Response | 64 |
| 8.5. | Pharmacodynamic (PD) Parameters | 64 |
| 8.6. | Biomarkers Analyses | 64 |
| 8.7. | Other Variables Analyses | 64 |
| 8.7.1. | Patient Reported Outcomes | 64 |
| 9. | CHANGES FROM THE PROTCOL SPECIFIED STATISTICAL ANALYSES | 66 |
| 10. | REFERENCES | 67 |
| 11. | APPENDICES | 68 |
| 11.1. | Data Derivation Details | 68 |
| 11.1.1. | Windows Convention for Handling Partial and Missing Dates | 68 |
| 11.2. | Interim Analysis Statistical Analysis Plan | 70 |
| 11.3. | Formula for Wilson Method | 71 |
| 11 4 | Mock-up Tables and Listings | 72 |

### LIST OF TABLES

| Table 15.1.1 | Subject Disposition (All Screened Subjects) |
|---|---|
| Table 15.1.2.1 | Demographic and Baseline Characteristics (Full Analysis Set) |
| Table 15.1.2.2 | Demographic and Baseline Characteristics (Per-Protocol Analysis Set) |
| Table 15.1.2.3 | Demographic and Baseline Characteristics (Safety Analysis Set) |
| Table 15.1.3 | Study Drug Exposure (Safety Analysis Set) |
| Table 15.1.4.1 | Prior Medications by ATC Class and Preferred Term (Safety Analysis Set) |
| Table 15.1.4.2 | Concomitant Medications by ATC Class and Preferred Term (Safety Analysis Set) |
| Table 15.2.1.1 | Analysis of Progression Free Survival (PFS) (Full Analysis Set) |
| Table 15.2.1.2 | Analysis of Progression Free Survival (PFS) (Per Protocol Analysis Set) |
| Table 15.2.1.3 | Subgroup Analysis of Progression Free Survival (PFS) (Full Analysis Set) |
| Table 15.2.1.4 | Analysis of Progression Free Survival (PFS) for Different HRG Cutoffs (Full Analysis Set) |
| Table 15.2.2.1 | Analysis of Overall Survival (OS) (Full Analysis Set) |
| Table 15.2.2.2 | Analysis of Overall Survival (OS) (Per Protocol Analysis Set) |
| Table 15.2.2.3 | Subgroup Analysis of Overall Survival (OS) (Full Analysis Set) |
| Table 15.2.2.4 | Analysis of Overall Survival (OS) for Different HRG Cutoffs (Full Analysis |
| | Set) |
| Table 15.2.3.1 | Best Overall Tumor Response and Objective Response Rate (ORR) (Full |
| 14010 10.2.3.1 | Analysis Set) |
| Table 15.2.3.2 | Best Overall Tumor Response and Objective Response Rate (ORR) (Per |
| 1 4010 13.2.3.2 | Protocol Analysis Set) |
| T-1-1- 15 2 4 | |
| Table 15.2.4 | Duration of Objective Response/Stable Disease and Time to Response/Disease Progression (Full Analysis Set) |
| Table 15.2.5 | Summary of Chang and the Percent Change from Baseline in the Sum of |
| 1able 13.2.3 | Longest Diameters of Target Lesions (Full Analysis Set) |
| Table 15.3.1.1 | Overview of Number (%) of Subjects Reporting Treatment-Emergent |
| 14010 13.3.1.1 | Adverse Events (Safety Analysis Set) |
| Table 15.3.1.2 | Number and Percentage of Subjects with Treatment-emergent Adverse |
| | Events Summarized by Worst CTCAE Grade, System Organ Class, and |
| | Preferred Term (Safety Analysis Set) |
| Table 15.3.1.3 | Number and Percentage of Subjects with Treatment-emergent Serious |
| | Adverse Events Summarized by Worst CTCAE Grade, System Organ Class, |
| | and Preferred Term (Safety Analysis Set) |
| Table 15.3.1.4 | Number and Percentage of Subjects with Treatment-emergent Adverse |
| | Events Related to Patritumab/Placebo Summarized by Worst CTCAE Grade, |
| T. 11. 15.2.1.5 | System Organ Class, and Preferred Term (Safety Analysis Set) |
| Table 15.3.1.5 | Number and Percentage of Subjects with Treatment-emergent Adverse |
| | Events Related to Cetuximab Summarized by Worst CTCAE Grade, System |
| Table 15.3.1.6 | Organ Class, and Preferred Term (Safety Analysis Set) Number and Percentage of Subjects with Treatment-emergent Adverse |
| 14016 13.3.1.0 | Events Related to Cisplatin/Carboplatin Summarized by Worst CTCAE |
| | Grade, System Organ Class, and Preferred Term (Safety Analysis Set) |
| Table 15.3.1.7 | Number and Percentage of Subjects with Treatment-emergent Serious |
| - 3010 10.0.1.7 | |

| | Adverse Events Related to Patritumab/Placebo Summarized by Worst |
|---|---|
| | CTCAE Grade, System Organ Class, and Preferred Term (Safety Analysis |
| | et) |
| | Number and Percentage of Subjects with Treatment-emergent Serious |
| A | Adverse Events Related to Cetuximab Summarized by Worst CTCAE Grade, |
| | ystem Organ Class, and Preferred Term (Safety Analysis Set) |
| Table 15.3.1.9 N | Number and Percentage of Subjects with Treatment-emergent Serious |
| A | Adverse Events Related to Cisplatin/Carboplatin Summarized by Worst |
| C | CTCAE Grade, System Organ Class, and Preferred Term (Safety Analysis |
| S | et) |
| Table 15.3.1.10 N | Number and Percentage of Subjects with Potential Hy's Law Event by Worst |
| C | CTCAE Grade, System Organ Class, and Preferred Term (Safety Analysis |
| | let) |
| Table 15.3.4.1 S | ummary of Results and Change from Baseline in Laboratory Tests – |
| | Iematology (Safety Analysis Set) |
| | ummary of Results and Change from Baseline in Laboratory Tests – |
| | Chemistry (Safety Analysis Set) |
| | hift Table of CTCAE Grade in Labor tory Tests – Hematology (Safety |
| | analysis Set) |
| | hift Table of CTCAE Grade in Labora ory Tests – Chemistry (Safety |
| | analysis Set) |
| | Number and Percentage of Subjects with Liver Enzymes (ALT, AST) and |
| | Total Bilirubin (TBL) Elevation (Safety Analysis Set) |
| | cummary of Vital Signs and Change from Baseline (Safety Analysis Set) |
| | ummary of 12-Lead ECG and Change from Baseline (Safety Analysis Set) |
| | ummary of Subjects M eting Pre-Specified QT and QTcB/QTcF Criteria Safety Analysis Se) |
| | hift Table of ECOG S tus (Safety Analysis Set) |
| | ummary of L ft Ventricular Ejection Fraction (LVEF) Value and Change |
| fi | rom Baseline (Safety Analysis Set) |
| Table 15.4.1.1 S | ummary of Patritumab Concentration (ug/mL) from Sparse PK Sampling |
| (1 | Pharmacokinetics Analysis Set) |
| Table 15.4.1.2 S | ummary of Patritumab Concentration (ug/mL) from Intensive PK Sampling |
| | t Cycle 1 (Pharmacokinetic Analysis Set) |
| | ummary of Cetuximab Concentration (ug/mL) from Intensive PK Sampling |
| | t Cycle 1 (Pharmacokinetic Analysis Set) |
| | lummary of Cisplatin Concentration (ug/mL) from Intensive PK Sampling at Cycle 1 (Pharmacokinetic Analysis Set) |
| | , |
| | ummary of Carboplatin Concentration (ug/mL) from Intensive PK |
| S | ampling at Cycle 1 (Pharmacokinetic Analysis Set) |
| Table 15.4.2.1 S | ummary of Patritumab PK Parameters at Cycle 1 (Pharmacokinetic |
| | analysis Set) |
| | ummary of Cetuximab PK Parameters at Cycle 1 (Pharmacokinetic |
| | analysis Set) |
| | nummary of Cisplatin PK Parameters at Cycle 1 (Pharmacokinetic Analysis |
| | et) |
| | , |
| | lummary of Carboplatin PK Parameters at Cycle 1 (Pharmacokinetic Analysis Set) |

| Table 15.4.2.5 | Statistical Analysis of PK Parameters for Cetuximab, Cisplatin, and Carboplatin at Cycle 1 (Pharmacokinetic Analysis Set) |
|---|---|
| Table 15.5.1.1 | Summary of Actual Results and Change from Baseline in FACT-H&N Total Score, FACT-H&N Subscale (HNS) Score, HNS Individual Symptom Score, and FACT-H&N Symptom Index (FHNSI) Score (FACT-H&N Analysis Set) |
| Table 15.5.1.2 | Statistical Analysis of the Change from Baseline in the FACT-H&N total score, the FACT-H&N HNS, HNS individual symptom score, and the FACT-H&N FHNSI score (FACT-H&N Analysis Set) |
| Table 15.5.1.3 | Summary of Actual Results and Change from Baseline in EQ-5D Index (EQ-5D Analysis Set) |
| Table 15.5.1.4 | Summary of Actual Results and Change from Baseline in VAS Score (EQ-5D Analysis Set) |



### LIST OF FIGURES

| Figure 15.1.1 | CONSORT diagram |
|---|---|
| Figure 15.2.1.1 | Kaplan-Meier Plot of Progression Free Survival (PFS) by Treatment<br>Group (Full Analysis Set) |
| Figure 15.2.1.2 | Forest Plot of Progression Free Survival (PFS) for Selected Subgroups (Full Analysis Set) |
| Figure 15.2.1.3 | Kaplan-Meier Plot of Progression Free Survival (PFS) for Different HRG Cutoffs by Treatment Group (Full Analysis Set) |
| Figure 15.2.1.4 | Forest Plot of Progression Free Survival (PFS) for Different HRG<br>Cutoffs (Full Analysis Set) |
| Figure 15.2.2.1 | Kaplan-Meier Plot of Overall Survival (OS) by Treatment Group (Full Analysis Set) |
| Figure 15.2.2.2 | Forest Plot of Overall Survival (OS) for Selected Subgroups (Full Analysis Set) |
| Figure 15.2.2.3 | Kaplan-Meier Plot of Overall Survival (OS) for Different HRG<br>Cutoffs by Treatment Group (Full Analysis Se) |
| Figure 15.2.2.4 | Forest Plot of Overall Survival (OS) for Different HRG Cutoffs (Full Analysis Set) |
| Figure 15.2.3.1 | Waterfall Plot of Best (Minimum) Per nt Change in Sum of Longest Diameters from Baseline in T rget Lesions (Full Analysis Set) |
| Figure 15.2.4 | Swimmer Plot of Duration of Response (Full Analysis Set) |
| Figure 15.4.1.1 | Mean Plasma Concentration of Patritumab by Time from Sparse PK Sampling (Pharmacokinetic Analysis Sets) |
| Figure 15.4.1.2 | Mean Plasma Concentration of Patritumab by Time from Intensive PK Sampling (Pharmacokinetic Analysis Sets) |
| Figure 15.4.1.3 | Mean Plasma Con entration of Cetuximab by Time from Intensive PK Sampling (Pharmacok netic Analysis Sets) |
| Figure 15.4.1.4 | Mean Plasm Concentration of Cisplatin by Time from Intensive PK Sampling (Pharmacokinetic Analysis Sets) |
| Figure 15.4.1.5 | Mean Plasm Concentration of Carboplatin by Time from Intensive PK Sampling (Pharmacokinetic Analysis Sets) |
| Figure 15.4.2.1 | Boxplot of Patritumab PK Parameters at Cycle 1 (Pharmacokinetic Analysis Sets) |
| Figure 15.4.2.2 | Boxplot of Cetuximab PK Parameters at Cycle 1 by Treatment (Pharmacokinetic Analysis Sets) |
| Figure 15.4.2.3 | Boxplot of Cisplatin PK Parameters at Cycle 1 by Treatment (Pharmacokinetic Analysis Sets) |
| Figure 15.4.2.4 | Boxplot of Carboplatin PK Parameters at Cycle 1 by Treatment (Pharmacokinetic Analysis Sets) |
| Figure 15.5.1.1 | Plot of Cumulative Distribution Function of Change from Baseline on FACT-H&N HNS Score (FACT-H&N Analysis Set) |
| Figure 15.6.1 | Heregulin (HRG) Distritubution, Full Analysis Set |

### LIST OF DATA LISTINGS

| Listing 16.2.1.1 | Subject Disposition |
|---|---|
| Listing 16.2.1.1 | Deaths |
| Listing 16.2.2.1 | Inclusion/Exclusion Criteria |
| Listing 16.2.2.2 | Informed Consent |
| | Protocol Deviation |
| Listing 16.2.2.3 | |
| Listing 16.2.3 | Subject Inclusion in Analysis Sets |
| Listing 16.2.4.1 | Demographic Data |
| Listing 16.2.4.2 | Pregnancy Test Results |
| Listing 16.2.4.3 | Medical/Surgical History |
| Listing 16.2.4.4.1 | Cancer History for SCCHN |
| Listing 16.2.4.4.2 | Prior Head and Neck Systemic Cancer Therapy |
| Listing 16.2.4.4.3 | Prior Radiation Therapy |
| Listing 16.2.4.5 | Prior/Concomitant Medication |
| Listing 16.2.4.6 | Non-Drug Treatment/Procedures |
| Listing 16.2.5.1.1 | Investigational Drug Patritumab Adminis ration |
| Listing 16.2.5.1.2 | Cetuximab, Cisplatin, and Carboplatin Administration |
| Listing 16.2.5.1.3 | Patritumab, Cetuximab, and Cisplatin/Carboplatin Exposure |
| Listing 16.2.5.2.1 | Patritumab Pharmacokinetic Sample Collection Time and Results |
| Listing 16.2.5.2.2 | Cetuximab Pharmacokinetic Sample Collection Time and Results |
| Listing 16.2.5.2.3 | Patritumab Pharmacokinetic Sample Collection Time and Results |
| Listing 16.2.5.2.4 | Cetuximab Pharmacokinetic Sample Collection Time and Results |
| Listing 16.2.6.1.1 | Target Tumor Assessment |
| Listing 16.2.6.1.2 | Non-Target Tumor Assessment |
| Listing 16.2.6.1.3 | Overall Tumor Ass ssment |
| Listing 16.2.6.2 | Progression-Fre Survival and Overall Survival |
| Listing 16.2.6.3 | Subjects with Complete Response (CR), Partial Response (PR), or Stable Dis ase (SD) |
| Listing 16.2.7.1 | Adv se Event |
| Listing 16.2.7.2 | Serious Adverse Events, Including those Leading to Deaths |
| Listing 16.2.7.3 | Adverse Events Leading to Study Drug Discontinuation |
| Listing 16.2.7.4 | Adverse Event Leading to Study Drug Interruption or Dose Reduction |
| Listing 16.2.7.5 | Adverse Events of Interest |
| Listing 16.2.8.1.1 | Laboratory Data – Hematology |
| Listing 16.2.8.1.2 | Laboratory Data – Chemistry |
| Listing 16.2.8.1.3 | Laboratory Data – Urinalysis |
| Listing 16.2.8.1.4 | Laboratory Data – Coagulation |
| Listing 16.2.8.2.1 | Clinically Significant Laboratory Abnormalities or Abnormalities of |
| | CTCAE Grade 3/4 Hematology |
| Listing 16.2.8.2.2 | Clinically Significant Laboratory Abnormalities or Abnormalities of |
| | CTCAE Grade 3/4 Chemistry |
| Listing 16.2.8.2.3 | Subjects with Liver Enzymes (ALT, AST) and Total Bilirubin (TBL) |
| | Elevation (Safety Analysis Set) |
| Listing 16.2.8.3.1 | Vital Signs |
| Listing 16.2.8.3.2 | 12 Lead ECG |
| Listing 16.2.8.3.3 | Physical Examination |
| Listing 16.2.8.3.4 | Eastern Cooperative Oncology Group (ECOG) Score |
| | 1 Troperante checked croap (1000) secte |

| Listing 16.2.8.3.5 | Echocardiogram |
|--------------------|-----------------------------------------------|
| Listing 16.2.8.4.1 | Human Anti-Humanized Antibody (HAHA) |
| Listing 16.2.8.4.2 | Tumor Tissue Collection and Biomarker Results |
| Listing 16.2.9.1.1 | FACT-H&N Item Scores |
| Listing 16.2.9.1.2 | FACT-H&N Total and Subscale Scores |
| Listing 16.2.9.2 | EQ-5D Scale Scores |



### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| ABBREVIATION | DEFINITION |
|---|---|
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUC | Area under curve |
| AUC <sub>0-21d</sub> | Area under curve at last time point |
| C <sub>max</sub> | Maximum observed circulating concentration |
| CR | Complete response |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ECG | Electrocardiograph |
| ECOG | Eastern Cooperative Oncology Group |
| EOI | End of infusion |
| EQ-5D-5L | EuroQoL-5 Dimensions-5 Levels |
| EWB | Emotional well-being |
| FACT-H&N | Functional Assessment of Cancer Therapy-Head and Neck |
| FHNSI | FACT-Head and Neck Symptom Index |
| FWB | Functional well-being |
| GFR | Glomerular filtration rate |
| НАНА | Human antihuman antibody |
| HNS | FACT-Head and Neck Subscale |
| HPV | Human p pilloma virus |
| HRG | Heregulin (product neuregulin-1 gene [nRG1]) |
| ILD | Interstitial Lung Disease |
| IV | Intraven us |
| IXRS | Interactive Web/Voice Response System |
| LD | longest diameters |
| LVEF | Left ventricular ejection fraction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MUGA | Multigated acquisition (scan) |
| NCI | National Cancer Institute |
| ORR | Objective response rate |
| OS | Overall survival |
| PFS | Progression-free survival |
| PK | Pharmacokinetic or pharmacokinetics |
| PR | Partial response |
| PROs | Patient reported outcomes |
| PWB | Physical well-being |
| QTc (QTcB; QTcF) | Heart rate-corrected QT interval (by Bazett's; by Fridericia's) |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious adverse event |

| ABBREVIATION | DEFINITION |
|--------------|----------------------------------------------|
| SAP | Statistical analysis plan |
| SCCHN | Squamous cell carcinoma of the head and neck |
| SD | Stable disease |
| SWB | Social well-being |
| TEAE | Treatment-emergent adverse event |
| ULN | Upper limit of normal |
| WBC | White Blood Count |



### 1. SCOPE

This Statistical Analysis Plan (SAP) is created based on Protocol U31287-A-U203 version 4.0, 13 JUN 2016. This version describes in detail the statistical methodology and the statistical analyses to be conducted for the above mentioned protocol. The analysis plan may change due to unforeseen circumstances. Any deviations to the planned statistical analyses specified within the SAP will be justified in writing and presented within the clinical study report.



### 2. STUDY OBJECTIVES

### 2.1. Primary Objectives

• To evaluate PFS in the HRG high expression population from subjects treated with patritumab + cetuximab + platinum-based therapy compared to placebo + cetuximab + platinum-based therapy

### 2.2. Secondary Objectives

- Evaluate OS
- Evaluate objective response rate (ORR)
- Refine the cutoff between HRG high and low xpression based on clinical data from this study
- Assess the population PK of patritumab in subjects with SCCHN
- Assess the PK parameters of serum cetuximab and platinum concentrations when cetuximab and cisplatin or carboplatin (platinum-based therapy) are coadministered with patritumab in subgroup (n = 30) of subjects
- Evaluate the incidence of HAHA formation (anti-patritumab antibodies)
- Evaluate the safety and tolerability of the combination of patritumab + cetuximab + platinum-based herapy in first-line treatment of subjects with SCCHN

### 2.3. Exploratory Objectives

- Duration of response, time to response, time to disease progression, duration of SD from subjects treated with patritumab + cetuximab + platinum-based therapy compared to those treated on placebo + cetuximab + platinum-based therapy
- Explore potential exposure-response and possibly other biomarker relationships
- Evaluate disease specific patient reported outcomes (PROs) using the Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N) which assesses:
  - Physical well-being
  - Functional well-being
  - Social/Family well-being
  - Emotional well-being
  - Head and neck cancer symptoms

- Evaluate head and neck cancer symptoms using the FACT-Head and Neck Symptom Index (FHNSI), a 10-item instrument comprising items from the FACT-H&N
- Evaluate PROs using the EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire, which assesses five dimensions:
  - Mobility
  - Self-care
  - Usual activities
  - Pain/discomfort
  - Anxiety/depression

### 3. STUDY DESIGN

#### 3.1. General Study Design and Plan

This is a multicenter, randomized, placebo-controlled, double blind Phase 2 study to evaluate the PFS and safety in recurrent/metastatic first-line SCCHN in subjects treated with patritumab plus cetuximab plus platinum-based therapy compared with subjects randomized to the control arm consisting of placebo plus cetuximab plus platinum-based therapy.

Adult subjects with metastatic SCCHN originating from the oral cavity, oropharynx, hypopharynx, and larynx with documented disease recurrence following previous treatment for non-metastatic disease will be studied.

Approximately 105 subjects will be randomized 1:1 to the patritumab and the control arms stratified by HRG value (high versus low) and HPV status (positive vs negative). Approximately 70 HRG-high and approximately 35 HRG-low subjects will be randomized. When one HRG stratum is filled with the required sample size, the enrollment in that HRG stratum will cease. The initial cut-off for HRG high versus low before randomization was set using the median HRG delta Ct value (0.93) of commercial tissue samples and was increased based on further samples to 1.50 on 29JUL2016. See Figure 3.1.1 for a schematic of the study d sign

Figure 3.1.1: Phase 2 Study Design



The enrolled subjects will be stratified by HRG (high, low) and HPV (positive, negative)

There will be two treatment arms:

- 1. Patritumab + cetuximab + platinum-based therapy with HRG high and HRG low subjects
- 2. Placebo + cetuximab + platinum-based therapy with HRG high and HRG low subjects

Figure 3.1.2 illustrates the order and timing of the treatments involved.



Figure 3.1.2: Order and Timing of Treatments

Patritumab initial loading dose is 18 mg/kg IV (or placebo) over 60 minutes followed in cycle 2 and beyond with a maintenance dose of 9 mg/kg IV over 60 minutes ( $\pm$  10 minutes) every three weeks. Infusion time can be extended to a maximum of 120 minutes for subjects unable to tolerate the 60 minute infusion. Cetuximab initial dose at 400 mg/m² IV is given as a 2-hour infusion followed by 250 mg/m² over 60 minutes weekly.

One hour after the end of the cetuximab administration (on the weeks when cetuximab and platinum therapy are coadministered) infuse with either:

- Cisplatin at 100 mg/m² IV infused over 1 hour, every three weeks up to a maximum of 6 cycles Pretreatment hydration with 2 liters of fluid prior to a cisplatin infusion is recommended and should adhere to institutional standards. Adequate hydration and urinary output must be maintained during the following 24 hours. Other pretreatments such as anti-emetic prophylaxis and posttreatments such as hydration are up to the discretion of the Investigator. This can be given in a separate infusion during patritumab and cetuximab infusion; or
- Carboplatin, IV bolus over 30-60 minutes, every 3 weeks for a maximum of 6 cycles. AUC 5 is the target. The carboplatin dose will be calculated using the Calvert formula: Carboplatin Dose (mg) = 5 x (glomerular filtration rate [GFR] + 25). Estimated serum creatinine clearance (mL/min) calculated using the modified Cockcroft-Gault equation also be used as an estimate for GFR. The carboplatin dose is required to be re-calculated for every dosing based on the current GFR (or creatinine clearance as an estimate of GFR as per the protocol).

Pre- and post-treatments are up to the discretion of the investigator.

For the purpose of collecting survival data, the duration of the study will be until all subjects have died or a minimum of 13 months after the last subject is randomized whichever comes first, approximately 22 months for PFS and 25 months for OS.

The screening period is up to 14 days. Each cycle of treatment will be 21 days. There is no limit to how many cycles for patritumab and cetuximab treatment. Treatment will continue without interruption in subjects with CR, partial response PR, or SD. However, platinum treatment (cisplatin or carboplatin) will be given up to a maximum of 6 cycles. Subject participation is expected to be approximately 20 months.

Subjects who demonstrate benefit from therapy may continue in the extension phase (Section 6.5) to receive treatment until progressive disease (PD), toxicity, withdrawal of consent, or starting another treatment for cancer therapy.

The study evaluation schedule is provided in Table 3.1.1 and Table 3.1.2

Table 3.1.1: Schedule of Events

| | Tissue<br>screen | Screen | Random- | Cycle 1 (Weeks 1-3) | | | | | | | | Cycle 4 & all Subsequent Cycles | End of<br>Cycle 6<br>& Every<br>4 Cycles | Every<br>6<br>weeks | End-of-<br>Study<br>Treatment<br>Visit | 40 Days<br>After<br>Last<br>Dose <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5010011 | | ILWU VI | | Day 1 | | Day 2 | D. 2 | ъ о | Day 15 | Day 1 | B 1 | | | | |
| Assessment | | | | Predose | Dosing | EOI | Day 2 | Day 3 | рау о | Day 15 | Day 1 | Day 1 | | | | |
| Visit Window (Days) | | -14 unless<br>otherwise<br>indicated | | | | | | | | | | | | | 21 days<br>after last<br>dose <sup>a</sup> | |
| Informed consent for tumor tissue | X | | | | | | | | | | | | | | | |
| Informed consent (s) b | | X | | | | | | | | | | | | | | |
| Medical history<br>(including smoking<br>history) &<br>demographics | | X | | | | | | | 14 | | | | | | | |
| Inclusion / Exclusion | | X | | | | | | | | | | | | | | |
| Physical exam | | X | | X | | | | | X | X | X* | X* | | | X | |
| Vital signs | | X | | X | | X | | | X | X | X* | X* | | | X | |
| Height & weight c | | X | | X d | | | | | | | X*d | X* <sup>d</sup> | | | X <sup>d</sup> | |
| ECOG | | X | | X | | | 7 | | X | X | X | X | | | X | |
| Echo or MUGA e | | X | | | | | | | | | X e | X e | | | X | |
| ECG (12-lead) e | | X | | | | 1 | | | | | | | | | X | |
| Con Meds | | X | | X | | X | | | X | X | X* | X* | | | X | |
| Adverse Events | X f | X | | X | 7 | X | | | X | X | X* | X* | | | X | X <sup>g</sup> |
| PRO assessments h | | | | X | | | | | | | X | X | | | X | |
| CBC differential & platelets i | | X | | X d | | | | | X d | X d | X* d | X* <sup>d</sup> | | | X <sup>d</sup> | |
| Serum chemistries <sup>1</sup> | | X | | X d | | | | | X d | X d | X* d | X* d | | | X d | |
| GFR or estimated | | | | | | | | | | | | | | | | |
| serum creatinine clearance j | | X | | X | | | | | | | X | X | | | | |
| Coagulation | | X | | | | | | | | | | | | | | |
| Urinalysis | | X | | | | | | | | | | | | | X | |
| IxRS | | _ | X | | | | | | | | | | | | | |
| Intense PK k | | | | X d | | X | X | X | X | X | $X^{\dagger}$ | | | | | |
| Sparse PK (all) | | | | X d | | X | | | | | X | | | | X | |
| HAHA sample | | | | X d | | | | | | | X | | | | X | |
| Pregnancy test m | | X | | | | | | | | | | | | | X | |

| | Tissue<br>screen | Screen | Random-<br>ization | Cycle 1 (Weeks 1-3) | | | | | | | Cycles 2 & 3 | | End of<br>Cycle 6<br>& Every<br>4 Cycles | Every<br>6<br>weeks | End-of-<br>Study<br>Treatment<br>Visit | 40 Days<br>After<br>Last<br>Dose <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5010011 | | Lawron | | Day 1 | | Day 2 | Day 3 | Day & | Day 15 | Day 1 | Day 1 | | | | |
| Assessment | | | | Predose | Dosing | EOI | Day 2 | Day 3 | Day 0 | Day 13 | Day 1 | Day 1 | | | | |
| Patritumab Adm <sup>n</sup> | | | | | X | | | | | | X | X | | | | |
| Cetuximab Adm <sup>o</sup> | | | | | X | | | | X | X | X | X | | | | |
| Platinum Adm <sup>p</sup> | | | | | X | | | | | | X | X | | | | |
| PGx sample q | | | | X d | | | | | | | | | | | | |
| Tumor assessments <sup>r</sup> | | X | | | | | | | | | | | | X s | X | |
| Survival follow-up | | | | | | | | | | | | | | | | X <sup>t</sup> |
| Additional biomarker blood samples <sup>u</sup> | | | | X <sup>u</sup> | | | | | 10 | | X <sup>u</sup> | | X <sup>u</sup> | | X <sup>u</sup> | X <sup>u</sup> |

- a Last dose of any study drug administered.
- b Informed consent for main study (mandatory) and pharmacogenomics (optional).
- c Height measured only at Screening.
- d These assessments can be performed within 3 days prior to visit.
- e Echocardiograms/MUGA scans will be performed at Screening, Cycle 3, every third subsequent cycle, and End-of-Study Visit. Additional echocardiograms/MUGA scans and electrocardiograms may be performed at the discretion of the investigator. The same test (echocardiogram or MUGA) must be used for a subject throughout the study.
- f Collect SAEs only related to the biopsy procedure.
- g At 40 days after the last dose of study drug, a telephone call will epl ced to the subject to record adverse events.
- h PRO assessments will be administered before any study-rela ed procedures are performed.
- i Results must be available prior to dosing.
- j At Screening, either GFR or the estimated serum creatinin clear nce (mL/min) as an estimate of GFR will be calculated. The estimated serum creatinine clearance rate (CrCl; mL/min) will be calculated using the modified Cockcroft-Gault equation (Appendix 17.1). The estimated GFR will also be calculated before each cisplatin or carboplatin administration. This will be performed only until completion of chemotherapy.
- k Intensive serum PK in a subgroup of 30 subjects samples will be collected. See **** in the protocol for detailed information on sampling times.
- 1 See  in the protocol for detailed information on sampling times.
- m Pregnancy test must be confirmed negative before dosing. Additional pregnancy testing may be done at the discretion of the Investigator and/or if required by local regulations for women of child-bearing potential.
- Patritumab administered initially at 18 mg/kg and thereafter 9 mg/kg every 3 weeks as a continuous intravenous infusion over 60 minutes (±10 minutes). Infusion times can be extended to a maximum of 120 minutes for subjects unable to tolerate the 60-minute infusion.
- o Cetuximab infusions administered initially at 400 mg/m<sup>2</sup> IV over 2 hours and 250 mg/m<sup>2</sup> over 1 hour weekly. Cetuximab is administered 60 minutes after patritumab administration. Cetuximab is given on Days 1, 8, and 15.
- P Cisplatin infusions administered at 100 mg/m<sup>2</sup> IV over 1 hour and every 3 weeks up to a maximum of 6 cycles. For pre- and post-treatment hydration see Section Error!

  Reference source not found. in the protocol and according to institutional standards. Creatinine clearance required prior to cisplatin administration. Cisplatin administered 1 hour after cetuximab administration. If carboplatin is selected instead of cisplatin, administer carboplatin at AUC of 5 over 30-60 minutes every 3 weeks for a maximum of 6 cycles. See Section  in the protocol for carboplatin.
- q Genetic sampling is optional.
- r Tumor measurements will be assessed per RECIST Version 1.1. Baseline scans to be performed as part of eligibility during Screening. Existing radiographic scans can be used for the baseline evaluation if the scans were performed within 4 weeks prior to randomization.
- s Tumor assessments are to be performed every 6 weeks to Week 24 (+/- 3 days), then every 12 weeks (+/- 7 days) thereafter.
- t After discontinuation from study treatment, follow-up information for survival will be obtained per telephone approximately every 3 months for a minimum of 13 months.
- u Additional biomarker samples:
  Collect blood sample for cfDNA predose Cycle 1 Day 1, predose Cycle 2 Day 1, End of Cycle 6, predose every 4 Cycles, at progression (end of study treatment), and 40 days after last dose of study drug administered.
  - Collect blood samples for exosome at: predose Cycle 1 Day 1, predose Cycle 2 Day 1, and End of Cycle 6. Refer to the laboratory manual for instructions on collection and management of samples.
- \* Can be collected on Days 8 and 15 in all subsequent cycles at the discretion of the Investigator.
- † Corresponds to Cycle 1, Day 21 (504 hrs)—see  in the protoc 1.

Table 3.1.2: Schedule of Events for Extension Phase

| | Additional cycles | | Every 3 months | End of<br>Treatment | 40 days after last dose <sup>a</sup> |
|---|---|---|---|---|---|
| | Predose | Dosing | | | |
| Visit Window (Days) | | | | | |
| Physical Exam | X | | | X | |
| Vital Signs | X | | | X | |
| Adverse Events | X | | C | | X |
| CBC diff and platelets <sup>b</sup> | X b | | 1 | X b | |
| Serum chemistries b | X b | | | X b | |
| HAHA and PK sample <sup>c</sup> | | | X | | |
| Patritumab Adm <sup>d</sup> | | X | | | |
| Cetuximab Adm <sup>e</sup> | | X | | | |
| Additional biomarker blood samples | | | X | X | X |

- a Last dose of any study drug administered.
- b CBC and chemistries must be performed within 3 days of dosing
- For subjects with positive HAHA at the End of Study Trea ment visit, dditional serum HAHA samples should be collected every 3 months up to 1 year from the last dose of study drug or if the subject starts another ther py for canc r, or withdraws consent from the study, whichever occurs first.
- d Patritumab administered at 9 mg/kg every 3 weeks as continuous intravenous infusion over 60 minutes (±10 minutes). Infusion times can be extended to a maximum of 120 minutes for subjects unable to tolerate the 60 minute infusion.
- e Cetuximab is infused at 250 mg/m<sup>2</sup> over 1 hour weekly. Cetuximab can be administered directly after patritumab administration.



#### 3.2. Study Population

Adult subjects with metastatic SCCHN originating from the oral cavity, oropharynx, hypopharynx, and larynx with documented disease recurrence following previous treatment for non-metastatic disease will be enrolled. A subject is considered enrolled in the study upon the Investigator or designee obtaining written informed consent from the subject, and upon determination that all inclusion and exclusion criteria have been satisfied.

#### 3.3. Randomization and Blinding

#### 3.3.1. Randomization

Approximately 105 subjects who have an HRG expression value and HPV status (+/-) will be assigned randomly in a blinded manner by the Interactive Web/Voice Response System (IXRS) to the patritumab or the control arms in a 2 1 stratification (approximately 70 HRG-high and approximately 35 HRG-low subjects)

The IXRS will manage the number of HRG-high and HRG-low patients randomized. Once the maximum number of HRG-low subjects has been randomized, the IXRS will not allow enrollment of additional HRG-low subjects. To ensure balance between treatment groups, subjects will additionally b stratified according to HPV status (positive, negative).

Randomization to treatment groups will be achieved using IXRS. The time between randomization and the initiation of treatment should be as short as possible and no more than 3 business days.

# 3.3.2. Blinding

This study is randomized, placebo-controlled, double blinded study. The treatment assignments will be blinded to the subjects, the investigators, site staff, and all persons involved in reviewing the clinical data, including CRO personnel in clinical and trial management and Sponsor personnel, with the exception of the Data Monitoring Committee, who will review the unblinded clinical data on an ongoing basis.

#### 3.3.2.1. Unblinding at Primary Analysis

At the point of primary analysis, as defined in Section 7 of this SAP, the treatment assignment for all subjects randomized will only be unblinded to CRO and sponsor statisticians and programmers directly involved in performing the analyses after data are reconciled and cleaned and a snapshot of the clean database is created. To minimize potential bias, subjects and investigators will not be informed about individual treatment assignment until study closure. Any datasets containing potentially unblinded information (i.e., patritumab PK and HAHA) will have their access restricted. The study statistician will maintain a list of the individuals who have access to individual treatment assignments and/or data that potentially unblinds the study. This list will include the date and level of unblinding and rationale for unblinding.

#### 3.3.2.2. Unblinding at Study Closure

For the purpose of database lock and generation of the clinical study report (CSR), the study will be considered closed when OS data will be considered mature. At study closure, all subjects will be unblinded for final analysis after the final database is locked. Any subject remaining on study treatment and appears to continue to benefit (ie, SD or better) from treatment may continue to receive study treatment.

# 3.3.2.3. Emergency Unblinding

In the case of a rare emergency where, in the opinion of the Investigator, discontinuation of study drug is not sufficient and study treatment must be unblinded to evaluate further course of medical treatment. The investigator is encouraged to contact the CRO medical monitor to discuss their rationale for unblinding. However, to prevent delays to the investigator or medical personnel responding to a potentially emergent situation, unblinding of the study treatment will not be dependent pon the investigator receiving approval from the CRO medical monitor. The method for determining a subject's treatment assignment once a subject is randomized in the study is through the IxRS. The investigator and one designated subinvestigator will have access to perform emergency unblinding in the IxRS. The treatment assignment of the selected subject randomized at their site will be revealed to the investigator performing the IxRS call upon completion of the emergency unblinding call. The investigat r must contact CRO medical monitor by telephone with an explanation of the need for opening the treatment assignment code within 24 hours of opening the code. A detailed procedure is described in the protocol.

#### 3.4. Study Assessments

The table in Section 3.1, above, presen s the visit schedule and procedures of the study to be conducted at each visit.

# 4. SAMPLE SIZE DETERMINATION

The primary efficacy endpoint is PFS. The sample size for this study is based on the number of required PFS events in the HRG-high stratum. For PFS, a clinically meaningful improvement is defined as 79% increase from median PFS of 4.2 months in the control arm to median PFS of 7.5 months in the patritumab arm (that is a HR of 0.56). A total of 70 HRG-high subjects will be randomized to observe 53 PFS events in the HRG high stratum assuming a one-sided alpha of 0.10, 80% power, and a 1:1 randomization ratio between 2 arms, a 12-month enrollment and 10-month follow-up, and 10% dropouts.

Under 2:1 (HRG high vs. low) stratification, a total of approximately 105 subjects (70 HRG high subjects and 35 HRG low subjects) will be randomized in both strata to observe at least 75 PFS events. The sample size from bo h strata combined will provide approximately 81% power to detect a HR=0.56 in PFS assuming one-sided alpha of 0.05 and other same assumptions above if HRG high stratum does not show statistical significance in PFS.

The sample size computation is performed using the test based on Survival Superiority Trials: Two Sample Test – Logrank Test: Given Accrual Duration and Study Duration in the EAST software (version 5.3, Cytel Inc.).

# 5. STUDY VARIABLES

# 5.1. Efficacy Variables

Efficacy variables include PFS, OS, ORR (CR and PR), duration of response, time to response, time to disease progression, and duration of SD.

Tumor response assessments, including subjects who discontinued from treatment, will be performed every 6 weeks ( $\pm$  3 days) for the first 24 weeks independent of treatment cycle until disease progression, death, start of new anticancer therapy, withdrawal of subject consent, lost to follow-up, or study closure, whichever occurs first. After 24 weeks, tumor assessments will be performed every 12 weeks ( $\pm$  7 days).

# **5.1.1.** Primary Efficacy Variable

The primary efficacy variable is PFS. PFS is defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1 as assessed by investigator) or death due to any cause. Progressive Disease is defined as  $\geq 20\%$  increase in the sum of diameters of target lesions; taking as reference the mallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions s also considered progression).

Subjects with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "clinical progression." Every effort should be made to document objective progression even after discontinuation of treatment. Symptomatic deterioration is not a descriptor of an objective response: it is a reason for stopping study therapy. The objective response status of such subjects is to be determined by evaluation of target and non-target disease. If a radiographic tumor assessment has not been performed within 4 weeks of the time of clinical progression, then another radiographic assessment should be performed without waiting for the next regularly scheduled scan.

For equivocal findings of progression (ie, very small and uncertain new lesions, cystic changes, or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

The rules for censored cases are defined as follows:

1. Subjects who are alive with no objective documentation of radiographic disease progression by the data cut-off date for the PFS analyses will be censored at the date of the last post-baseline evaluable tumor assessment. The evaluable tumor assessment is defined as the overall response for tumor assessment being not "Inevaluable" recorded on the Case Report Form (CRF) page "overall tumor assessment". If there is no post-baseline evaluable tumor assessment, the subject will be censored at the date of randomization.

- 2. Subjects who start other anti-cancer therapy including surgical or radiologic intervention given with curative intent prior to progression or death will be censored at the date of the last post-baseline evaluable tumor assessment prior to starting other anti-cancer therapy. If there is no post-baseline evaluable tumor assessment prior to starting other anti-cancer therapy, the subject will be censored at the date of randomization.
- 3. Subjects who progress or die after ≥2 consecutive missed tumor assessment visits will be censored at the date of the last evaluable tumor assessment prior to progression or death. In this study, progression or death after ≥2 consecutive missed tumor assessment visits is defined as progression or death that occurs more than 13 weeks (two tumor assessment visits plus 1 week visit window) since the last post-baseline evaluable tumor assessment. If there is no post-baseline evaluable tumor assessment prior to the tumor assessment of progressive disease or death and progression or death occurs more than 13 weeks since the date of randomization, the subject will be censored at the date of randomization;
- 4. Subjects without baseline tumor assessment will be censored at the date of randomization.

# 5.1.2. Secondary Efficacy Variables

Secondary efficacy variables include OS and ORR (CR and PR).

# 5.1.2.1. Overall Survival (OS)

OS is defined as the time from the date of randomization to death due to any cause. Subjects who are alive at the time of data cut off for OS analysis will be censored at the last contact date at which the subject is known to be alive.

Survival status data will be obtained from deaths reported in the CRFs and Survival follow-up communications every 3 months after a subject discontinues from study treatment.

The last contact date is defined as the last date the subject was known to be alive at the analysis cut-off. The date will be the latest date among the following:

- Last non-missing assessment/onset date captured under the following eCRF pages (or if a date of assessment/onset is not available the "date of visit" for the eCRF page can be used): adverse events, vital signs, physical examination, ECOG PS, ECG, Echocardiogram or MUGA scan, safety laboratory test, tumor assessment, patient-reported outcomes assessment, hospitalization and also assessment date in third-party data such as PK, HAHA etc.
- Last dosing date of study medication, last date of concomitant medications, and last date of non-drug treatments/procedures.
- Start date of subsequent anti-cancer therapy administered after study treatment discontinuation.
- Date of Last Contact collected on the survival follow up page of the eCRF.

• Date of Last Contact collected on the final subject status (or end of study status) page of the eCRF.

# 5.1.2.2. Object Response Rate (ORR)

ORR is defined as the proportion of subjects with the best overall response of CR or PR. A confirmation of CR/PR is not required for this study as per RECIST Version 1.1.

The best overall response is defined as the best response (in the order of CR, PR, SD, and PD) among all overall responses recorded from the start of treatment until the subject is withdrawn from the study. The best overall response of PD corresponds to disease progression (assessment based upon tumor measurements and recorded on the CRF page "overall tumor assessment") for the first valid post-treatment tumor assessment. If there is no post-treatment tumor assessment, the best overall response will be assigned as "Inevaluable". In the case of a best overall response of SD, measurements must have met the SD criteria at least once after study entry at a minimum time interval from baseline. A best overall response of SD must be assessed a minimum of 39 days (6 weeks – 3 day visit window) after the date of randomization. If this minimum requirement is not met, the best overall response will be determined starting with the next tumor assessment. If there is no next tumor assessment, the best overall response will be assigned as "Inevaluable".

# **5.1.3.** Exploratory Efficacy Variables

Duration of response, time to response, time to disease progression and duration of SD will be exploratory efficacy variables examined in this study.

#### 5.1.3.1. Duration of Response

Duration of response is defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease (disease progression as assessed based upon tumor measurements and recorded on the CRF page "overall tumor assessment"). If a subject is discontinued or is lost to follow-up with no documentation of progressive disease, duration of response is defined as the time from the date of the first documentation of objective response to the date of the last evaluable tumor assessment as a censored value. The rules for censored cases are defined as follows:

Subjects who progress after  $\geq 2$  consecutive missed tumor assessment visits will be censored at the date of the last evaluable tumor assessment prior to the tumor assessment of progressive disease. In this study, progression after  $\geq 2$  consecutive missed tumor assessment visits is defined as progression that occurs more than 13 weeks (two tumor assessment visits plus 1 week visit window) since the last post-baseline evaluable tumor assessment. Subjects who start other anti-cancer therapy prior to progression will be censored at the date of the last post-baseline evaluable tumor assessment prior to starting other anti-cancer therapy.

Duration of response will be measured for responding subjects (PR or CR) only.

#### **5.1.3.2.** Time to Response

Time to response is defined as the time from the date of randomization to the date of the first documentation of objective response (CR or PR). Time to response will be measured for responding subjects (PR or CR) only.

#### **5.1.3.3.** Time to Disease Progression (TTP)

Time to progression is defined as the time from the randomization date to the date of first objective documentation of radiographic disease progression (per RECIST v1.1 as assessed by investigator). Objective documentation of disease progression is based upon "Overall Response" recorded as "Progressive Disease (PD)" on the CRF page: "overall tumor assessment". The rules for censored cases of TTP and duration of response are similar to the censoring of PFS, except that subjects who die before disease progression is document are censored for the former.

#### **5.1.3.4.** Duration of Stable Disease (SD)

Duration of stable disease is defined for subjects whose best response is SD as the time from the date of randomization to the date of the first documentation of progressive disease (disease progression as assessed based upon tumor measurements and recorded on the CRF page "overall tumor assessment"). Censoring rules are the same as described above for duration of response.

#### 5.2. Safety Variables

#### **5.2.1.** Adverse Events

The following safety variables will be assessed in this study according to the Schedule of Events (Table 3.1.1 and Table 3.1.2) in Section 3.1.

- A Treatment-eme g nt adverse event (TEAE) is defined as an Adverse Event (AE) that emerges during treatment, having been absent at pretreatment, or reemerges during treatment, having been present at baseline but stopped prior to treatment, or worsens in severity since treatment relative to the pretreatment state, when the AE is continuous. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, Version XX.X), and graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
- AEs of Special Interest
- Interstitial Lung Disease (ILD)
  - ILD is defined as an acute onset of new or progressive pulmonary symptoms, such as dyspnea, cough or fever.
- Combined Elevations of Aminotransferases and Bilirubin
   Hepatic events, both serious and nonserious, presenting with combined abnormalities meeting criteria for a potential "Hy's law" case [i.e., Alanine

aminotransferase (ALT) or Aspartate aminotransferase (AST)  $\geq$  3 x ULN, with simultaneous total bilirubin  $\geq$  2 x ULN].

# **5.2.2.** Clinical Laboratory Evaluations

Safety laboratory assessments will include hematology, serum chemistry, coagulation, and urinalysis.

- Coagulation (only at Screening): prothrombin time, international normalized ratio, and partial thromboplastin time
- Hematology: CBC including hemoglobin, hematocrit, white blood cell count (WBC) with 5 part differential (including absolute neutrophil count), red blood cell, and platelet count
- Serum chemistry: bicarbonate, calcium, phosphorus, magnesium, albumin, glucose, serum creatinine, uric acid, total protein, urea, AST, ALT, lactic dehydrogenase, alkaline phosphatase, total and direct bilirubin, sodium, potassium, and chloride
- Routine urinalysis: dipstick and microscopy (if indicated), including protein, specific gravity, glucose, and blood
- Serum or urine β-HCG pregnancy t st

At Screening, creatinine clearance (mL min) or GFR will be calculated. This will also be done before each cisplatin or carboplatin administration.

# 5.2.3. Vital Signs

Vital sign measurements include blood p essure, heart rate, temperature, height, and weight.

### 5.2.4. ECG

A 12-lead ECG will be performed within 14 days prior to Screening, at the End of Study Treatment visit, and during the study at the discretion of the Investigator.

#### **5.2.5.** Physical Examinations

Physical examinations will evaluate the following body systems/organs: respiratory, cardiovascular, gastrointestinal, musculoskeletal, genitourinary/reproductive (optional), psychiatric (optional), hematological, neurological, immunological, head, eyes, ears, nose and throat, and other. Abnormal physical examination findings that are new or changed will be reported as AEs.

#### 5.2.6. Other Safety Variables

An echocardiogram or multigated acquisition (MUGA) scan will be performed at screening, and at End-of-Study Treatment visit and during the study at the discretion of the Investigator.

The presence of anti-patritumab neutralizing antibody in serum will be assessed. Blood samples will be taken on Day 1 of Cycle 1 (preinfusion), Cycle 2 (preinfusion), Cycle 3 (preinfusion), and at End-of-Study Treatment visit. For subjects with positive anti-patritumab neutralizing antibody on the serum sample drawn at the end of study treatment visit, additional serum samples should be obtained for antibodies, until the antibody level returns to baseline (or becomes negative) or up to 1 year from the last dose of study drug or if the subject starts another therapy for cancer, whichever occurs first.

#### 5.3. Pharmacokinetic Variables

#### **5.3.1.** Concentration Data

Serum concentrations for patritumab will be collected at Cycles 1- 3 and at End of Study Treatment (Table 8.1 of the Protocol).

For a subset of 30 subjects, a blood sample for PK analyses of patritumab, cetuximab, and platinum concentrations will be obtained at the time points, relative to the start of patritumab infusion at Cycle 1 (Table 8.2 of the Protocol) This will be an intense pharmacokinetic (PK) assessment.

# 5.3.2. Pharmacokinetic (PK) Parameters

PK parameters (AUC<sub>0-21d</sub> and Cmax) will be calculated from the individual concentrations of patritumab, cetuximab, cisplatin and carboplatin using non-compartmental methods. PK parameters will be derived for the intensive PK sampling (i.e. Cycle 1) for patritumab, cetuximab cisplatin and carboplatin.

# 5.4. Pharmacodynamic (PD) Variables

Not Applicable.

#### 5.5. Biomarkers

A predictive biomarker will be analyzed with the intent of identifying those subjects who might derive clinical benefit from treatment with patritumab. Heregulin is the candidate biomarker prospectively selected as the single predictive biomarker. Heregulin messenger RNA will be measured in tumor samples using a quantitative reverse transcription polymerase chain reaction assay.

HPV status or p16 will be evaluated in all tumor tissue in this study.

Further exploratory tissue, soluble, or genomic biomarkers in subject tissue and blood samples (possibly including circulating cell-free DNA and exosomes) may be analyzed based on emerging scientific knowledge to better understand the target disease and also the effects of study treatment.

#### 5.6. Other Variables

# **5.6.1.** Eastern Cooperative Oncology Group Performance Status

The Eastern Cooperative Oncology Group (ECOG) performance status will be determined at Screening, and then at each scheduled visit throughout the study.

# **5.6.2.** Patient Reported Outcomes

Patient-reported outcomes will be used to evaluate study treatment in subjects treated with patritumab + cetuximab + platinum-based therapy compared to placebo + cetuximab + platinum-based therapy.

# Functional Assessment of Cancer Therapy—Head and Neck (FACT-H&N) Instrument

The FACT-H&N contains 4 general subscales (total 27 items) measuring physical well-being (PWB), functional well-being (FWB), social well-being (SWB), emotional well-being (EWB), and a Head and Neck Cancer symptom-sp cific subscale – the 12-item Head and Neck Additional Concerns Subscale (HNS). Each of the 39 FACT- H&N items is rated on 5-point scales, ranging from 0=not at all to 4=very much, where higher scores represent more favorable patient-reported outcomes.

Combining the 10 symptom-related items out of the 39 FACT-H&N items – "I have a lack of energy" (PWB item 1), "I have nausea" (PWB item 2), "I have pain" (PWB item 4), "I worry that my condition will get worse" (EWB item 6), "I am content with the quality of my life right now" (FWB item 7), "I have trouble breathing" (Additional Concerns item 3), "I can swallow naturally and easily" (Additional Concerns item 7), "I am able to communicate with others" (Additional Concerns item 10), "I can eat solid foods" (Additional Concerns item 11), and "I have pain in my mouth, throat or neck" (Additional Concerns item 12) - yields a 10-item FACT-Head and Neck Symptom Index (FHNSI).

Specifically, 7 specific summary scores will be evaluated,

- PWB score
- FWB score
- SWB score
- EWB score
- HNS score
- FHNSI score
- FACT-H&N total score

The FACT-H&N Total Score ranges from 0-156. The PWB score, SWB score and EWB score range from 0 to 28. The EWB score ranges from 0 to 24. The HNS score and the FHNSI score ranges from 0 to 48. The FACT-H&N total score, PWB score, FWB score,

SWB score, EWB score, HNS score and FHNSI score will be analyzed as exploratory efficacy parameters.

Use following algorithm to determine the individual subscale scores:

- Physical well-being (PWB): PWB score = Sum (GP1-GP7) x 7/number of nonmissing items. If the number of missing items (GP1-GP7) is greater than 3, then set PWB score = missing.
- Social well-being (SWB): SWB score = Sum (GS1-GS7) x 7/number of nonmissing items. If the number of missing items (GS1-GS7) is greater than 3, then set SWB score = missing.
- Emotional well-being (EWB): EWB score = Sum (GE1-GE6) x 6/number of nonmissing items. If the number of missing items (GE1-GE6) is greater than 3, then set EWB score = missing.
- Functional well-being (FWB): FWB score = Sum (GF1-GF7) x 7/number of nonmissing items. If the number of missing items (GF1-GF7) is greater than 3, then set FWB score = missing.
- Additional Concern (HNS): HCS score = Sum (H&N1-H&N12) x 12/number of nonmissing items. If the number of missing above items is greater than 6, then set HCS score = missing.
- Additional Concern (HNS): HCS score = Sum (H&N1-H&N12) x 12/number of nonmissing items. If the number of missing above items is greater than 6, then set HCS score = missing.
- FHNSI: FHNSI score = Sum of 10 symptom-related items x 10/number of nonmissing items. If the number of missing above items is greater than 5, then set FHNSI score = missing.
- FACT-H&N total score: FACT-H&N score = Sum (PWB, SWB, EWB, GFB, HCS). If any of the above items is missing, then set FACT-H&N score = missing.

#### **EuroQoL-5 Dimensions-5 Levels Instrument**

The EQ-5D-5L is a preference based measure of health status that is now widely used in clinical trials, observational studies, and other health surveys.

The EQ-5D-5L consists of 2 pages – the EQ-5D-5L descriptive system and the EuroQoL Visual Analogue scale (EQ VAS). The descriptive system comprises the following 5 domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each domain has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box with the most appropriate statement in each of the 5 domains. This decision results in a 1-digit number expressing the level selected for that domain. The digits for 5 domains can be combined in a 5-digit number or profile describing the respondent's health state.

As index-based values have not been evaluated for the EQ-5D-5L at this time, crosswalk value sets developed based on the EQ-5D-3L index-based values will be applied. The crosswalk value set for the United Kingdom will be used for analyses overall and for all regions. The value set provides an index score for each health state and can be accessed at:

(http://www.euroqol.org/fileadmin/user\_upload/Documenten/Excel/Crosswalk\_5L/EQ-5 D-5L Crosswalk Value Sets.xls).

The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'. This information is used as a quantitative measure of health as judged by the individual respondents. The instructions for the EQ VAS asks respondents to 'mark an X on the scale to indicate how your health is TODAY' and then to 'write the number you marked on the scale in the box below.

# 6. ANALYSIS SETS

# 6.1. Analysis Sets Definitions

# 6.1.1. Full Analysis Set

The full analysis set (FAS) will be based on the intent-to-treat principle and will comprise all subjects randomized into the study. Subjects will be analyzed as randomized.

# 6.1.2. Safety Analysis Set

The safety analysis set includes all subjects who received any amount of study medication. Subjects will be analyzed according to actual treatment received.

# 6.1.3. Per-Protocol Analysis Set

The per-protocol analysis set will include all subjects in the FAS who have completed at least 1 cycle of treatment, and who were sufficiently compliant with the protocol and without major protocol violation. Full criteria for defining sufficient compliance will be finalized and documented prior to database unblinding.

# 6.1.4. Pharmacokinetic Analysis Set

The PK analysis set will include all sub ects who have received at least 1 dose of study drugs and have evaluable patritumab or cetuximab concentrations.

### 6.1.5. Patient Reported Outcome Analysis Set

There will be 2 PRO Analysis Sets:

- FACT-H&N An lysis Set
- EQ-5D Analysis Set.

The FACT-H&N Analysis Set will include all subjects in the Full Analysis Set who complete the FACT-H&N assessment at Cycle 1 Day 1, at least partially in a manner that permits imputation of missing responses, according to the approach described in Section 5.6.2.

The EQ-5D Analysis Set will include all subjects in the Full Analysis Set who complete the EQ-5D assessment at Cycle 1 Day 1, at least partially in a manner that permits imputation of missing responses, according to the approach described in Section 5.6.2.

#### 6.2. Protocol Deviations

A list of protocol deviations for the study report will be presented in a data listing.

#### **6.3.** Treatment Misallocations

The following rules of reporting efficacy and safety results (eg, under which treatment group) for subjects with errors in treatment allocation will be applied.

#### If subjects are:

- Randomized but not treated, then they will be reported under their randomized treatment group for efficacy analysis. However, they are by definition excluded from the safety analysis as actual treatment is missing.
- Treated but not randomized, then by definition they will be excluded from the efficacy analyses since randomized treatment is missing, but they will be reported under the treatment they actually received for all safety analyses.
- Randomized but took incorrect treatment, then they will be reported under their randomized treatment group for all efficacy analyses, but will be reported under the treatment they actually received for all safety analyses.



# 7. GENERAL STATISTICAL CONSIDERATIONS

This is a multicenter randomized Phase 2 study designed to evaluate the safety and efficacy of patritumab in combination with cetuximab and platinum-based therapy in recurrent/metastatic first-line SCCHN. The primary analyses for this study will occur when at least 53 PFS events have been observed in the HRG high stratum.

At the point of primary analysis for PFS, the treatment assignment for all randomized subjects will be unblinded to designated study personnel for the analysis after data are reconciled and cleaned and a snapshot of the clean database is created. To minimize potential bias, subjects and Investigators will not be informed about individual treatment assignment until study closure.

Final analyses will occur after study closure with mature OS data (i.e., when all subjects have died or a minimum of 13 months after the last subject is randomized whichever comes first). At the time of study closure, subjects who are demonstrating clinical benefit (SD or better) from study treatment may be offered an opportunity to continue study treatment on the extension phase.

Assessments of change from baseline to post b seline or the ratio of post baseline to baseline will include only those subjects with both baseline and post baseline measurements. The last nonmissing value of a variable taken before the first dose of study drug will be used as the baseline value, unless otherwise specified. In general, missing or dropout data will not be imput d for the purpose of data analysis. Descriptive summary statistics (n, mean, median, standard deviation, and range) will be calculated for continuous variables, and for categorical variables, the number and percentage in each category will be displayed by treatment group.

Study Day is calculated as  $< date - 1^{st}$  study treatment date + 1 >. The date of the first study treatment is Day 1

# 7.1. Adjustment for Covariates

No other covariate adjustments will be applied for primary and secondary efficacy analyses, except for the stratification variables if applicable. The PRO analyses will use baseline values of the dependent variable as a covariate in a mixed model.

# 7.2. Handling of Dropouts or Missing Data

For a description of the handling of censored data for efficacy endpoints such as OS, PFS and TTP, see Section 5.1 above. Imputation of partial or missing AE onset date and concomitant medication date, incomplete tumor assessment dates, and incomplete dates for last contact or death are specified in Section 11.1. The missing data handling for the analyses on patient reported outcomes is described in 5.6.2.1.

#### 7.3. Interim Analyses and Data Monitoring

An independent Data Monitoring Committee (DMC) will be established for this study and will review the ongoing safety of the study participants and monitor the overall

conduct of the clinical trial. The DMC will review accumulating safety data at periodical basis. Based on its ongoing review of the unblinded safety data, the DMC will outline any serious safety concerns and make recommendations to continue, modify, suspend, or terminate the study.

Details on the membership, responsibilities and working procedures of the Independent DMC will be described in the DMC Charter, provided as a separate document in the study file. The same independent Data Analysis Group statistician responsible for providing the safety data will also provide efficacy data (for proper assessment of the risk/benefits of continuing treatment and study) to the DMC for review.

#### 7.4. Multicenter Studies

There will be approximately 35 sites in Europe. Site as a factor will not be formally examined in this study.

# 7.5. Multiple Comparisons/Multiplicity

This study has only one primary efficacy variable PFS. The testing hypotheses to compare PFS the patritumab arm versus the control arm will be performed in two sequential steps in pre-defined populations (Freidlin 2012 et al). The primary analysis is PFS comparison between the patritumab arm and the control arm in HRG-high stratum of the FAS (Step 1). If the testing in Step 1 is significant, then no further testing will be performed in Step 2 and the 80% confid n e intervals of the hazard ratio in HRG low stratum will be estimated. If the testing in Step 1 is not significant, then the testing in FAS (HRG high + low) will be performed in Step 2 (See Section 8.2.1). The results from both steps will be used to guide the decision on future Phase 3 designs. Since this is a proof of concept study, no adjustment for multiplicity will be performed.

# 7.6. Examination of Subgroups

As exploratory analyses, subgroup analysis (e.g. age, sex, HRG, HPV, primary tumor site, etc) for selective efficacy endpoints will be conducted (Section 8.2.4).

# 8. STATISTICAL ANALYSIS

# 8.1. Study Population Data

#### 8.1.1. Subject Disposition

Subject disposition will be summarized by randomized treatment group and overall for All Screened Subjects. The number and percentage of subjects in the Full Analysis Set, the Per Protocol Analysis Set, the Safety Analysis Set, the Pharmacokinetics Analysis Set, and the PRO Analysis Sets will be presented. Subject status (ongoing, if any, and discontinued from study treatment) and the reasons for discontinuation (as reported on CRF EOT page) will be summarized in this table. All percentages, except those for All Screened Subjects, will be based on the Full Analysis Set. A listing will present data relevant to subject disposition.

#### **8.1.2.** Protocol Deviations

Protocol deviations collected by clinical team, as well as those identified in the CRF data will be provided in a listing.

Protocol deviations will be finalized prior to database lock.

# 8.1.3. Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized by treatment group and overall for the FAS as well as the HRG-high stratum of the FAS, Per-Protocol analysis set (if substantial differences such as >5% as compared to the FAS), and Safety Analysis Set. If two sets of subjects are dentical to each other, analysis will only be performed once.

Demographic characteristics consist of age, gender, race, and ethnicity. A subject's age in years is calculated using the informed consent date and the birth date [(consent date-birthdate)/365.25]. Age will additionally be categorized as ( $\leq$  65, > 65) for reporting purposes.

Baseline characteristics consist of height, weight, tumor stage at study entry, tumor grade, prior systemic cancer therapy (Yes or No), prior radiation therapy (Yes or No), time from diagnosis of SCCHN to study treatment, histology subtype, HRG value, HPV Status, tobacco history (cigarettes and cigars), ECOG performance status, and ECG findings at baseline.

Individual subject listings of all demographic, baseline characteristics, SCCHN cancer history, medical and surgical history including prior cancer history and prior cancer surgery, and prior cancer therapy will be provided.

# 8.2. Efficacy Analyses

Efficacy analyses will be performed on the FAS and per-protocol analysis set as well as HRG strata. Subjects will be analyzed according to the treatment assigned at randomization.

#### 8.2.1. Analysis of Primary Efficacy Variables

The primary efficacy endpoint is PFS as defined in Section 5.1.1 of this SAP. Progression will be determined based on the investigators' assessment.

The primary efficacy analysis will be the comparison of PFS between the patritumab arm and the control arm in HRG-high stratum of the FAS using the stratified log-rank test. For a description of the handling of censored data for efficacy endpoint PFS, see Section 5.1 above.

The testing hypotheses to compare PFS for the patritumab arm versus the control arm will be performed in two sequential steps (Freidlin 2012 et al). In step 1, the null hypothesis that PFS is the same for both arms in the HRG high stratum of FAS is tested at the one-sided 0.10 significance level. If this test in step 1 does not reject the null hypothesis, then in step 2A, the null hypothesis that PFS is the same for both arms in the FAS (HRG high stratum + low stratum) will be t s ed at the one-sided 0.05 significance level. If the test in step 1 is rejected, then in st p 2B, the two-sided 80% confidence interval (CI) for hazard ratio (HR) of PFS in the HRG low stratum of the FAS will be estimated.

The comparison of PFS between the patritumab arm and the control arm will be performed using a log-rank test stratified by the stratification factors.

Hypothesis testing for superiority with regard to PFS will be performed with a 1-sided hypotheses setting.

Suppose that  $S_A(t)$  and  $S_P(t)$  are the cumulative survival functions for PFS in patritumab and control treatment groups, respectively. The null hypothesis  $H_0$  with PFS:

 $H_0$ :  $S_A(t) = S_P(t)$  for all  $t \ge 0$  (identical survival functions for both groups) will be tested against the 1-sided alternative hypothesis  $H_A$ :

 $H_A$ :  $S_A(t) \ge S_P(t)$  for all  $t \ge 0$  and  $S_A(t) > S_P(t)$  for at least some t > 0

(improvement in PFS in the patritumab group over the control group)

The stratified log-rank test will be conducted using SAS PROC LIFETEST where the STRATA statement will include the treatment group and the stratification factors [HPV (positive vs other) and HRG (high vs. low, only for the FAS) at randomization]. The 1-sided p-value will therefore be obtained and  $H_0$  will be rejected if p-value  $\leq$  the prespecified 1-sided alpha.

The Kaplan-Meier product-limit method will be used to estimate the distribution of PFS for the patritumab arm versus the control arm. The median PFS for each treatment group will be based on the Kaplan-Meier estimate and the 95% confidence intervals for each treatment group will be calculated using the method of Brookmeyer and Crowley. The

median and confidence interval will be reported in months, and days will be converted to months by dividing by 30.4. The corresponding Kaplan-Meier curves will also be presented.

Estimates of HR between 2 arms along with their two-sided 80% and 95% CIs will be calculated using stratified Cox proportional hazards regression model. SAS PROC PHREG with the treatment group as the model covariate and stratification factors [HPV (positive vs other) and HRG (high vs. low) at randomization] as the STRATA variables will be used for this model. The Efron's method will be used to handle ties.

The above analysis for PFS will be repeated for the per-protocol analysis set. A separate analysis which includes clinical progression as a PFS event will be done as a sensitivity analysis.

# 8.2.2. Analysis of Secondary Efficacy Variables

#### 8.2.2.1. Overall Survival

OS will be analyzed in the same manner as for PFS. Estimates of HR between the patritumab arm and the control arm along with their two-sided 80% and 95% CIs will be calculated using stratified Cox proportional hazards regression model. SAS PROC PHREG with the treatment group as the model covariate and stratification factors at randomization as the STRATA variables will be used for this model. The Efron's method will be used to handle ties. The corresponding Kaplan-Meier curves will also be presented.

#### 8.2.2.2. Objective Response Rate

The number and the percentage of the subjects with the best overall tumor responses of either CR or PR (the objective response) will be tabulated by treatment group. Percentages will be calculated based on the number of subjects in the respective treatment group. The differences in the ORR between the control arm and patritumab arm will be presented along with two-sided 80% and 95% CIs based on the Wilson's score method with continuity correction.

In addition, the percent change from baseline will be calculated for the sum of longest diameters (LD) for all target lesions at each post-treatment evaluation for each subject, if applicable. The percent change in the sum of longest diameters from baseline in target lesions will be summarized by treatment group and assessment time with descriptive statistics; the largest decrease from baseline will also be summarized and displayed in the waterfall plots.

Best overall response and tumor assessments (target lesions, non-target lesions and overall) will be listed for all subjects in the Full Analysis Set. Percent change from the nadir (i.e., minimum sum of LD, including baseline, if that is the minimum value, up to the preceding tumor assessment) will be presented in the listing for target lesions.

# 8.2.2.3. Cutoff for HRG Expression

HRG expression value will be summarized by treatment group for overall, HRG-high, and HRG-low group with summary statistics. The distribution of HRG values will be plotted with histogram and normal curves.

HRG expression values will be dichotomized at alternative cutoffs to form new HRG-high and HRG-low groups. Analysis of PFS and OS specified in Section 8.2.1 and Section 8.2.2.1 will be performed for newly classified HRG high and low groups at alternative cutoffs. The results will be used to select optimum HRG cutoff.

# 8.2.3. Analysis of Exploratory Efficacy Variables

Exploratory efficacy endpoints include duration of response, time to disease progression, and duration of SD.

#### 8.2.3.1. Duration of Response

The distribution of duration of response as defined in Section 5.1.4.1 of this SAP will be presented as Kaplan Meier plot, together with response duration quartiles for responding subjects (PR or CR). Median time to response will be stimated along with two-sided 80% and 95% CIs using Kaplan-Meier methods

#### 8.2.3.2. Time to Response

The distribution of time to response as defined in Section 5.1.4.2 of this SAP will be presented as Kaplan Meier plot, together with response duration quartiles for responding subjects (PR or CR). Median time to response will be estimated along with two-sided 80% and 95% CIs using Kaplan Meier methods.

#### 8.2.3.3. Time to Disease Progression

Median time to disease progres ion will be estimated along with two-sided 80% and 95% CIs using Kaplan-Meier methods by treatment. In addition, summary statistics for 25% and 75% percentiles will be estimated using Kaplan-Meier methods.

#### **8.2.3.4.** Duration of Stable Disease

The distribution of duration of stable disease as defined in Section 5.1.4.4 of the SAP will be presented as Kaplan Meier plot, together with response duration quartiles for responding subjects with the best response of stable disease. In addition, median duration of stable disease will be estimated along with two-sided 80% and 95% CIs using Kaplan-Meier methods.

#### 8.2.4. Sensitivity and Subgroup Analysis

#### 8.2.4.1. Sensitivity Analysis

Sensitivity analysis for PFS will be performed by including both RECIST progression disease and clinical progression as PFS events. If HRG cutoff is changed during subject enrollment and stratification, the subject HRG status (High versus Low) will be redefined

using the changed HRG cutoff into new HRG high and low cohorts. Statistical analysis for PFS and key secondary endpoints will be conducted for the new HRG cohorts as a sensitivity analysis.

# 8.2.4.2. Subgroup Analysis

The subgroup analyses for PFS and OS specified in Section  and Section  will be performed for the subgroups below if data warrants:

- Age ( $\leq 65$ , > 65 yrs)
- Sex (Female, Male)
- Race (White, Non-white)
- HPV status (Postive, Negative)
- HRG subgroups (alternative cutoffs)
- Primary tumor site (oral cavity, oropharynx, hypopharynx, and larynx)
- ECOG performance status (0, 1)
- Platinum-based therapy (cisplatin carboplatin; n.b., subjects treated with both will be excluded)
- Tumor grade (well- or mod rately differentiated, poorly differentiated)
- Previous treatment (neoadjuvant chemotherapy, radiochemotherapy)
- Baseline FACT-H&N total score (≤ median, > median)

A Cox proportional hazards regression with treatment as the only covariate will be applied. Forest plots will be presented for both PFS and OS.

#### 8.3. Safety Analyses

All analyses involving safety data (extent of exposure, TEAEs, clinical laboratory results, vital signs, ECG, echocardiograms/MUGAs, physical exam, HAHA, and ECOG performance status) will be performed on the Safety Analysis Set. No inferential statistical analysis is planned for safety data. Descriptive statistics will be calculated for quantitative safety data and frequency counts and percentages will be compiled for classification of qualitative safety data. All percentages will be calculated based on the number of subjects in the Safety Analysis Set. If the number of subjects with available data does not allow for the reliable estimation of variability at a scheduled time point, no summary statistics will be presented for that time point. Unless otherwise noted, baseline values will be the last non-missing assessment collected prior to first dose of study drug.

#### **8.3.1.** Adverse Events

A treatment-emergent AE (TEAE) is defined as an adverse event that has an onset date on or after the first dose of patritumab/Placebo, or worsens in severity after the first dose of patritumab/Placebo relative to the pre-treatment state. An adverse event that occurs more than 30 days after the last dose of study medication will not be included as a TEAE, unless it is considered drug related.

Adverse events will be coded using the Medic 1 Dictionary for Regulatory Activities (MedDRA) and summarized for the number and percentage of subjects reporting treatment emergent AEs. AEs/toxicities and laboratory test results (hematology and blood chemistry) will be graded according to the NCI CTCAE, Version 4.03. The number and percentage of subjects reporting TEAEs will be tabulated by the worst CTCAE grade, system organ class, and preferred term with a breakdown by treatment group. Similarly, the number and percentage of subjects reporting treatment emergent serious adverse events (SAEs) will be tabulated, as well as TEAEs and treatment emergent SAEs considered related to patritum b, cetuximab, and cisplatin/carboplatin.

At each level of subject summarization, a subject will be counted once if he/she reports one or more occurrences of the same system organ class/preferred term/grade. For treatment-emergent (serious) adverse event toxicity tables tabulated on subject level, a subject with two or more treatment-emergent adverse events with the same preferred term will be counted only once for that term using the most severe toxicity. For a given subject, if the toxicity grade is missing for all treatment-emergent adverse events with the same preferred term, the treatment-emergent adverse events will be counted only once for that term under the "Missing" CTCAE toxicity category. In the presence of a subject who has both missing and non-missing CTCAE toxicity grades for adverse events with the same preferred term, the missing CTCAE toxicity of the adverse event will be treated as the lowest toxicity grade. In addition, a subject who reported two or more treatment-emergent adverse events with the same system organ class will be counted only once in the system organ class total, and subjects with two or more treatment-emergent adverse events in different system organ classes will be counted only once in the overall total.

A by-subject AE (including treatment emergent) data listing including, but not limited to, verbatim term, preferred term, system organ class, CTCAE grade, and relationship to study drug will be provided.

SAEs reported from tumor biopsies collected during Screening will be recorded, but not included in the primary analysis.

Deaths, other SAEs, and other significant AEs, including those leading to permanent discontinuation of subjects from patritumab, cetuximab, and cisplatin/carboplatin will be listed.

# 8.3.2. Clinical Laboratory Evaluations

For continuous laboratory parameters, values and their changes from baseline at each visit will be summarized, as well as the maximum and minimum post-treatment values, and values for the last observation on treatment. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration plus 7 days.

Repeated or unscheduled tests will not be summarized fo each scheduled visit, but will be included for summaries of maximum and minimum post-treatment values.

Clinical laboratory test results (hematology and blood chemistry) will be graded according to the NCI CTCAE, Version 4.03. Test results will also be flagged as low or high relative to the normal reference ranges. For each test, subjects will be characterized based on their worst severity grade observed during post-baseline period, based on CTCAE criteria and/or normal reference ranges. For parameters where CTCAE criteria are applicable, a shift table presenting the 2-way frequency tabulation of baseline and the worst post-baseline CTCAE grades will be provided. If absolute neutrophil or lymphocyte counts are not reported in the lab data, but percent differentials and total WBC are available, the absolut counts will be derived by the formula: differential count = 100\*differential(%)/WBC and will be reported with the same units as WBC. Derived differentials will be used for NCI-CTCAE toxicity grading, and will not be reported with a normal range. Derived values that do not meet the NCI-CTCAE criteria for grade 2 or higher toxicity will be reported as grade <1 and as being within normal range. If the result of a liver function test is below a certain threshold (e.g., AST reported as <10), then it will be reported as grade <1 and as being within normal range.

Abnormal clinical laboratory test results deemed of clinical significance or of CTCAE Grade 3 or 4 will be listed.

#### **8.3.3.** Liver Function Parameters

Subjects with elevated post-baseline ALT, AST or Total Bilirubin that fall into the following categories will be identified. Number and percentage of these subjects will be tabulated for each cohort and in total.

- AST  $\geq$  3 × Upper Limit of Normal range (ULN)
- ALT  $>= 3 \times ULN$
- AST  $\geq$  3 × ULN or ALT  $\geq$  3 × ULN

- AST  $>= 5 \times ULN$
- ALT  $>= 5 \times ULN$
- AST  $\geq$  5 × ULN or ALT  $\geq$  5 × ULN
- Total Bilirubin >= 2×ULN
- AST  $>= 3 \times ULN$  and Total Bilirubin  $>= 2 \times ULN^a$
- ALT  $\ge 3 \times ULN$  and Total Bilirubin  $\ge 2 \times ULN$
- (AST  $\ge$  3 × ULN or ALT  $\ge$  3 × ULN) and Total Bilirubin  $\ge$  2×ULN

Total Bilirubin  $\ge 2 \times \text{ULN}$  is defined as at least one case of post-dose  $\ge 2 \times \text{ULN}$  occurred between the first incidence date and 30 days after the last incidence date of ALT  $\ge 3 \times \text{ULN}$  post treatment. Same rule applies to the last 2 categories.

#### 8.3.4. Vital Signs

Values and change from baseline for vital signs, incl. ding systolic blood pressure, diastolic blood pressure, pulse, body temperature, and weight will be summarized by treatment group and scheduled time of evaluation (including end-of-treatment visit), as well as for the maximum and minimum post-treatment values, the values at the end-of-treatment visit, and values for the last observation on treatment for the Safety Analysis Set. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration plus 7 days.

Repeated or unscheduled tests will not be summarized for each scheduled visit, but will be included for summaries of maximum and minimum post-treatment values. A comprehensive listing of vital signs will be provided.

#### 8.3.5. ECG

Values and change from baseline for ECG parameters, including heart rate, PR interval, RR interval, QRS duration, QT interval, QTcB (QT / RR\*\*1/2), and QTcF (QT / RR\*\*1/3), will be summarized for each treatment group and in total at scheduled time of evaluation (including end-of-treatment visit).

In addition, the following notable ECG interval values for each parameter will be evaluated:

QTcB and QTcF:

- New >450 msec
- New >480 msec
- New >500 msec
- Increase from baseline >30 msec
- Increase from baseline >60 msec

Note that "New" implies a newly occurring ECG abnormality. It is defined as an abnormal ECG finding at post-baseline that is not present at baseline, e.g., QTc New > 480 msec implies QTc > 480 msec pose-baseline and QTc  $\leq 480 \text{ msec}$  at baseline.

A subject with multiple occurrences of a newly occurring abnormality is counted only once per abnormality.

The percentage of subjects with newly occurring qualitative ECG abnormalities is based on the total number of subjects who are at risk of developing this abnormality in the category. For each individual abnormal finding, this is defined as the number of subjects with both baseline and post baseline evaluations and a normal value at baseline.

If a QTc record is missing but the records of QT interval and RR are available then QTc should be derived using the formula above. If RR is missing but heart rate (HR) is available, QTc should be derived using the following formulae:

- QTcF = QT x  $(HR/60)^{1/3}$
- OTcB = OTx  $(HR/60)^{1/2}$

Data from ECGs will also be presented in the data listings using the Safety Analysis Set.

# 8.3.6. Dosing and Extent of Exposure

The number of IV received will be summarized for patritumab, cetuximab, and cisplatin/carboplatin, respectively, for subjects in Safety Analysis Set.

Treatment duration in weeks for patritumab and cisplatin/carboplatin is calculated as (date of the last dose – date of the first dose + 21)/7.

Cycle duration in days is calculated as (date of Day 1 of next cycle – date of Day 1 of present cycle). Cycle duration is not calculated for the last cycle. Average cycle duration will be calculated for each subject.

Treatment duration for cetuximab is calculated as Duration (weeks): (date of the last dose - date of the first dose + 7)/7

For all study treatment expect carboplatin:

- Total cumulative dose (mg/kg) is defined as the sum of all doses (mg/kg) taken by a subject.
- Total cumulative dose (mg) is calculated as total cumulative dose (mg/kg) x weight (kg).
- Dose intensity (mg/kg/cycle/dose) is calculated as 3\*(total cumulative dose(mg/kg)/(Duration(weeks)\*(number of planned doses/cycle))
- Relative dose intensity (%) is calculated as 100\*(dose intensity/(planned protocol dose)

For carboplatin:

• Total cumulative dose (mg) is defined the sum of all doses (mg) taken by a subject.

- Dose intensity is calculated as 3\*(total cumulative dose(mg)/Duration(weeks)
- Relative dose intensity (%) is calculated as 100\*(dose intensity)(planned protocol dose (mg)) where the planned protocol dose is 5x(creatinine clearance + 25) (i.e., target of 5 AUC), and the creatinine clearance is calculated using the modified Cockcroft-Gault equation (Protocol Appendix 17.1).

For the purpose of counting cycle, a subject is considered to be treated in a cycle if they receive the Day 1 dose. Treatment duration (in weeks and cycles), total cumulative dose, dose intensity, relative dose intensity, doses not completed, dose reductions, and number of IV received will be summarized using descriptive statistics, and listed for each subject in the Safety Analysis Set. Average cycle duration and number of cycles delayed, defined as time from last cycle > 21 days,) will be reported for patritumab. Subjects' dose modification will also be listed for patritumab, cetuximab, and cisplatin/carboplatin.

#### **8.3.7.** Prior and Concomitant Medications

Prior and concomitant medications will be coded using he World Health Organization (WHO) drug dictionary. Prior and concomitant medications will be summarized by treatment group, ATC2 class, and preferred term. A subject who takes one or more medications under any given ATC2 class and preferred term will be counted once for the ATC2 class and preferred term.

For the summary, medications taken prior to the first dose of study medication will be classified as prior medications, while medications taken on or after the first dosing will be classified as concomitant medications. Medications taken prior to the first dosing but with a missing stop date or with a stop date either on or after the first dosing or marked as "continuing" will also be conside ed c ncomitant medications for the summary. A listing of prior and concomitant medications by subject will be provided for the Safety Analysis Set.

# 8.3.8. Physical Examinations

A listing of physical examination data by subject for the Safety Analysis Set will be provided.

#### 8.3.9. Analysis of Other Safety Variables

HAHA results (positive as determined by titer values, if positive on screening, and detection of neutralizing antibody, if needed) will be listed to identify subjects with positive HAHA.

ECOG performance status at baseline and scheduled time of evaluation (including end of Treatment visit) will be summarized by treatment group and in total for Safety Analysis Set. A two-way frequency tabulation for baseline and each study visit will be provided for ECOG performance status.

Left ventricular ejection fraction (LVEF) will be summarized using descriptive statistics for actual values and for changes from baseline by cohort by scheduled time of evaluation including the end of treatment visit as well as for the minimum and maximum post-baseline values and for the last observation on treatment. The last observation on

treatment value is defined as the last non-missing value on or prior to end of treatment duration plus 7 days. Repeated or unscheduled tests will not be summarized for each scheduled visit, but will be included for summaries of maximum and minimum post-baseline values and the last observation on treatment.

A listing of ECOG performance status will be presented.

A listing of echocardiogram by subject for the Safety Analysis Set will be provided.

#### 8.4. Pharmacokinetic Analyses

#### **8.4.1.** Concentration Data

Concentrations below the lower limit of quantitation (BLQ) will be set to zero for the calculation of descriptive statistics. If any of the concentrations at a time point is BLQ, the geometric mean of the concentrations at this partic lar time point will not be calculated and will be presented as "NC" in the summary t bles. PK data will be listed for the pharmacokinetic analysis sets.

#### 8.4.1.1. Sparse Patritumab PK

Serum concentrations for patritumab at Cycles 1-3 and at End of Study Treatment will be listed and summarized with descriptive statistics using the PK Analysis set. Mean plasma concentration of patritumab versus time will be plotted on both linear scale and semilogarithm scale.

#### **8.4.1.2. Intensive PK**

Intensive PK refers to samples taken during Cycle 1 (Day 1 to Day 21 for patritumab, Day 1 to Day 8 for cetuximab Day 1 to Day 3 for cisplatin or carboplatin). Individual concentration profiles versus time by treatment group for each study drug will be plotted on linear and logarithmic scales. Concentrations will be summarized by treatment and nominal timepoint. Individual PK parameters will be listed and summarized by treatment.

The PK parameters, area under curve at last time point (AUC<sub>last</sub>) and  $C_{max}$  will be summarized and listed by treatment groupfor each drug using the PK Analysis set. Box plots of AUC<sub>last</sub> and  $C_{max}$  versus treatment will be presented.

# 8.4.2. Analysis of Pharmacokinetic (PK) Parameters

The intensive PK parameters, area under curve at last time point (AUC $_{last}$ ) and  $C_{max}$  will be summarized and compared for cetuximab and platinum concentration by treatment arms for the PK Analysis set. The possible drug-drug interactions between patritumab plus cetuximab or cisplatin/carboplatin, the PK of serum cetuximab and platinum concentrations will be compared with and without patritumab using an ANOVA model with treatment as factor. AUC $_{last}$  and  $C_{max}$  will be log-transformed prior to analysis. The geometric mean ratios and their two-sided 90% CIs for AUC $_{last}$  and  $C_{max}$  between the patritumab arm and the placebo arm will be calculated using the exponentiation of the differences and their CIs between treatments least square mean from the ANOVA. The ratios and their two-sided 90% CIs will be expressed relative to the placebo arm.

#### 8.4.3. Population Pharmacokinetic (PK) and Exposure Response

For all subjects, sparse samples for serum patritumab concentrations will be assessed using population PK methods. The relationship between exposure and response will be explored using population PK modeling. These analyses are outside the scope of this SAP and details of those analyses will be included in a separate document for population PK and exposure response analyses.

#### 8.5. Pharmacodynamic (PD) Parameters

Not Applicable.

# 8.6. Biomarkers Analyses

The study has baseline HRG biomarker and HPV status assessments to determine the stratification factors of HRG and HPV. Baseline HRG cutoff will be used for all specified efficacy analyses. As exploratory analyses, the HRG cutoff will be refined using graphic technique, data distribution, maximum likelihood methods, and clinical benefit of HRG high group. Selected efficacy analyses for the HRG high stratum will be performed using the refined HRG cutoff as additional exploratory analyses. Further biomarker evaluations will be summarized descriptively.

Baseline HRG values will be summarized and listed.

# 8.7. Other Variables Analyses

# 8.7.1. Patient Reported Outcomes

The FACT-H&N total score (FACT-G +disease specific subscale score), the FACT-H&N individual subscale scores (Physical Well Being (PWB), Social Well Being (SWB), Emotional Well Being (EWB), Functional Well Being (FWB)), FACT-G total score, and the FACT-H&N FHNSI sco and change from baseline will be summarized by visit and treatment group using the FACT-H&N Analysis Set.

#### For each post-baseline assessment:

- Observed range; Mean (SD) by treatment group (overall, HPV+ and HPB-) will be reported for each of the scores listed above.
- The entire Cumulative Distribution Function (CDF) of change from baseline on FACT-G, FACT-H&N FHNSI and FACT-H&N total score will be presented as a continuous plot of the change from baseline on the X-axis and the cumulative percent of subjects experiencing that change on the Y-axis for each treatment group.

Change from baseline in the FACT-H&N total score (FACT-G +disease specific subscale score), the FACT-H&N individual subscale scores, FACT-G total score, and the FACT-H&N FHNSI score, will also be evaluated using mixed longitudinal modeling for the FACT-H&N Analysis Set. The model will include treatment, time, treatment-by-time interaction, and baseline as fixed effects. The unstructured option for the REPEATED statement in PROC MIXED will be used to model the within subject covariance

structure. LS means along with 95% CIs by timepoint and LS mean differences between the control arm and patritumab arm along with two-sided 95% CIs for each timepoint will be derived.

For these analyses, PRO values obtained at the end of treatment visit or at any scheduled timepoint with fewer than 5 subjects in the placebo arm or patritumab arm will not be included.

Descriptive statistics for the actual value and change from baseline will be computed for the EQ-5D-5L health profile utilities and EQ-5D VAS by scheduled time of evaluation (including end of treatment visit) for all subjects and by treatment group using the EQ-5D Analysis Set. Results of the EQ VAS will be presented as a measure of overall self-rated health status.



# 9. CHANGES FROM THE PROTCOL SPECIFIED STATISTICAL ANALYSES

No changes have been issued.



# 10. REFERENCES

- 1. Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, et al. Toxicity and Response Criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5:649 55.
- 2. Cella DF. Manual: Functional Assessment of Cancer Therapy (FACT) Scales and Functional Assessment of HIV Infection (FAHI) Scale. Chicago: Rush-Presbyterian-St. Luke's Medical Center (1994).
- 3. D'Antonio LL, Zimmerman GJ, Cella DF, & Long, S.A. Quality of life and functional status measures in patients with head and neck cancer. *Arch Otolaryngol Head Neck Surg.* 1996; 122, 482-487.
- 4. Yount S, List M, Du H, et al. A randomized validation study comparing embedded versus extracted FACT head and neck symptom index scores. *Qual Life Res.* 2007;16:1615-26.
- 5. The EuroQol Group (1990). EuroQoL-a new facility for the measurement of health-related quality of life. *Health Policy*. 1990;16(3):199-208.
- 6. Brooks R. EuroQoL: the current state of play. *Health Policy*. 1996; 37(1):53-72.
- 7. Freidlin B, McShane LM, Polley M-Y C, et al. Randomized phase II trial designs with biomarkers. *J Clin Oncol* 2012;30:3304-3309.
- 8. Kaplan, E. L.; Meier, P. (1958). "Nonparametric estimation from incomplete observations". J. Amer. Statist. Assn. 53 (282): 457–481.
- 9. Brookmeyer, R. and Crowley, J. (1982), "A Confidence Interval for the Median Survival Time," Biometrics, 38, 29–41.
- 10. Newcombe, R. (1998). Two-Sided confidence intervals for the single proportion: comparison of seven methods. Statistics in Medicine, 17, 857-872.
- 11. Newcombe, R. (1998). Interval estimation for the difference between independent proportions: comparison of eleven methods. Statistics in Medicine, 17, 873-890

# 11. APPENDICES

#### 11.1. Data Derivation Details

#### 11.1.1. Windows Convention for Handling Partial and Missing Dates

No imputation will be performed for any dates other than adverse event onset dates and concomitant medication start and stop dates. A complete date may be necessary in order to determine if an adverse event or medication should be included in the summary/analysis (i,e., if the event is treatment emergent or the medication is prior or concomitant). The conventions specified below will be used for this purpose only. The original partial or missing dates rather than the imputed dates will be presented in the listing.

#### **Adverse Events Onset Date**

If the AE onset date is missing in which the day, month, and year are all unknown or only the day is known, the AE onset date is set to the date of first dose of study medication.

For the partial AE onset date,

- If the year is present and the month and day are missing or the year and day are present and the month is m ssing
  - If year = year of first dose then set month and day to month and day of first dose
  - If year < year of first dose, then set month and day to December 31<sup>st</sup>.
  - If year > year of first dose, then set month and day to January 1<sup>st</sup>.
- If the month and year are present and the day is missing:
  - If year=year of first dose and if month = month of first dose then set day to day of first dose date if month < month of first dose then set day to last day of month if month > month of first dose then set day to 1<sup>st</sup> day of month If year < year of first dose then set day to last day of month If year > year of first dose then set day to 1<sup>st</sup> day of month
- If the imputed AE onset date is after AE stop date, then set the onset date to the AE stop date.

#### **Prior and Concomitant Medications Date**

If the start date of medication is completely missing in which the day, month, and year are all unknown or only the day is known, then the start date will not be imputed.

For the partial start date of medication,

- If the year is present and the month and day are missing or the year and day are present and the month is missing, set month and day to January 1.
- If the year and month are present and the day is missing, set day to 1<sup>st</sup> day of month.
- If the imputed start date of medication is after the non-imputed end date of medication, then the start date will be set to the end date of medication.

If the end date of medication is completely missing which the day, month, and year are all unknown or only the day is known, then the end date will not be imputed.

For the partial end date of medication,

- If the year is present and the month and day are missing or the year and day are present and the month is missing, set month and day to December 31.
- If the year and month are present and the day is missing, set day to last day of the month.

# **Incomplete Tumor Assessment Dates**

All dates for tumor assessment must be completed with day, month and year.

- If one or more measurement dates (e.g. X-ray, CT-scan for target and non-target tumor lesions) are incomplete but other measurement dates are available, this/these incomplete date(s) are not considered for calculation of the assessment date.
- If all measurement dates have no day recorded, the 1<sup>st</sup> of the month is used.
- If the month is not completed, for any of the assessments, the respective assessment will be onsidered to be at the midpoint of previous and following assessment dates.

#### **Incomplete Dates for Last Contact or Death**

All dates are expected to be completed with day, month, and year.

If the day/month is missing, the 1<sup>st</sup> of the month/year will be used for incomplete death dates or dates of last contact.
SAP U31287-A-U203 Version 1.0, 29 November 2016

# 11.2. Interim Analysis Statistical Analysis Plan

Safety data and efficacy data will be prepared for the purpose of DMC reviews, and the frequency and extent of such data reviews will follow the DMC charter for Study U31287-A-U203. In general, the statistical methodology and TLF shells in the SAP will be a framework to generate outputs for DMC reviews. The independent Data Analysis Group (DAG) will perform the analysis. Operating details of the DAG are included in the DMC charter.



SAP U31287-A-U203 Version 1.0, 29 November 2016

### 11.3. Formula for Wilson Method

## Wilson Method

Use the following formula to compute a  $(1-\alpha)$ % confidence interval for a single proportion using the Wilson method with continuity correction:

$$L = \frac{\hat{p}_i + \frac{z^2}{2n_i} - \frac{1}{2n_i} - z\sqrt{\frac{\hat{p}_i[n_i(1 - \hat{p}_i) + 1]}{n_i^2} + \frac{z^2 - 2 - 1/n_i}{4n_i^2}}}{1 + \frac{z^2}{n_i}}$$

$$U = \frac{\hat{p}_i + \frac{z^2}{2n_i} + \frac{1}{2n_i} + z\sqrt{\frac{\hat{p}_i[n_i(1 - \hat{p}_i) - 1]}{n_i^2} + \frac{z^2 + 2 - 1/n_i}{4n_i^2}}}{1 + \frac{z^2}{n_i}}$$

where  $\hat{p}_i$  denotes the sample proportion for group i and n the group sample size. All statistical constants will be computed using appropriate SAS functions. Note: if  $\hat{p}_i$ =0, L must be taken as 0; if  $\hat{p}_i$ =1, U is then 1. In case L is calculated to be less than 0, set L to 0; and similarly set U to 1 if U is calculated to be larger than 1.

Confidence limits for the difference in ORR between each of the U3-1287 (AMG888) groups and placebo based on Wilson (Newcombe) score will use the method below.

Denote the lower and upper Wilson score (with continuity correction) confidence limits for  $p_1$  as  $L_1$  and  $U_1$  and the lower and upper confidence limits for  $p_2$  as  $L_2$  and  $U_2$  (where L and U are defined above). The Wilson score (with continuity correction) confidence limits for the proportion diff ence  $(d=p_1-p_2)$  are computed as

$$d_{L} = (\hat{p}_{1} - \hat{p}_{2}) - z\sqrt{L_{1}(1 - L_{1})/n_{1} + U_{2}(1 - U_{2})/n_{2}}$$

$$d_{U} = (\hat{p}_{1} - \hat{p}_{2}) + z\sqrt{U_{1}(1 - U_{1})/n_{1} + L_{2}(1 - L_{2})/n_{2}}$$

SAP U31287-A-U203 Version 1.0, 29 November 2016

## 11.4. Mock-up Tables and Listings

The date on which the first dose of study medication (including placebo) is administered is considered as Day 1 of the study. For events occurring on or after the start of treatment, study day is calculated as the event date minus the date of first administration of study medication plus 1 day. For events occurring before the start of treatment, study day is calculated as the event date minus the date of first administration of study medication.

Raw measurements will be reported to the number of significant digits as captured electronically or on the CRF. The mean and median will be displayed to one decimal place beyond the number of decimal places the original parameter is presented, and the measure of variability (e.g., standard deviation) will be displayed to two decimal places beyond the number of decimal places the original parameter is presented. Minimums and maximums will be reported to the same number of significant digits as the parameter. Calculated percentages will be reported with 1 decimal place. When count data are presented as category frequencies and corresponding percentages, the percent will be suppressed when the count is zero. Show a 'Missing row' after the last category if there are missing observations for the variable.

P-values will be reported to 4 decimal places (SAS format pvalue6.4). Values less than 0.0001 will be displayed as <0.0001. Values greater than 0.9995 will be displayed as 1.0000. Unless otherwise indicated, 1-sided p-values are presented in the tables.

All tables will summarize data for the overall study population and by the high and low HRG expression strata. For disposition tables and safety tables the order will be overall, high, and low. For efficacy tables the order will be high, low, and overall.

Listings will be presented for each part and sorted by subject ID. When available, listings will also be sorted by study day.

Unless otherwise indicated continuous variables will be summarized using the following descriptive statistics: the number of subjects (n), mean, standard deviation, median, minimum, and maximum. The frequency and percentage of observed levels will be reported for categorical measures. Percentages will be based on the number of subjects in the relevant analysis set. All statistical analyses will be performed in SAS Version 9.1 or higher

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.1: Subject Disposition
All Screened Analysis Set

**HRG High** 

| HRG High | | | |
|---|---|---|---|
| | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| Subject Accounting | (N=xxx) | (N=xxx) | (N=xxx) |
| Screened | | | |
| Screened, But Not Randomized | | <b>A</b> | xxx [a] |
| Randomized | | | |
| Randomized but Not Dosed | xxx (xx.x) | xxx ( x.x) | xxx (xx.x) |
| Analysis Set | | ~10 | |
| Full Analysis Set (Intent to Treat Set)[b] | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Safety Analysis Set | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Per-Protocol Analysis Set | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| PK Analysis Set | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| FACT-H&N Analysis Set | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| EQ-5D Analysis Set | xxx (xxx ) | xxx (xxx.x) | xxx (xxx.x) |
| _ u =, | | | ` ' |
| Treatment Status | | | |
| Ongoing on the Study Treatment | xx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Discontinued from Study Treatment | xxx xx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Primary Reason for Discontinuation from | | | |
| Study Treatment Adverse Event | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Progressive Disease per RECIST | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Clinical Progression | xxx (xxx.x) | XXX (XXX.X) | xxx (xxx.x) |
| Lost to Follow-up | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Death | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Protocol Violation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Withdrawal by subject | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Study Terminated by Sponsor | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Other | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Notes: Percentages are based on the number of subjects in the Full Analysis Set.

Source Data: adam.adsl; Listing 16.2.1.1

<sup>[</sup>a] Subjects who had signed ICF and were screened but not randomized are not included in the total number of Full Analysis Set.

<sup>[</sup>b] The full analysis set (FAS) will be based on the intent-to-treat principle and will include all subjects randomized into the study.

<sup>[</sup>c] On-study Death is defined as death occurred on or after first dose date till 21 days after last dose date of any study drug.

Protocol U31278-A-U203

Page x of y rogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.1: Subject Disposition All Screened Analysis Set

HRG High

| TINO TIIgii | Patritumab + cetuximab + cisplatin or carboplatin | Placebo + cetuximab + cisplatin or carboplatin | Total |
|---|---|---|---|
| Subject Accounting | (N=xxx) | (N=xxx) | (N=xxx) |
| Extension Treatment Status | | | |
| Ongoing on the Study Treatment | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Discontinued from Study Treatment | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Primary Reason for Discontinuation from Study | , | | , |
| Treatment | | | |
| Adverse Event | xxx (xxx.x) | xxx (xxx ) | xxx (xxx.x) |
| Clinical Progression | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Lost to Follow-up | xxx (xxx.x) | xxx (xxx x) | xxx (xxx.x) |
| Death | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Protocol Violation | xxx (xxx.x) | x (xxx.x) | xxx (xxx.x) |
| Withdrawal by subject | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Study Terminated by Sponsor | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Progressive Disease per RECIST | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Other | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| On-Study Death [c] | xxx (xxx.x | xxx (xxx.x) | xxx (xxx.x) |
| Primary cause of On-Study Death | | | |
| Adverse Event | xx (x x x) | xxx (xxx.x) | xxx (xxx.x) |
| Disease Progression | xx (xxx x) | xxx (xxx.x) | xxx (xxx.x) |
| Unknown | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Other | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Notes: Percentages are based on the number of subjects in the Full Analysis Set.

Source Data: adam.adsl; Listing 16.2.1.1

<sup>[</sup>a]: Subjects who had signed ICF and were screened but not randomized are not included in the total number of Full Analysis Set.

<sup>[</sup>b] The full analysis set (FAS) will be based on the intent-to-treat principle and will comprise all subjects randomized into the study.

<sup>[</sup>c] On-study Death is defined as death occurred on or after first dose date till 21 days after last dose date of any study drug.

<run date time>

Page x of y

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

HRG High

| eg | Patritumab + cetuximab + | Placebo + cetuximab + | Total |
|---|---|---|---|
| | cisplatin or carboplatin (N=xxx) | cisplatin or carboplatin<br>(N=xxx) | Total<br>(N=xxx) |
| Age (yrs) [a] | (** 700*) | (11 7551) | (11 7001) |
| n | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX |
| Maximum | xx | xx | XX |
| <=65 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >65 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gender | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <=65 | | | |
| >65 | | | |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <=65 | | | |
| >65 | | | |
| Race | | | |
| White | xx (xx. %) | xx (xx.x%) | xx (xx.x%) |
| Black or African American | (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asian | xx ( x.x%) | xx (xx.x%) | xx (xx.x%) |
| American Indian or Alaskan Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Native Hawaiian/Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other/Specify | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other/opedity | ^^ (^^.^ /0) | ^^ (^^.^/0) | ^^ (^^.^ /0) |

Notes: Denominator for percentages is the number of subjects in the Full Analysis Set.

The baseline value is defined as the last non-missing value before initial administration of study treatment.

Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16.2.4.4.3, 16.2.4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

<sup>[</sup>a] Age in years is calculated using the informed consent date and the birth date.

Protocol U31278-A-U203

Page x of y

cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

HRG High

| | Patritumab + cetuximab + | Placebo + cetuximab + | T-4-1 |
|---|---|---|---|
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Height (cm) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX |
| Maximum | XX | XX | XX |
| Veight (kg) | | , 1 | |
| n | XX | XX | XX |
| Mean | XX.X | x x | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Minimum | xx | XX | xx |
| Maximum | XX | XX | xx |
| listology | | | |
| Squamous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (x x%) | xx (xx.x%) | xx (xx.x%) |
| Curo | /ai (ai 2/3) | 70t (70ti)*/*/ | 70t (70ti7t70) |
| Histologic Grade | | | |
| Well Differentiated | xx ( x.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderately Differentiated | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Poorly Differentiated | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Undifferentiated | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Unknown | | , , | |
| OHNHOWH | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: Denominator for percentages is the number of subjects in the Full Analysis Set.

Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16.2.4.4.3, 16.2.4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

The baseline value is defined as the last non-missing value before initial administration of study treatment.

<sup>[</sup>a] Age in years is calculated using the informed consent date and the birth date.

Protocol U31278-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

**HRG High** 

| HRG High | | | |
|---|---|---|---|
| | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Tumor Staging at Study Entry | | | |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <u> </u> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| IIA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| IIB | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| III<br>IVA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| IVB | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| IVC | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Outer | XX (XX.X70) | XX (XX.X/0) | XX (XX.X70) |
| Time from Initial Diagnosis of SCCHN to Study | | .10 | |
| reatment (month) [b] | | | |
| n<br>Maar | XX | XX | XX |
| Mean<br>SD | XX.X | XX.X | XX.X |
| | XX.XX | xx.xx | XX.XX |
| Median | XX.X | xx.x | XX.X |
| Minimum | xx | xx | XX |
| Maximum | xx | xx | XX |
| <6 months | xx xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 6-12 months | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| >12 months | xx (xx.x% | xx (xx.x%) | xx (xx.x%) |
| Cancer Type | <b>Y</b> | | |
| Oral Cavity | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Oropharynx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypopharynx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Larynx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: Denominator for percentages is the number of subjects in the Full Analysis Set.

The baseline value is defined as the last non-missing value before initial administration of study treatment.

<sup>[</sup>a] Age in years is calculated using the informed consent date and the birth date.

<sup>[</sup>b] For the partial Initial Diagnosis of SCCHN date, if the month and year are present and the day is missing, then set day to the 1st day of month. Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16.2.4.4.3, 16.2.4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

Protocol U31278-A-U203

Page x of y rogname <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

**HRG High** 

| | Patritumab + cetuximab + | Placebo + cetuximab + | |
|---|---|---|---|
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Cigarette Use | | | |
| Current | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Former | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Never | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Duration of Cigarette (years) | | | |
| n | XX | xx | XX |
| Mean | XX.X | xx.x | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX |
| Maximum | XX | xx | XX |
| Cigar Use | | | |
| Current | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Former | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Never | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Duration of Cigar (years) | | | |
| n , | X | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Minimum | xx | XX | XX |
| Maximum | XX | xx | XX |

Notes: Denominator for percentages is the number of subjects in the Full Analysis Set.

The baseline value is defined as the last non-missing value before initial administration of study treatment.

<sup>[</sup>a] Age in years is calculated using the informed consent date and the birth date.

<sup>[</sup>b] For the partial Initial Diagnosis of SCCHN date, if the month and year are present and the day is missing, then set day to the 1st day of month. Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16.2.4.4.3, 16.2.4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

Protocol U31278-A-U203

Page x of y rogname <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

**HRG High** 

| | Patritumab + cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | Placebo + cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Prior Systemic Cancer Therapy | (************************************** | (************************************** | (********* |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Best Response to Prior Systemic Cancer<br>Therapy | | | |
| CR | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PR | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SD | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PD | xx (xx.x%) | xx ( x.x%) | xx (xx.x%) |
| Not Applicable | xx (xx.x%) | xx (xx %) | xx (xx.x%) |
| Unknown | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Prior Radiation Therapy | . ( | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline ECOG Performance Status | | | |
| 0 - Fully Active | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 - Restricted in Physically Strenuous | xx ( x x%) | xx (xx.x%) | xx (xx.x%) |
| Activity | | ( 173) | () |
| 2 - Ambulatory and Capable of All Self- | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| are | | , | , , |
| 3 – Capable of Only Limited Self Care | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 – Completely Disabled | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: Denominator for percentages is the number of subjects in the Safety Analysis Set.

The baseline value is defined as the last non-missing value before initial administration of study treatment.

<sup>[</sup>a] Age in years is calculated using the informed consent date and the birth date.

Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16.2.4.4.3, 16.2.4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

Protocol U31278-A-U203

Page x of y

<run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.2.1: Demographic and Baseline Characteristics Full Analysis Set

| IRG High | | • | |
|---|---|---|---|
| | Patritumab + cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | Total<br>(N=xxx) |
| Baseline 12-Lead ECG | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Not Clinically Significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Clinically Significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Heregulin (HRG) | | | |
| n | XX | XX | XX |
| Mean | XX.X | xx x | XX.X |
| SD | XX.XX | XX.X | XX.XX |
| Median | XX.X | xx.x | XX.X |
| Minimum | XX | xx | XX |
| Maximum | XX | xx | XX |
| | A/ | | |

Notes: Denominator for percentages is the number of subjects in the Safety Analysis Set

Source Data: adam.adsl; Listing 16.2.4.1, 16.2.4.4.1, 16.2.4.4.2, 16 2 4.4.3, 16.2 4.4.4, 16.2.4.6, 16.2.8.3.2, 16.2.8.3.4, 16.2.8.4.2.

Programming Note: continue for HRG Low and Overall on the next page

Programming note: Present 'Missing' as a category if here is at least one subject in a row.

Using the table shell of 15.1.2.1 for following 3 tables:

Table 15.1.2.2: Demographic and Baseline Characteristics Per Protocol Analysis Set

Change first line footnote to: Denominator for percentages is the number of subjects in Per Protocol Analysis Set

Table 15.1.2.3: Demographic and Baseline Characteristics Safety Analysis Set

Change first line footnote to: Denominator for percentages is the number of subjects in Safety Analysis Set

The baseline value is defined as the last non-missing value before in all administration of study treatment.

<sup>[</sup>a] Age in years is calculated using the informed consent date a d the irth date.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYYY)

Table 15.1.3: Study Drug Exposure Safety Analysis Set

HRG High

| | | Patritumab + | cetuximab + | Placebo + cetuximab + | | | | |
|---|---|---|---|---|---|---|---|---|
| | cisplatin or carboplatin | | | | | cisplatin or carboplatin | | |
| | Patritumab | Cetuximab | Carboplatin | Cisplatin | Placebo | Cetuximab | Carboplatin | Cisplatin |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| Treatment Duration (weeks) | , | , | , | , | • | , | , | , , |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.X | XX.X | XX.X | XX.X | XX X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | | | 1 | | |
| Treatment Duration (cycles) | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | xx | XX | XX | XX | XX |
| Number of IVs Received per Subject | | | | | | | | |
| n | XX | XX | X | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | X.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.X | XX.X | X X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX |
| Number of Cubicate with a F IV | ( | ( | ( | ( | ( | (0( ) | (0/ ) | ( |
| Number of Subjects with <5 IVs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects with 5 - <10 IVs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects with 10 - <15 IVs | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) |
| Number of Subjects with 15 - <20 IVs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects with >20 IVs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: For Patritumab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

Source Data: adam.adex, adam.adda; Listing 16.2.5.1.1, 16.2.5.1.3. Programming Note: continue for HRG Low and Overall on the next page

For Cetuximab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 7)/7. Treatment duration (in cycles)

is calculated as (date of the last dose – date of the first dose + 7)/21.

For Carboplatin or Cisplatin, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the list dose + 21)/21.

<sup>[</sup>a] Refer to SAP Section 8.3.6 for definitions for Cumulative Dose Received per Subject, Dose Intensity, and Relative Dose Intensity, and Cycle Duration...

Protocol U31278-A-U203

Page x of y

<run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.3: Study Drug Exposure Safety Analysis Set

HRG High

| | | Placebo + cetuximab + cisplatin or carboplatin | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | cisplatin or carboplatin | | | | | | | |
| | Patritumab<br>(N=xxx) | Cetuximab<br>(N=xxx) | Carboplatin (N=xxx) | Cisplatin (N=xxx) | Placebo<br>(N=xxx) | Cetuximab<br>(N=xxx) | Carboplatin (N=xxx) | Cisplatin (N=xxx) |
| Cumulative Dose Received per Subject | | | | | | | | |
| (mg) [a] | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | xx x | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX XX | XX.XXX | XX.XXX | XX.XXX |
| Minimum | XX.X | XX.X | XX.X | XX.X | X.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX | XX | XX | XX | XX |
| Maximum | xx | XX | XX | XX | xx | XX | XX | XX |
| Cumulative Dose Received per Subject (mg/kg) | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | X | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX | XX | Xx |
| Dose Intensity (mg/kg/cycle/dose) [a] | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX |

Notes: For Patritumab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

For Cetuximab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 7)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 7)/21.

For Carboplatin or Cisplatin, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

[a] Refer to SAP Section 8.3.6 for definitions for Cumulative Dose Received per Subject, Dose Intensity, and Relative Dose Intensity, and Cycle Duration..

Source Data: adam.adex; Listing 16.2.5.1.1, 16.2.5.1.2, 16.2.5.1.3. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.3: Study Drug Exposure Safety Analysis Set

Overall

| Patritumab (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) Placebo (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) Placebo (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) Placebo (N=xxxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) Placebo (N=xxxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Placebo + cetuximab + | | | | | cetuximab + | | | |
|---|---|---|---|---|---|---|---|---|---|
| N=xxx | atin | cisplatin or carboplatin | | | | carboplatin | | | |
| N=xxx | oplatin Cisplatin | Carboplatin | Cetuximab | Placebo | Cisplatin | Carboplatin | Cetuximab | Patritumab | |
| n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx </th <th></th> <th>(N=xxx)</th> <th>(N=xxx)</th> <th>(N=xxx)</th> <th>(N=xxx)</th> <th></th> <th>(N=xxx)</th> <th>(N=xxx)</th> <th></th> | | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | | (N=xxx) | (N=xxx) | |
| Mean xx.xx | | | | | | | | | Relative Dose Intensity (%) [a] |
| SD xx.xxx xx.xxx xx.xxx xx.xxx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx <t< td=""><td>XX XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td></td></t<> | XX XX | XX | XX | XX | XX | XX | XX | XX | |
| Minimum XX.X | XX.XX XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | Mean |
| Median Maximum XX | .XXX XX.XXX | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | SD |
| Maximum xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx <t< td=""><td>x.x xx.x</td><td>XX.X</td><td>XX.X</td><td>xx x</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>Minimum</td></t<> | x.x xx.x | XX.X | XX.X | xx x | XX.X | XX.X | XX.X | XX.X | Minimum |
| Cycle Duration (Days) n xx | XX XX | XX | XX | XX | XX | XX | XX | XX | Median |
| n XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX </td <td>XX XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>Maximum</td> | XX XX | XX | XX | XX | XX | XX | XX | XX | Maximum |
| n XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX </td <td></td> <td></td> <td></td> <td></td> <td>. (</td> <td></td> <td></td> <td></td> <td>Ovela Devetia (Deve</td> | | | | | . ( | | | | Ovela Devetia (Deve |
| Mean xx.xx xx.x xx.x< | | | | | | | | | |
| SD xx.xxx xx.xx | | XX | | | | | | | |
| Minimum xx.x | | XX.XX | | | | | | | |
| Median Maximum XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <th< td=""><td></td><td>XX.XXX</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | | XX.XXX | | | | | | | |
| Maximum xx Cycles Delayed n xx | | XX.X | | | | | | | |
| Cycles Delayed n xx | | XX | | | | | | | |
| n xx xx xx xx xx xx xx | xx Xx | XX | XX | XX | XX | XX | XX | XX | Maximum |
| n xx xx xx xx xx xx xx | | | | | | | | | Cycles Delayed |
| | xx xx | XX | XX | XX | XX | XX | XX | XX | |
| | | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | Mean |
| | | XX.XXX | | | | | | | |
| | | XX.X | | | | | | | Minimum |
| Median xx x xx xx xx xx xx | | XX | | | | | | | |
| Maximum xx xx xx xx xx xx | | XX | | | | | | | |

Notes: For Patritumab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

For Cetuximab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 7)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 7)/21.

For Carboplatin or Cisplatin, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

[a] Refer to SAP Section 8.3.6 for definitions for Cumulative Dose Received per Subject, Dose Intensity, and Relative Dose Intensity, and Cycle Duration..

Source Data: adam.adex; Listing 16.2.5.1.1, 16.2.5.1.2, 16.2.5.1.3.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.3: Study Drug Exposure Safety Analysis Set

### Overall

| Patritumab | | | Cisplatin | Placebo | | | Cisplatin |
|---|---|---|---|---|---|---|---|
| (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX | XX | XX | XX | XX | XX | XX | XX |
| XX.XX | XX.XX | XX.XX | XX.XX | XX X | XX.XX | XX.XX | XX.XX |
| XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |
| XX | XX | XX | X | XX | XX | XX | XX |
| XX | xx | xx | XX | XX | XX | xx | Xx |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx ( x.x%′ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.xx)<br>xx.xx<br>xx.xx<br>xx.x<br>xx<br>xx<br>xx<br>xx<br>xx<br>xx | cisplatin or Patritumab (N=xxx) Cetuximab (N=xxx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.xx xx.xx xx (xx.xx xx.xx xx (xx.xx xx xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xxx) (N=xxx) (N=xxx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx xx xx xx xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx xx xx xx | Cisplatin or carboplatin Patritumab (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | Cisplatin or carboplatin Patritumab (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin (N=xxx) Placebo (N=xxx) xx (xx.x%) xx (xx.x%) | Cisplatin or carboplatin Cisplatin or cisplatin or cisplatin or cisplatin or cisplatin Patritumab (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cisplatin Placebo (N=xxx) Cetuximab (N=xxx) xx (xx.x%) xx | Cisplatin or carboplatin Cisplatin or carboplatin Patritumab (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) Cetuximab (N=xxx) Carboplatin (N=xxx) xx (xx.x%) xx (xx.x%) |

Notes: For Patritumab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/2.

For Cetuximab, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 7)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first do + 7)/21.

For Carboplatin or Cisplatin, treatment duration (in weeks) is calculated as (date of the last dose – date of the first dose + 21)/7. Treatment duration (in cycles) is calculated as (date of the last dose – date of the first dose + 21)/21.

[a] Refer to SAP Section 8.3.6 for definitions for Cumulative Dose Received per Subject, Dose Intensity, and Relative Dose Intensity, and Cycle Duration...

Source Data: adam.adex; Listing 16.2.5.1.1, 16.2.5.1.2, 16.2.5.1.3.

Protocol U31278-A-U203

Page x of y

cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.1.4.1: Prior Medications by ATC Class and Preferred Term Safety Analysis Set

**HRG High** 

| | Patritumab + cetuximab + cisplatin or carboplatin | Placebo + cetuximab + cisplatin or carboplatin | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Subjects with any Prior Medications | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC 2 Class x | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx ( x.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | x (xx.x) | xx (xx.x) |
| Preferred Term n | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC 2 Class y | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term n | xx (xx x) | xx (xx.x) | xx (xx.x) |
| ATC 2 Class z | xx ( x.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term n | x (xx.x) | xx (xx.x) | xx (xx.x) |

Notes: Denominator for percentages is the number of subjects in the Safety Analysis Set.

Medications taken prior to the first dose of study medication will be classified as prior medications.

Subjects may have more than one medication per ATC classification and preferred term. At each level of subject summarization, a subject was counted once if he/she reported one or more medications.

Medications were coded using the WHO Drug Dictionary (Version XXX).

Source Data: adam.adcm; Listing 16.2.4.5

Table 15.1.4.2: Concomitant Medications by ATC Class and Preferred Term Safety Analysis Set

Programming note: Replace the second sentence with "Medications taken on or after the first dose of study medication will be classified as concomitant medications".

First row should state 'Subjects with any Concomitant Medications'




Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.1.1: Analysis of Progression Free Survival (PFS) Full Analysis Set

**HRG High** 

| HRG High | | | |
|---|---|---|---|
| Statistics | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | |
| | (N=xxx) | (N=xxx) | |
| Subject (%) with Events | xx (xx.x%) | xx (xx.x%) | |
| Subject (%) without Events (Censored) | xx (xx.x%) | xx (xx.x%) | |
| Median PFS (months) [a] | xx.x | XX.X | |
| 95% CI | [xx.x; xx.x] | [xx x; xx.x] | |
| Disers the second second selection in | | | • |
| Stratified Log-rank p-value [b] | | | 0.xxxx |
| og-rank p-value (Unstratified) <sup>[c]</sup> | | | 0.xxxx |
| Stratified Cox Regression Analysis [D] | | | |
| Hazard Ratio (relative to Placebo) | | | X.XXXX |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one<br>Instratified Cox Regression Analysis <sup>[c]</sup> | | | 0.xxxx |
| Hazard Ratio (relative to Placebo) | | | x.xxxx |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one | NUY | | 0.xxxx |
| PFS Rate at 3 Months [d] | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 6 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 9 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 12 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |

Notes: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first. See the SAP for the handling of censored cases.

- [a] Median PFS is from Kaplan-Meier analysis. CI for median was computed using the Brookmeyer-Crowley method.
- [b] Stratified log-rank test adjusted for stratification factors: HRG (high vs low; overall only) and HPV (positive vs other) at randomization.
- [c] Log-rank test did not adjust for stratification factors.
- [d] Estimate and CI for PFS rate at the specified timepoint are from Kaplan-Meier analysis.

Source Data: adam.adtte; Listing 16.2.6.1

Programming note: If insufficient #'s of subject progress then certain proportions are not estimable and the estimate and corresponding confidence interval will be omitted.

Use table shell of 15.2.1.1 to generate following tables:

Table 15.2.1.2: Analysis of Progression Free Survival (PFS)
Per Protocol Analysis Set



Protocol U31278-A-U203

Page x of y rogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.1.3: Subgroup Analysis of Progression Free Survival (PFS)
Full Analysis Set

| Overall | | | |
|---|---|---|---|
| Subgroup/<br>Statistic | Patritumab + cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | |
| Age | | | |
| <65 | VV V | | |
| Median PFS (months) <sup>[a]</sup><br>95% CI | xx.x<br>[xx.x; xx.x] | xx.x<br>[xx.x; xx.x] | |
| Hazard Ratio (relative to Placebo) <sup>[b]</sup><br>95% CI for Hazard Ratio<br>p-value for hazard ratio equal to one | [^^.^, ^^.^] | [[, ,, | x.xxxx<br>[x.xxxx, x.xxxx]<br>0.xxxx |
| >=65 | <b>~</b> | | |
| Median PFS (months) [a] | XX.X | XX.X | |
| 95% CI<br>Hazard Ratio (relative to Placebo) <sup>lbj</sup> | [xx.x; xx.x] | [xx.x; xx.x] | X.XXXX |
| 95% CI for Hazard Ratio<br>p-value for hazard ratio equal to one | 40 | | [x.xxxx, x.xxxx]<br>0.xxxx |
| Sex | | | |
| Female | | | |
| Median PFS (months) [a] | XX.X | XX.X | |
| 95% CI | x.x; xx.x] | [xx.x; xx.x] | |
| Hazard Ratio (relative to Placebo) <sup>[b]</sup> | | | X.XXXX |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one | | | 0.xxxx |
| Male<br>Median PFS (months) <sup>[a]</sup> | XX.X | XX.X | |
| 95% CI | [xx.x; xx.x] | [XX.X; XX.X] | |
| Hazard Ratio (relative to Placebo) <sup>[b]</sup> | [AAA, AAA] | [MAN, MAN] | x.xxxx |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one | | | 0.xxxx |

Notes: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first. See the SAP for the handling of censored cases.

Source Data: adam.adtte; Listing 16.2.6.1

Programming note: Continue for subgroups in Section 8.2.4.2 of SAP.

<sup>[</sup>a] Median PFS is from Kaplan-Meier analysis. CI for median was computed using the Brookmeyer-Crowley method.

<sup>[</sup>b] Log-rank test did not adjust for stratification factors.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.1.4: Analysis of Progression Free Survival (PFS) for Different HRG Cutoffs
Full Analysis Set

HRG Cutoff: HRG >= XX.XX

| HRG Cutoff: HRG >= XX.XX | | | |
|---|---|---|---|
| Statistics | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | |
| | (N=xxx) | (N=xxx) | |
| Subject (%) with Events | xx (xx.x%) | xx (xx.x%) | |
| Subject (%) without Events (Censored) | xx (xx.x%) | xx (xx.x%) | |
| Median PFS (months) <sup>[a]</sup> | xx.x | XX.X | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| Stratified Cox Regression Analysis <sup>[b]</sup> | | | |
| Hazard Ratio (relative to Placebo) | | | x.xxxx |
| 95% CI for Hazard Ratio | × 1 | | [x.xxxx, x.xxxx] |
| 80% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| Instratified Cox Regression Analysis <sup>[c]</sup> | | | |
| Hazard Ratio (relative to Placebo) | | | X.XXXX |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| 80% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| PFS Rate at 3 Months <sup>[d]</sup> | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 6 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 9 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| PFS Rate at 12 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |

Notes: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first. See the SAP for the handling of censored cases.

- [a] Median PFS is from Kaplan-Meier analysis. CI for median was computed using the Brookmeyer-Crowley method.
- [b] Stratified Cox PH regression adjusted for stratification factors: HPV (positive vs other) and HRG (high vs. low, only for the FAS) at randomization.
- [c] Cox PH regression did not adjust for stratification factors.
- [d] Estimate and CI for PFS rate at the specified timepoint are from Kaplan-Meier analysis.

Programming note: If insufficient #'s of subject progress then certain proportions are not estimable and the estimate and corresponding confidence interval will be omitted.

Programming Note: continue for different HRG Cutoff

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYYY)
Table 15.2.2.1: Analysis of Overall Survival (OS)

Full Analysis Set

HRG High

| IRG High | | | |
|---|---|---|---|
| Statistics | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | |
| | (N=xxx) | (N=xxx) | |
| Subject (%) with Events | xx (xx.x%) | xx (xx.x%) | |
| Subject (%) without Events (Censored) | xx (xx.x%) | xx (xx.x%) | |
| Median PFS (months) [a] | XX.X | XX.X | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| stratified Log-rank p-value <sup>[b]</sup> | | | 0.xxxx |
| og-rank p-value (Unstratified) [c] | 4 | | 0.xxxx |
| Stratified Cox Regression Analysis <sup>[b]</sup> | | | |
| Hazard Ratio (relative to Placebo) | | | x.xxxx |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one | | | 0.xxxx |
| Instratified Cox Regression Analysis <sup>[c]</sup><br>Hazard Ratio (relative to Placebo) | | | x.xxxx |
| 95% CI for Hazard Ratio | | | [x.xxxx, x.xxxx] |
| p-value for hazard ratio equal to one | | | 0.xxxx |
| FS Rate at 3 Months [d] | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [XX.X; XX.X] | |
| PFS Rate at 6 Months | XX.X% | XX.X% | |
| 95% CI | [xx.x; xx.x] | [XX.X; XX.X] | |
| PFS Rate at 9 Months | XX.X% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |
| FS Rate at 12 Months | xx.x% | xx.x% | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | |

Notes: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first. See the SAP for the handling of censored cases.

- [a] OS is defined as the time from the date of randomization to death due to any cause.
- [b] Stratified log-rank test adjusted for stratification factors: HPV (positive vs other) at randomization.
- [c] Log-rank test did not adjust for stratification factors.
- [d] Estimate and CI for OS rate at the specified timepoint are from Kaplan-Meier analysis.

Source Data: adam.adtte; Listing 16.2.6.1

Daiichi Sankyo Pharma Development Protocol U31278-A-U203

Page x of y

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Use table shell of 15.2.2.1 to generate following tables:

Table 15.2.2.2 Analysis of Overall Survival (OS)
Per Protocol Analysis Set

Change the first line of footnote to: OS is defined as the time from the date of randomization to death due to any cause. Change the PFS in table and footnotes to OS.

Use table shell of 15.2.1.3 to generate following tables:

Table 15.2.1.3: Subgroup Analysis of Overall Surviva (OS) Full Analysis Set

Change the first line of footnote to: OS is defined as the time from the date of randomization to death due to any cause. Change the PFS in table and footnotes to OS.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.2.3: Analysis of Overall Survival (OS) for Different HRG Cutoffs Full Analysis Set

HRG Cutoff: HRG <= XX.XX

| Statistics | Patritumab + cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | |
|---|---|---|---|
| Subject (%) with Events<br>Subject (%) without Events (Censored) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | |
| Median PFS (months) [a]<br>95% CI | xx.x<br>[xx.x; xx.x] | xx.x<br>[xx x; xx.x] | |
| Stratified Cox Regression Analysis <sup>[D]</sup> Hazard Ratio (relative to Placebo) 95% CI for Hazard Ratio 80% CI for Hazard Ratio Unstratified Cox Regression Analysis <sup>[C]</sup> Hazard Ratio (relative to Placebo) 95% CI for Hazard Ratio 80% CI for Hazard Ratio | | | x.xxxx [x.xxxx, x.xxxx] [x.xxxx, x.xxxx] x.xxxx [x.xxxx, x.xxxx] [x.xxxx, x.xxxx] |
| PFS Rate at 3 Months <sup>[d]</sup> 95% CI PFS Rate at 6 Months 95% CI PFS Rate at 9 Months 95% CI PFS Rate at 12 Months 95% CI | xx.x%<br>xx.x; xx.x]<br>xx.x%<br>[xx.x; xx.x]<br>xx.x%<br>[xx.x; xx.x]<br>xx.x%<br>[xx.x; xx.x] | xx.x% [xx.x; xx.x] | |

Notes: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first. See the SAP for the handling of censored cases.

- [a] OS is defined as the time from the date of randomization to death due to any cause..
- [b] Stratified Cox PH regression adjusted for stratification factors: HPV (positive vs other) at randomization.
- [c] Cox PH regression did not adjust for stratification factors.
- [d] Estimate and CI for OS rate at the specified timepoint are from Kaplan-Meier analysis.

Programming note: If insufficient #'s of subject progress then certain proportions are not estimable and the estimate and corresponding confidence interval will be omitted.

Programming Note: continue for different HRG Cutoff

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.3.1: Best Overall Tumor Response and Objective Response Rate (ORR) Full Analysis Set

| | i uli Alialysis | 361 | |
|---|---|---|---|
| HRG High | <u> </u> | | |
| | Patritumab + cetuximab + | Placebo + cetuximab + | |
| | cisplatin or carboplatin | cisplatin or carboplatin | |
| Subjects with measurable disease | (N=xxx) | (N=xxx) | |
| Subject with Measurable Disease at Baseline, n (%) | xx (xx.x) | xx (xx.x) | |
| Objective Response (CR, PR) | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | |
| 95% CI [a] | [xx.x; xx.x] | [xx.; xx x] | |
| Between-arm difference (relative to placebo) | [88.8, 88.8] | [70%, 7, 70%, 7] | |
| 95% CI [b] | | .10 | [xx.x; xx.x] |
| 80% CI [b] | | | |
| 00 % Ci [b] | | | [xx.x; xx.x] |
| Complete Response (CR) | | | |
| | xx (xx.x%) | xx (xx.x%) | |
| n (%)<br>95% CI [a] | [xx.x; x x] | [xx.x; xx.x] | |
| 90 % OI [a] | [^^.^, ^ ^] | [^^.^, ^^.^] | |
| Partial Response (PR) | | | |
| n (%) | xx (xx.x ) | xx (xx.x%) | |
| 95% CI [a] | [xx.x; xx.x] | [xx.x; xx.x] | 95% CI [a] |
| 33 /0 GI [a] | [٨٨.٨, ٨٨.٨] | [^^.^, ^^.^] | 35 /0 OI [a] |
| Stable Disease (SD) | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | |
| 95% CI [a] | | | |
| 95% CI [a] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Progressive Disease (PD) | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | |
| 95% CI [a] | [xx.x; xx.x] | [xx.x; xx.x] | |
| 30 /0 OI [a] | [^^.^, | [^^.^, ^^.^] | |
| Inevaluable | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | |
| 11 ( /0 ) | AX (AX.A /0) | AA (AA.A /0) | |

Note: Denominator for percentages is the number of subjects with measurable disease.

The best overall response is the best response (in the order of CR, PR, SD, and PD) among all overall responses recorded from the start of treatment until the subject withdraws from the study. If there is no post-baseline tumor assessment or all post-baseline tumor assessments with overall response of Inevaluable captured in the CRF, the best overall response is classified as Inevaluable.

- [a] Based on Wilson's score method for single proportion with continuity correction.
- [b] Based on Wilson's score method for the difference of two proportions with continuity correction.

## U31287-A-U203 Statistical Analysis Plan | VV-TMF-2768034 | 1.0

Source Data: adam.adrs; Appendices 16.2.6.1.3, 16.2.6.3 Programming Note: continue for HRG Low and Overall on the next page

The following table follows Table 15.2.3.1:

Table 15.2.3.2 Best Overall Tumor Response and Objective Response Rate (ORR)
Per Protocol Analysis Set


Downloaded

Protocol U31278-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Programming Note: continue for different HRG Cutoff.

Table 15.2.4: Duration of Objective Response/Stable Disease and Time to Response/Disease Progression in Months Full Analysis Set

| HRG | High |
|-----|------|

| | Patritumab + cetuximab + | Placebo + cetuximab + |
|---|---|---|
| | cisplatin or carboplatin | cisplatin or carboplatin |
| | (N=xxx) | (N=xxx) |
| Ouration of Objective Response [a] | | |
| Subjects with Objective Response | XX | XX |
| n. (%) subjects with radiographic disease progression | xx (xx.x%) | xx (xx.x%) |
| Median | XX.XX | XX.XX |
| 95% CI for Median | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| 80% CI for Median | [xx.xx, xx xx] | [xx.xx, xx.xx] |
| 1 <sup>st</sup> Quantile | XX XX | XX.XX |
| 3 <sup>rd</sup> Quantile | XX.XX | XX.XX |
| Min, Max | XX.X XX.X* | XX.X*, XX.X |
| Ouration of Stable Disease [a] | | |
| Subjects with Stable Disease | XX | XX |
| n (%) subjects with radiographic disease progression | xx (xx.x%) | xx (xx.x%) |
| Median | XX.XX | XX.XX |
| 95% CI for Median | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| 80% CI for Median | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| 1 <sup>st</sup> Quantile | XX.XX | XX.XX |
| 3 <sup>rd</sup> Quantile | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X* | XX.X*, XX.X |

#### Notes:

Duration of objective response is defined for subjects with CR/PR as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease.

Duration of SD is defined for subjects whose best response is SD as the time from the randomization date to the date of the first documentation of progressive disease.

Time to response is defined as the time from the randomization date to the date of the first documentation of objective response (CR or PR).

Time to disease progression is defined as the time from the randomization date to the date of first objective documentation of disease progression. See the SAP for the handling of censored cases.

[a] Median, 1st and 3rd quantiles are from Kaplan-Meier Estimate. CI for median was computed using the Brookmeyer-Crowley method. Minimum and maximum include the censored observations where using "+" after value indicates censoring.

Source Data: adam.adtte; Listing 16.2.6.2, 16.2.6.3

Protocol U31278-A-U203

Page x of y

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.4.: Duration of Objective Response/Stable Disease and Time to Response/Disease Progression in Weeks Full Analysis Set

HRG High

| xx (xx.x%)<br>xx.xx<br>[xx.xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx<br>xx.xx | xx (xx.x%)<br>xx.xx<br>[xx.xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx<br>xx.xx |
|---|---|
| xx.xx [xx.xx, xx.xx] [xx.xx, xx.xx] xx.xx xx.xx | xx.xx<br>[xx.xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx |
| [xx.xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx<br>xx.xx | [xx.xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx |
| [xx.xx, xx.xx]<br>xx.xx<br>xx.xx | [xx.xx, xx.xx]<br>xx.xx |
| [xx.xx, xx.xx]<br>xx.xx<br>xx.xx | xx.xx |
| XX.XX | |
| | vv vv |
| var | ۸۸.۸۸ |
| xx.x, xx.x | xx.x, xx.x |
| xx ( x.x%) | xx (xx.x%) |
| XX.XX | XX.XX |
| [x xx, xx.xx] | [xx.xx, xx.xx] |
| [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| XX.XX | XX.XX |
| XX.XX | XX.XX |
| XX.X, XX.X | XX.X, XX.X |
| | xx.xx<br>[x xx, xx.xx]<br>[xx.xx, xx.xx]<br>xx.xx<br>xx.xx |

### Notes

Duration of objective response is defined for subjects with CR/PR as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease.

Duration of SD is defined for subjects whose best response is SD as the time from the randomization date to the date of the first documentation of progressive disease.

Time to response is defined as the time from the randomization date to the date of the first documentation of objective response (CR or PR).

Time to disease progression is defined as the time from the randomization date to the date of first objective documentation of disease progression. See the SAP for the handling of censored cases.

[a] Median, 1<sup>st</sup> and 3<sup>rd</sup> quantiles are from Kaplan-Meier Estimate. CI for median was computed using the Brookmeyer-Crowley method. Minimum and maximum include the censored observations where using "+" after value indicates censoring.

Source Data: adam.adtte; Listing 16.2.6.2, 16.2.6.3

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.5: Summary of Change and the Percent Change from Baseline in the Sum of Longest Diameters (mm) of Target Lesions Full Analysis Set

HRG High

| | | tritumab + cetuxima<br>isplatin or carbopla<br>(N-xxx) | | | Placebo + cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| Visit | Result<br>(mm) | Change<br>(mm) | % Change | Result | Change | % Change |
| Baseline | | , | - | | <u> </u> | |
| n | XX | | | XX | | |
| Mean | XX.X | | | XX.X | | |
| SD | XX.XX | | 4 K | XX.XX | | |
| Median | XX.X | | | XX.X | | |
| Minimum | XX. | | | XX. | | |
| Maximum | xx | | (O) | xx | | |
| Week X | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX. | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX. | XX | XX. | XX. | XX. | XX. |
| Maximum | XX | ХХ | XX | XX | XX | XX |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Time points with data from fewer than 5 subjects overall are not summarized. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of minimum post -baseline values.

Source Data: adam.adrs; Listing 16.2.6.1.3

Protocol U31278-A-U203

<run date time>

Page x of y

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.2.5: Summary of Change and the Percent Change from Baseline in the Sum of Longest Diameters (mm) of Target Lesions Full Analysis Set

HRG High

| Patritumab + cetuximab + | Placebo + cetuximab + |
|--------------------------|--------------------------|
| cisplatin or carboplatin | cisplatin or carboplatin |
| (N-xxx) | (N=xxx) |

| | | (14 ////) | | | (14-7///) | |
|---|---|---|---|---|---|---|
| Visit | Result | Change | | | • | |
| | (mm) | (mm) | % Change | Result | Change | % Change |
| Week N | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX. | XX. | XX | XX. | XX. | XX. |
| Maximum | XX | XX | XX | XX | XX | XX |
| Minimum Post-baseline Value<br>(Nadir) | | | 1 | | | |
| n | XX | | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX. | XX. | XX. | XX. | XX. | XX. |
| Maximum | XX | XX | XX | XX | XX | XX |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Time points with data from fewer than 5 subjects overall are not summarized. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of minimum post-baseline values.

Source Data: adam.adrs; Listing 16.2.6.1.3

Protocol U31278-A-U203

Page x of y rogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.1: Overview of Number (%) of Subjects Reporting Treatment-Emergent Adverse Events Safety Analysis Set

**HRG High** 

| | Patritumab+ cetuximab + | Placebo + cetuximab + | |
|---|---|---|---|
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Freatment-Emergent Adverse Events (TEAE) Worst CTCAE Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | · · · (· · ) | | (// |
| TEAE Related to Patritumab Worst CTCAE Grade | xx (xx.x%) | xx ( x x%) | xx (xx.x%) |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Wildering | AA (AA.A70) | λλ (λλ.λ/υ) | AA (AA.A70) |
| TEAE Related to Cetuximab Worst CTCAE Grade | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | xx (xx.x% | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (x x%) | xx (xx.x%) | xx (xx.x%) |
| <br>>=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE Related to Cisplatin<br>Worst CTCAE Grade | <b>&gt;</b> | | |
| TEAE Related to Carboplatin Worst CTCAE Grade | | | |
| ••• | | | |

Notes: In the presence of a subject who has both missing and non-missing CTCAE grades for adverse events, the missing CTCAE grade of the adverse event is treated as the lowest severity grade.

Adverse events were coded using the MedDRA dictionary, Version XXX.

Source Data: adam.adae; Listing 16.2.7.2.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.1: Overview of Number (%) of Subjects Reporting Treatment-Emergent Adverse Events Safety Analysis Set

HRG High

| | Patritumab + cetuximab + | Placebo + cetuximab + | <b>-</b> |
|---|---|---|---|
| | cisplatin or carboplatin | cisplatin or carboplatin | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Treatment-Emergent SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Worst CTCAE Grade | | | |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx x%) | xx (xx.x%) |
| >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | | 1 | |
| Freatment-Emergent SAE Related to Patritumab Worst CTCAE Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| reatment-Emergent SAE Related to Cetuximab Worst CTCAE Grade | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx ( x.x%) | xx (xx.x%) | xx (xx.x%) |
| <br>>=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Freatment-Emergent SAE Related to Cisplatin Worst CTCAE Grade | | | |

. . .

Treatment-Emergent SAE Related to Carboplatin Worst CTCAE Grade

. . . .

Notes: In the presence of a subject who has both missing and non-missing CTCAE grades for adverse events, the missing CTCAE grade of the adverse event is treated as the lowest severity grade.

Adverse events were coded using the MedDRA dictionary, Version XXX.

Source Data: adam.adae; Listing 16.2.7.2.

Protocol U31278-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.1: Overview of Number (%) of Subjects Reporting Treatment-Emergent Adverse Events Safety Analysis Set

**HRG High** 

| пко підії | Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Discontinued Patritumab Due to TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Cetuximab Due to TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Cisplatin Due to TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Carboplatin Due to TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Patritumab Interruption TEAE leading to Patritumab Interruptio Related to Patritumab TEAE leading to Patritumab Dose Reduction TEAE leading to Patritumab Dose Reduction Related to Patritumab Discontinued Patritumab Due to TEAE Related to Patritumab | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Discontinued Cetuximab Due to TEAE<br>Related to Cetuximab | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Cisplatin Due to TEAE Related to Cisplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Carboplatin Due to TEAE Related to Carboplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Patritumab Due to Treatment Emergent SAE Discontinued Cetuximab Due to Treatment Emergent SAE Discontinued Cisplatin Due to Treatment Emergent SAE Discontinued Carboplatin Due to Treatment Emergent SAE | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

Notes: In the presence of a subject who has both missing and non-missing CTCAE grades for adverse events, the missing CTCAE grade of the adverse event is treated as the lowest severity grade.

Adverse events were coded using the MedDRA dictionary, Version XXX.

Source Data: adam.adae; Listing 16.2.7.2.

Page x of y run date time>

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.1: Overview of Number (%) of Subjects Reporting Treatment-Emergent Adverse Events Safety Analysis Set

HRG High

| Tirto riigii | Patritumab+ cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab +<br>cisplatin or carboplatin<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Discontinued Patritumab Due to Treatment Emergent SAE Related to Patritumab | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Cetuximab Due to Treatment Emergent SAE Related to Cetuximab | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Cisplatin Due to Treatment Emergent SAE Related to Cisplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Carboplatin Due to Treatment Emergent SAE Related to Carboplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Death Related to Patritumab | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Death Related to Cetuximab | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Death Related to Cisplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE leading to Death Related to Carboplatin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: In the presence of a subject who has both missing and non-m ssing CTCAE grades for adverse events, the missing CTCAE grade of the adverse event is treated as the lowest severity grade.

Adverse events were coded using the MedDRA dict onar Versio XXX.

Source Data: adam.adae; Listing 16.2.7.2.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.2: Number and Percentage of Subjects with Treatment-emergent Adverse Events Summarized by Worst CTCAE Grade,
System Organ Class, and Preferred Term
Safety Analysis Set

HRG High

| - | | Worst CTCAE | Patritumab+ cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|
| System Organ Class | Preferred Term | Grade | n (%) | n (%) | n (%) |
| Subjects with any TEAEs | | Any Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| , | | 5 | xx (xx.x%) | xx (x x%) | xx (xx.x%) |
| | | 4 | xx (xx.x%) | xx (xx %) | xx (xx.x%) |
| | | 3 | xx (xx.x%) | xx (xx.x ) | xx (xx.x%) |
| | | 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 1 | xx (xx.x%) | xx (x x%) | xx (xx.x%) |
| | | >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #1 | Any Preferred Term | Any Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 5 | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| | | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 3 | xx (x x%) | xx (xx.x%) | xx (xx.x%) |
| | | 2 | xx (xx. %) | xx (xx.x%) | xx (xx.x%) |
| | | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Missing | x (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: In the presence of a subject who has both missing and non-mis ing CTCAE grades for adverse events with the same preferred term, the missing CTCAE grade of the adverse event is treated as the lowes sever y grade.

Subjects may have more than one event per system organ class and preferred term. At each level of subject summarization, a subject was counted once if he/she reported one or more adverse events.

Adverse events were coded using the MedDRA dictionary, Version XXX.

Source Data: adam.adae; Listing 16.2.7.2.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.1.2: Number and Percentage of Subjects with Treatment-emergent Adverse Events Summarized by Worst CTCAE Grade,
System Organ Class, and Preferred Term
Safety Analysis Set

**HRG High** 

| - | | Worst CTCAE | Patritumab+ cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|
| System Organ Class | Preferred Term | Grade | n (%) | n (%) | n (%) |
| System Organ Class #1 | Preferred Term #1 | Any Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| , | | 5 <sup>°</sup> | xx (xx.x%) | xx (x x%) | xx (xx.x%) |
| | | 4 | xx (xx.x%) | xx (xx. %) | xx (xx.x%) |
| | | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 2 | xx (xx.x%) | xx ( x.x%) | xx (xx.x%) |
| | | 1 | xx (xx.x%) | x (xx x%) | xx (xx.x%) |
| | | >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #1 | Preferred Term N | Any Grade | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 5 | xx (xx x%) | xx (xx.x%) | xx (xx.x%) |
| | | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 3 | xx (x x%) | xx (xx.x%) | xx (xx.x%) |
| | | 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 1 | xx ( x.x%) | xx (xx.x%) | xx (xx.x%) |
| | | >=3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class N | Any<br>Preferred Term<br>Etc. | | Y | | |

Notes: In the presence of a subject who has both missing and non-missing CTCAE grades for adverse events with the same preferred term, the missing CTCAE grade of the adverse event is treated as the lowest severity grade.

Subjects may have more than one event per system organ class and preferred term. At each level of subject summarization, a subject was counted once if he/she reported one or more adverse events.

Adverse events were coded using the MedDRA dictionary, Version XXX.

Source Data: adam.adae; Listing 16.2.7.2.
Page x of y

Protocol U31278-A-U203

<run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

The following table follows 15.3.1.2:

Table 15.3.1.3: Number and Percentage of Subjects with Treatment-emergent Serious Adverse Events Summarized by Worst CTCAE Grade, System Organ Class, and Preferred Term Safety Analysis Set

First Row: Subjects with any treatment emergent SAEs

Table 15.3.1.4: Number and Percentage of Subjects with Treatment-emergent Adverse Events Related to Patritumab/Placebo Summarized by Worst CTCAE Grade, System Organ Class, and Preferred Term Safety Analysis Set

First Row: Subjects with any TEAEs related to Patritumab

Table 15.3.1.5: Number and Percentage of Subjects with Treatment-emerg t Adverse Events Related to Cetuximab Summarized by Worst CTCAE Grade, System Organ Class, and Preferred Term

Safety Analysis Set

First Row: Subjects with any TEAEs related to Cetuximab

Table 15.3.1.6: Number and Percentage of Subjects with reatment-emergent Adverse Events Related to Cisplatin/Carboplatin Summarized by Worst CTCAE Grade System Organ Class, and Preferred Term Safety Analysis Set

First Row: Subjects with any TEAEs related to Cisplatin/ Carbop atin

Table 15.3.1.7: Number and Percentage of Subjects with Treatment-emergent Serious Adverse Events Related to Patritumab/Placebo Summarized by Worst CTCAE Grade, System Organ Class, and Preferred Term

Safety Analysis Set

First Row: Subjects with any treatment emergent SAEs related to Patritumab

Table 15.3.1.8: Number and Percentage of Subjects with Treatment-emergent Serious Adverse Events Related to Cetuximab Summarized by Worst CTCAE Grade, System Organ Class, and Preferred Term

Safety Analysis Set

First Row: Subjects with any treatment emergent SAEs related to Cetuximab

Table 15.3.1.9: Number and Percentage of Subjects with Treatment-emergent Serious Adverse Events Related to Cisplatin/Carboplatin Summarized


Downloaded on one

Page x of y rogname<run date time>

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

by Worst CTCAE Grade, System Organ Class, and Preferred Term Safety Analysis Set

First Row: Subjects with any treatment emergent SAEs related to Cisplatin/Carboplatin

Table 15.3.1.10: Number and Percentage of Subjects with Adverse Events of Interest by Worst CTCAE Grade, System Organ Class, and Preferred Term Safety Analysis Set

First Row: Subjects with any adverse events of interest


Downloaded

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.4.1: Summary of Results and Change from Baseline in Laboratory Tests – Hematology Safety Analysis Set

### HRG High

| Lab Test (units) | Patritumab+ cetuximab + cisplatin or carboplatin(N=xxx) | | | cetuximab +<br>carboplatin<br>xxx) | | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Visit | Result | Change | Result | Change | Result | Change |
| Lab Test #1 (SI unit) Baseline | | | | | | |
| n | XX | | XX | | XX | |
| Mean | xx.x | | XX.X | | XX.X | |
| SD | XX.XX | | XX.XX | | XX.XX | |
| Median | XX.X | | XX.X | | XX.X | |
| Minimum | XX | | XX | | XX | |
| Maximum | xx | | XX | 1 | XX | |
| Cycle X Day X | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | xx | XX | X | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |

Note: The baseline value is defined as the last non-missing value before initia administration of study treatment. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration + 7. Perce tages are bised on the number of subjects meeting the defined criteria (m); the number of subjects with non-missing observations for the specified visit (n) is the denominator.

Source Data: adam.adlb; Listing 16.2.8.1.1

Programming Note: do not summarize Cycle 1 Day 1. Do not summarize coagulation parameters.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.4.1: Summary of Results and Change from Baseline in Laboratory Tests – Hematology Safety Analysis Set

HRG High

| | | cetuximab + | Placebo + ce | | _ | |
|---|---|---|---|---|---|---|
| | | carboplatin | cisplatin or o | | | tal |
| Lab Test (units) | | xxx) | (N=x> | | (N=xxx) | |
| Visit | Result | Change | Result | Change | Result | Change |
| Lab Test #1 (SI unit) | | | | | | |
| End of Treatment | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |
| | | | | 1 1 1 | | |
| Last Observation on Treatment | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |
| Maximum Post-Baseline Value | | | | | | |
| | | . 4 | | | | |
| Minimum Post-Baseline Value | | | | | | |
| Lab Test N | | | | | | |

#### Lab Test N....

Note: The baseline value is defined as the last non-missing value before initial administration of study treatment. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of last observation on treatment, maximum and minimum post-baseline values. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration + 7. Percentages are based on the number of subjects meeting the defined criteria (m); the number of subjects with non-missing observations for the specified visit (n) is the denominator.

Source Data: adam.adlb; Listing 16.2.8.1.1

Programming Note: do not summarize Cycle 1 Day 1. Do not summarize coagulation parameters.

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYYY)

The following table follows Table 15.3.4.1:

Table 15.3.4.2: Summary of Results and Change from Baseline in Laboratory Tests - Chemistry Safety Analysis Set

Source Data: adam.adlb; Listing 16.2.8.1.2




Downloaded

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.4.3: Shift Table of CTCAE Grade in Laboratory Tests – Hematology Safety Analysis Set

HRG High

| | | | | V | Vorst Post-basel | ine CTCAE Grad | de | | |
|---|---|---|---|---|---|---|---|---|---|
| Condition (Unit) | Baseline | < 1 | 1 | 2 | 3 | 4 | 3 or 4 | Total | Missing |
| Treatment | CTCAE Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n |
| Condition #1 | | | | | | | | | |
| Patritumab+ cetuximab + cisplatin or carboplatin | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| (n=xxx) | < 1 | | | | | | | | XX |
| | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | x (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 3 or 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Missing | XX | XX | xx | xx | xx | xx | XX | XX |
| Placebo + cetuximab + cisplatin or carboplatin | | xx (xx.x%) | xx (xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| (n=xxx) | < 1 | | | | | | | | XX |
| , | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 2 | xx (xx.x%) | x (x .x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 4 | xx (xx. %) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | 3 or 4 | x (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Missing | X | xx | xx | xx | xx | xx | xx | xx |

### Condition #2 . . . etc.

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment.

For each condition, percentages are based on the number of subjects in the Safety Analysis Set for each cohort with a baseline and at least one post-baseline assessment (that is, n in the first column). Subjects classified as missing have a missing test result.

Source Data: adam.ad b; Listing 16.2.8.1.1

Programming note: do not summarize coagulation parameters.

Page x of y rogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

The following table follows 15.3.4.3:

Table 15.3.4.4: Shift Table of CTCAE Grade in Laboratory Tests - Chemistry Safety Analysis Set

Source Data: adam.adlb; Listing 16.2.8.1.2




Downloaded

Protocol U31278-A-U203

Page x of y

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.4.5: Number and Percentage of Subjects with Liver Enzymes (ALT, AST) and Total Bilirubin (TBL) Elevation Safety Analysis Set

### **HRG High**

| Category | Patritumab+ cetuximab + cisplatin or carboplatin (N=xxx) | Placebo + cetuximab + cisplatin or carboplatin (N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Subjects with post-baseline AST | (11 700) | (11 700) | (11 700) |
| AST >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 5 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 8 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 10 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 20 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with post-baseline ALT | | | |
| ALT >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >= 5 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| $ALT >= 8 \times ULN$ | xx (xx x) | xx (xx.x) | xx (xx.x) |
| $ALT >= 10 \times ULN$ | x (xx.x) | xx (xx.x) | xx (xx.x) |
| $ALT \ge 20 \times ULN$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with post-baseline AST or ALT | | | |
| AST >= 3 x ULN or ALT >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 5 x ULN or ALT >= 5 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 8 x ULN or ALT >= 8 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 10 x ULN or ALT >= 10 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >= 20 x ULN or ALT >= 20 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TBL >= 2 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurent TBL >= 2 x ULN and AST >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurent TBL >= 2 x ULN and ALT >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurent TBL >= 2 x ULN and AST or ALT >= 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurent TBL $>= 2 x$ ULN and AST or ALT $>= 3 x$ ULN and ALP $>= 2 x$ U | JLN xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurent TBL >= 2 x ULN and AST or ALT >= 3 x ULN and ALP <= 2 x l | JLN xx (xx.x) | xx (xx.x) | xx (xx.x) |

Notes: ULN = Upper limit of normal ranges.

Concurrent is defined as at least one case of post-dose TBL >= 2 x ULN occurred between the first incidence date and 30 days after the last incidence date of the corresponding liver enzyme(s) >= 3 x ULN

Source Data: adam.adlb; Listing 16.2.8.1.1

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.5: Summary of Vital Signs and Change from Baseline Safety Analysis Set

**HRG High** 

| HRG High | Dotritures | actualmah I | Dlasska | actuvimah I | | |
|---|---|---|---|---|---|---|
| | Patritumab+<br>cisplatin or | | | cetuximab +<br>carboplatin | т, | otal |
| /ital Sign (units) | | | (N= | | (N=) | |
| Visit | (N=xxx)<br>Result Change | | Result | Change | | |
| VIOIL | resuit | Change | Result | Change | resuit | Change |
| ystolic Blood Pressure (mmHg) | | | | | | |
| Baseline | | | | | | |
| n | XX | | XX | | XX | |
| Mean | XX.X | | XX.X | | XX.X | |
| SD | XX.XX | | XX.XX | | XX.XX | |
| Median | XX.X | | XX.X | | XX.X | |
| Minimum | XX | | XX | | XX | |
| Maximum | XX | | XX | 1 K J | XX | |
| Cycle 1 Day 1 | | | | | | |
| Pre-infusion | | | | | | |
| n | XX | | XX | | XX | |
| Mean | XX.X | | XX | | XX.X | |
| SD | XX.XX | | XX.XX | | XX.XX | |
| Median | XX.X | | ХX | | XX.X | |
| Minimum | XX | | XX | | XX | |
| Maximum | XX | | XX | | XX | |
| Post-infusion | | | | | | |
| n | xx | XX | XX | XX | XX | xx |
| Ovela N. Davi N. | The state of the s | | | | | |
| Cycle N Day N | | · | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of last observation on treatment, maximum and minimum post-baseline values. The End of Treatment value is based on the CRF visit. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration + 7.

Source Data: adam.advs; Listing 16.2.8.3.1.

Programming note: continue table for Diastolic Blood Pressure, Pulse Rate, Temperature and Weight

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.5: Summary of Vital Signs and Change from Baseline Safety Analysis Set

HRG High

| | Patritumab+ | + cetuximab + | Placebo + o | etuximab + | | |
|---|---|---|---|---|---|---|
| | | r carboplatin | cisplatin or | | То | |
| Vital Sign (units) | | xxx) | (N=x | | (N=x | |
| Visit | Result | Change | Result | Change | Result | Change |
| Systolic Blood Pressure (mm Hg) End of Treatment | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | X.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |
| | | | | . 1 | | |
| Last Observation on Treatment | | | | | | |
| n | XX | XX | XX | Х | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | xx x | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | XX | XX | XX | XX | XX |
| Maximum Post-baseline Value | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | X.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | XX | XX | XX | XX | XX |
| Maximum | XX | xx | XX | XX | XX | XX |

Minimum Post-baseline Value

#### Lab Test N (SI unit)

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of last observation on treatment, maximum and minimum post-baseline values. The End of Treatment value is based on the CRF visit. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment duration + 7.

Source Data: adam.advs; Listing 16.2.8.3.1.

Programming note: continue table for Diastolic Blood Pressure, Pulse Rate, Respiratory Rate, Body Temperature and Weight

Protocol U31278-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.6.1: Summary of 12-Lead ECG and Change from Baseline Safety Analysis Set

HRG High

| Parameter (units) | Patritumab+<br>cisplatin or<br>(N=x | carboplatin<br>xx) | cisplatin o | cetuximab +<br>r carboplatin<br>exxx) | To<br>(N=) | |
|---|---|---|---|---|---|---|
| Visit | Result | Change | Result | Change | Result | Change |
| Heart Rate (bpm)<br>Baseline | | | | | | |
| n | XX | | XX | | Х | |
| Mean | XX.X | | XX.X | | XX.X | |
| SD | XX.XX | | XX.XX | $A \times J$ | XX.XX | |
| Median | XX.X | | XX.X | | XX.X | |
| Minimum | XX | | XX | | XX | |
| Maximum | XX | | XX | | XX | |
| End of Treatment | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.X | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | X.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX | X | XX | XX | XX | XX |
| Maximum | XX | xx | XX | XX | XX | XX |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. The End of Treatment value is based on the CRF visit

Source Data: adam.adeg; Listing 16.2.8.3.2.

Programming note: continue with PR interval, RR interval, QRS duration, QT interval, QTcB, and QTcF Programming Note: continue for HRG Low and Overall on the next page

Protocol U31278-A-U203

Page x of y rogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.6.2: Summary of Subjects Meeting Pre-Specified QT and QTcB/QTcF Criteria Safety Analysis Set

HRG High

| | Patritumab+ cetuximab + cisplatin | Placebo + cetuximab + cisplatin or carboplatin | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Maximum Over All Post- Baseline Evaluations | n (%) | `n (%) ´ | `n (%) ´ |
| Subjects with at least one baseline and one post-<br>baseline ECG evaluation | xx | xx | xx |
| QTcB | | | |
| New > 450 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| New > 480 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| New > 500 msec | xx (xx.x%) | xx (x x%) | xx (xx.x%) |
| Change from baseline >30 msec | xx (xx.x%) | xx xx.x%) | xx (xx.x%) |
| Change from baseline > 60 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QTcF | | | |
| New > 450 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| New > 480 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| New > 500 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Change from baseline >30 msec | xx ( x.x%) | xx (xx.x%) | xx (xx.x%) |
| Change from baseline > 60 msec | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Percentages are based on the number of subjects in the Safety Analysis Set for each cohort with at least one baseline and one post-baseline ECG assessment. "New" means the category of the QTc abnormality was not present at baseline and became present at least one post-baseline ECG assessment.

Source Data: adam.adeg; Listing 16.2.8.3.2.

Programming Note: continue for HRG Low and Overall on the next page

Downloaded

Protocol U31278-A-U203

Page x of y

cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY) Table 15.3.7: Shift Table of ECOG Status Safety Analysis Set

HRG High

| | | | | Pos | t-Baseline ECO | S PS | | | |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Baseline | 0 | 1 | 2 | 3 | 4 | 5 | Total | Missing |
| Treatment | ECOG PS | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n |
| Cycle 1 Day 1 | | | | | | | | | |
| Patritumab+ cetuximab + cisplatin | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| or carboplatin (n=xxx) | 0 | , , | , , | , , | | , , | , , | , , | XX |
| | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Missing | XX | XX | XX | XX | XX | XX | XX | XX |
| Placebo + cetuximab + cisplatin or | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Carboplatin (n=xxx) | 0 | , , | , , | | | , | , , | , , | XX |
| . , , | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x% | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Missing | `xx | xx | xx | xx | xx | `xx | xx | XX |

Cycle x Day 1

**End of Treatment** 

Last Observation on Treatment

Maximum Post-baseline Value

Minimum Post-baseline Value

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. For each test, percentages are based on the number of subjects in the Safety Analysis Set for each cohort with a baseline and at least one post-baseline ECOG assessment (that is, n in the first column).

Subjects classified as missing have a missing test result.

Source Data: adam.adgs; Listing 16.2.8.3.4.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.3.8: Summary of Left Ventricular Ejection Fraction (LVEF) Value and Change from Baseline Safety Analysis Set

HRG High

| Parameter (units) | Patritumab+<br>cisplatin oi<br>(N= | cisplatin or<br>(N= | cetuximab +<br>r carboplatin<br>xxxx) | Total<br>(N=xxx) | | |
|---|---|---|---|---|---|---|
| Visit | Result | Change | Result | Change | Result | Change |
| LVEF (%) | | | | | | |
| Baseline | | | | | | |
| n | XX | | XX | | XX | |
| Mean | XX.X | | XX.X | | xx x | |
| SD | XX.XX | | XX.XX | | XX.XX | |
| Median | XX.X | | XX.X | | XX.X | |
| Minimum | XX | | XX | . 1 | xx | |
| Maximum | XX | | xx | | XX | |
| Cycle X Day X | | | | | | |
| n | XX | XX | X | XX | XX | XX |
| Mean | XX.X | XX.X | XX | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX X | XX.X | XX.X | XX.X | XX.X |
| Minimum | xx | XX | XX | XX | XX | XX |
| Maximum | XX | X | XX | XX | XX | XX |
| Cycle N Day N | | $\mathcal{V}$ | | | | |
| End of Treatment | | | | | | |
| Last Observation on Treatment | | | | | | |
| Maximum Post-baseline Value | | | | | | |
| Minimum Post-baseline Value | | | | | | |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment. Repeated or unscheduled tests are not summarized for each scheduled visit, but are included for summaries of last observation on treatment, maximum and minimum post-baseline values. The End of Treatment value is based on the CRF visit. Last observation on treatment is defined as the last non-missing value on or prior to end of treatment period + 7.

Source Data: adam.adeg; Listing 16.2.8.3.5.

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.1: Summary of Patritumab Concentration (ug/mL) from Sparse PK Sampling Pharmacokinetic Analysis Set

HRG High

C1D1 C1D1 C2D1 C3D1 C3D1
ent Pre-Infusion End of Infusion Pre-Infusion Pre-Infusion End of Infusion End of Treatment

Sample Times

| Treatment | Pre-Infusion | End of Infusion | Pre-Infusion | Pre-Infusion | End of Infusion | End of Treatment |
|---|---|---|---|---|---|---|
| Patritumab+ cetuximab + | | | | | | |
| cisplatin or carboplatin | | | | | | |
| n | xx | xx | xx | xx | xx | xx |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | XX | XX | XX | XX |
| Geom. Mean | XX | XX | XX | XX | XX | XX |
| Geom. CV% | XX | XX | XX | XX | XX | XX |
| Minimum | XX.XXX | XX.XXX | XX.XXX | x.xxx | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XXX | XX.XXX | XX XXX | XX.XXX | XX.XXX | XX.XXX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | x xxx | XX.XXX | XX.XXX | XX.XXX |
| Maximum | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX | XX.XXX |

Notes: Concentrations below the lower limit of quantitation (BLQ) are et to zero fo the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time po t is not c lculated and is presented as "NC".

CXDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.1.

Programming Note: List scheduled times as shown in table 8 1 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.2: Summary of Patritumab Concentration (ug/mL) from Intensive PK Sampling at Cycle 1

Pharmacokinetic Analysis Set

HRG High

| | | | Sample | Times | | | |
|---|---|---|---|---|---|---|---|
| Treatment | C1D1<br>Pre-Infusion | C1D1<br>End of<br>Infusion | C1D1<br>3 Hours Post<br>Infusion | C1D1<br>4 Hours Post<br>Infusion | C1D1<br>5 Hours Post<br>Infusion | C1D1<br>6 Hours Post<br>Infusion | C1D1<br>7 Hours Posi<br>Infusion |
| Patritumab+ cetuximab + cisplatin or carboplatin | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | XX | XX | XX | XX | XX |
| Geom. Mean | XX | XX | XX | XX | XX | XX | XX |
| Geom. CV% | XX | XX | XX | XX | XX | XX | XX |
| Minimum | XX.XXX | XX.XXX | XX.XXX | x xxx | XX.XXX | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XXX | XX.XXX | XX X X | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Maximum | XX.XXX | XX.XXX | xx xxx | xx.xxx | XX.XXX | XX.XXX | XX.XXX |

Notes: Concentrations below the lower limit of quantitation (BLQ) a set t zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC".

CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.1.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31278-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.2: Summary of Patritumab Concentration (ug/mL) from Intensive PK Sampling at Cycle 1
Pharmacokinetic Analysis Set

**HRG High** 

| | | Sample Times | | |
|---|---|---|---|---|
| C1D2 | C1D3 | C1D8 | C1D15 | C1D21 |
| 24 Hours Post | 48 Hours Post | 168 Hours Post | 336 Hours Post | 504 Hours Post |
| Infusion | Infusion | Infusion | Infusion | Infusion |
| XX | xx | XX | xx | xx |
| xx.xxx | XX.XXX | XX.XXX | xx xxx | XX.XXX |
| XX.XXX | XX.XXX | XX.XXX | xx xxx | XX.XXX |
| XX.XXX | XX.XXX | XX.XXX | xx xx | XX.XXX |
| XX | XX | XX | xx | XX |
| XX | XX | XX | xx | XX |
| XX | XX | xx | xx | XX |
| XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| XX.XXX | XX.XXX | xx.x x | XX.XXX | XX.XXX |
| XX.XXX | XX.XXX | xx.xx | XX.XXX | XX.XXX |
| XX.XXX | XX.XXX | x.xxx | XX.XXX | XX.XXX |
| XX.XXX | XX.XXX | xx xxx | XX.XXX | XX.XXX |
| | 24 Hours Post Infusion XX XX.XXX XX.XXX XX.XXX XX XX X | 24 Hours Post Infusion XX XX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX XX | 24 Hours Post<br>Infusion 48 Hours Post<br>Infusion 168 Hours Post<br>Infusion XX XX XX XX XXXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX XX XX XX XX | 24 Hours Post<br>Infusion 48 Hours Post<br>Infusion 168 Hours Post<br>Infusion 336 Hours Post<br>Infusion XX XX XX XX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX.XXX XX XX XX XX XX |

Notes: Concentrations below the lower limit of quantitation (BLQ) ar-set to-ero-r the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not-alculated and is presented as "NC".

CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.1.

Programming Note: List scheduled times as shown in table 8 2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.3: Summary of Cetuximab Concentration (ug/mL) from Intensive PK Sampling at Cycle 1
Pharmacokinetic Analysis Set

HRG High

| | | | Sample Times | | | |
|---|---|---|---|---|---|---|
| Treatment | C1D1<br>Pre-Infusion | C1D1<br>End of Infusion | C1D1<br>4 Hours Post<br>Infusion | C1D1<br>5 Hours Post<br>Infusion | C1D1<br>6 Hours Post<br>Infusion | C1D1<br>7 Hours Post<br>Infusion |
| Patritumab + cetuximab + | | | | | | |
| cisplatin or carboplatin | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.XXX | XX.XXX | xx.xxx | X .XXX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | xx | XX | XX | XX |
| Geom. Mean | XX | XX | xx | XX | XX | XX |
| Geom. CV% | XX | XX | | | XX | XX |
| Minimum | XX.XXX | XX.XXX | xx xxx | XX.XXX | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | x.xxx | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XXX | XX.XXX | x .xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| Maximum | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Placebo + cetuximab + cisplatin or carboplatin | | | | | | |
| N | XX | xx | XX | xx | xx | xx |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |

Notes: Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC".

CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.2.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.3: Summary of Cetuximab Concentration (ug/mL) from Intensive PK Sampling at Cycle 1 Pharmacokinetic Analysis Set

HRC High

| HRG High | | | |
|--------------------------|---------------|---------------|----------------|
| | | | Sample Times |
| | C1D2 | C1D3 | C1D8 |
| | 24 Hours Post | 48 Hours Post | 168 Hours Post |
| Treatment | Infusion | Infusion | Infusion |
| Patritumab+ cetuximab + | | | |
| cisplatin or carboplatin | | | <b>A</b> |
| n | XX | xx | xx |
| Mean | XX.XXX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | XX |
| Geom. Mean | XX | XX | XX |
| Geom. CV% | xx | XX | XX |
| Minimum | xx.xxx | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | xx.x x |
| Median | XX.XXX | XX.XXX | XX.XX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | X.XXX |
| Maximum | XX.XXX | XX.XXX | xx xxx |
| Placebo + cetuximab + | | | |
| cisplatin or carboplatin | | | |
| N | xx | xx | XX |
| Mean | XX.XXX | XX.XX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX |
| Continue above | | | |

Notes: Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC".

CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.2.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.4: Summary of Cisplatin Concentration (ug/mL) from Intensive PK Sampling at Cycle 1 Pharmacokinetic Analysis Set

HRG HIgh

| | | S | ample Times | | | |
|---|---|---|---|---|---|---|
| Treatment | C1D1<br>Pre-Infusion | C1D1<br>End of Infusion | C1D1<br>6 Hours Post<br>Infusion | C1D1<br>7 Hours Post<br>Infusion | C1D2<br>24 Hours Post<br>Infusion | C1D3<br>48 Hours Post<br>Infusion |
| Datriture als I astronius als I | | | | | | |
| Patritumab + cetuximab + cisplatin | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX XX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | XX | XX | XX | XX |
| Geom. Mean | XX | XX | XX | XX | XX | XX |
| Geom. CV% | XX | XX | XX | XX | XX | XX |
| Minimum | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | XX XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XXX | XX.XXX | XX XXX | XX.XXX | XX.XXX | XX.XXX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Maximum | XX.XXX | XX.XXX | x xxx | XX.XXX | XX.XXX | XX.XXX |
| Placebo + cetuximab + cisplatin | | | | | | |
| N | xx | xx | xx | xx | xx | xx |
| Mean | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | XX.XXX | XX.XXX | xx.xxx | xx.xxx | XX.XXX | XX.XXX |

Notes: Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC". CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.3.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.1.5: Summary of Carboplatin Concentration (ug/mL) from Intensive PK Sampling at Cycle 1
Pharmacokinetic Analysis Set

HRG High

| | | | Sample Times | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | C1D1<br>Pre-Infusion | C1D1<br>End of Infusion | C1D1<br>5 Hours Post<br>Infusion | C1D1<br>6 Hours Post<br>Infusion | C1D1<br>7 Hours Post<br>Infusion | C1D2<br>24 Hours Post<br>Infusion | C1D3<br>48 Hours Post<br>Infusion |
| Patritumab + cetuximab + | | | | | | | |
| carboplatin | | | | | | | |
| N | XX | XX | XX | XX | xx | XX | xx |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SEM | XX | XX | XX | XX | XX | XX | XX |
| Geom. Mean | XX | XX | XX | XX | XX | XX | XX |
| Geom. CV% | XX | XX | XX | XX | XX | XX | XX |
| Minimum | XX.XXX | XX.XXX | XX.XXX | xx xxx | XX.XXX | XX.XXX | XX.XXX |
| 1 <sup>st</sup> Quartile | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 3 <sup>rd</sup> Quartile | XX.XXX | XX.XXX | XX XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Maximum | XX.XXX | XX.XXX | XX. XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Placebo + cetuximab + | | | | | | | |
| carboplatin | | | VY | | | | |
| N | XX | xx | XX | XX | XX | XX | XX |
| Mean | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |

Notes: Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC".

CxDx = Cycle x Day x

Source Data: adam.adpk; Listing 16.2.5.2.4.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.2.1: Summary of Patritumab PK Parameters at Cycle 1
Pharmacokinetic Analysis Set

| <u> </u> | Patritumab +<br>cisplatin or o<br>(N=x | carboplatin |
|---|---|---|
| | AUC <sub>last</sub> | $C_{max}$ |
| Cycle | (ug.day/mL) | (ug/mL) |
| Cycle 1 | | |
| Geometric mean<br>Geometric CV%<br>Arithmetic mean<br>Arithmetic SD<br>Median<br>Min | 100 | Y |
| VIIII | | |

Note: If there are less than 3 values in the data series only the min, max, an N a e presented. The other summary statistics are denoted as not calculated (NC). If one or more of the values in a data series is zero, then do not calculate the geometric mean and geometric CV% and denote them as not applicable (NA). If an entire concentration-time profile is BLQ, PK parameters will b reported as NC and set to missing for summary statistics. For the calculation for summary statistics of PK parameters, all NR and NC values in a data series are set to missing.

Source Data: adam.adpk; Listing 16.2.5.2.1.

Programming Note: List scheduled times as shown in table 8.2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

Max N

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.2.2: Summary of Cetuximab PK Parameters at Cycle 1
Pharmacokinetic Analysis Set

| HRG High | | | | |
|---|---|---|---|---|
| | Patritumab + cisplatin or c | carboplatin | Placebo + c<br>cisplatin or c | carboplatin |
| | (N=x | , | (N=x | |
| | $AUC_{last}$ | $C_{max}$ | $AUC_{last}$ | $C_{max}$ |
| Cycle | (ug.day/mL) | (ug/mL) | (ug.day/mL) | (ug/mL) |
| Cycle 1 | | | | |
| Geometric mean | | | | |
| Geometric CV% | | | | |
| Arithmetic mean | | | | |
| Arithmetic SD | | | | |
| Median | | .10 | | |
| Min | | | | |

Note: If there are less than 3 values in the data series only the min ma and N are presented. The other summary statistics are denoted as not calculated (NC). If one or more of the values in a data series is zero, then do not calculate the geometric mean and geometric CV% and denote them as not applicable (NA). If an entire concentration-time profile is BLQ PK parameters will be ported as NC and set to missing for summary statistics. For the calculation for summary statistics of K parameter all NR and NC values in a data series are set to missing.

Source Data: adam.adpk; Listing 16.2.5.2.1.

Programming Note: List scheduled times as shown in table 8 2 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

The following table follows Table 15.4.2.2:

Table 15.4.2.3 Summary of Cisplatin PK Parameters at Cycle 1 Pharmacokinetic Analysis Set

Table 15.4.2.4 Summary of Carboplatin PK Parameters at Cycle 1 Pharmacokinetic Analysis Set


Downloaded

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.4.2.5: Statistical Analysis of Cetuximab, Cisplatin, and Carboplatin PK Parameters at Cycle 1 Pharmacokinetic Analysis Set

HRG High

| - | Geomet<br>(9: | Ratio of Geometric LS means<br>(90% CI) | |
|---|---|---|---|
| | Patritumab + cetuximab + cisplatin or carboplatin | Placebo + cetuximab + cisplatin or carboplatin | |
| PK Parameter | (N=xxx) | (N=xxx) | Patritumab/Placebo |
| Cetuximab | | <b>A</b> | |
| AUC <sub>last</sub> | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| $C_{max}$ | XX.X | XX.X | xx.x |
| | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Cisplatin | | 1 ( ) | |
| AUC <sub>last</sub> | XX.X | XX.X | XX.X |
| | [xx.x, xx.x] | [xx.x xx x] | [xx.x, xx.x] |
| $C_{max}$ | XX.X | XX.X | XX.X |
| Carboplatin | [xx.x, xx.x] | [x .x, xx.x] | [xx.x, xx.x] |
| AUC <sub>last</sub> | XX.X | XX.X | XX.X |
| | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| $C_{max}$ | XX.X | XX.X | XX.X |
| | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Note: AUC<sub>last</sub> and C<sub>max</sub> will be log-transformed prior o nalysis. The geometric mean ratios and their two-sided 90% CIs for AUC<sub>last</sub> and C<sub>max</sub> between the patritumab arm and the placebo arm will be calculated using the e ponentiation of the differences and their CIs between treatments least square mean from the ANOVA. The ratios and their two-sided 90% CIs will be expressed relative to the placebo arm.

Source Data: adam.adpk; Listing 16.2.5.2.2

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.5.1.1: Summary of Actual Results and Change from Baseline in FACT-H&N Total Score, FACT-H&N Subscale (HNS) Score, HNS Individual Symptom Score, and FACT-H&N Symptom Index (FHNSI) Score FACT-H&N Analysis Set

| PRO Measure<br>Visit | | o + cisplatin or carboplatin<br>=xxx) | | + cisplatin or carboplatin |
|---|---|---|---|---|
| | Result | Change | Result | Change |
| ACT-H&N Total Score | | | | |
| Baseline | | | | |
| n | XX | | XX | |
| Mean | XX.X | | XX.X | |
| SD | XX.XX | | xx.xx | |
| Minimum | XX | | XX | |
| Median | XX.X | 1 ( ) | XX.X | |
| Maximum | XX | | XX | |
| Cycle 2 Day 1 | | | | |
| n | xx | xx | XX | XX |
| Mean | XX.X | xx.x | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | xx | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | xx | XX | XX |
| Cycle 3 Day 1 | | <i>y</i> | | |
| n | XX | xx | xx | XX |
| Mean | xx.x | XX.X | XX.X | xx.x |
| SD | xx.xx | XX.XX | XX.XX | XX.XX |
| Minimum | XX | xx | xx | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX |

Continue with Cycle 4 Day 1, Cycle 5 Day 1 and additional cycles as required. Last visit will be End of Study Treatment. Then continue with FACT-H&N Subscale (HNS) Score, HNS Individual Symptom Score, and FACT-H&N Symptom Index (FHNSI) Score

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment.

PRO assessments obtained at the end of treatment visit or at scheduled timepoints with fewer than 5 subjects in any treatment arm are not included.

Source Data: adam.adgs; Listing 16.2.9.1, 16.2.9.2

Cycle 5 Day 1

Overall

HDC High

XX.X

[xx.x, xx.x]

xx.x [xx.x, xx.x]

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.5.1.2: Statistical Analysis of the Change from Baseline in the FACT-H&N total score, the FACT-H&N HNS, HNS individual symptom score, and the FACT-H&N FHNSI score FACT-H&N Analysis Set

| | | | mean<br>% CI) | Difference between LS means (95% CI) |
|---|---|---|---|---|
| | _ | Patritumab + cetuximab + | Placebo + cetuximab + | · |
| PRO | | cisplatin or carboplatin | cisplatin or carboplatin | |
| Measure | Timepoint | (N=xxx) | (N=xxx) | Patritumab - placebo |
| FACT-H&N<br>total score | Cycle 2 Day 1 | xx.x | XX.X | xx.x |
| total occio | | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| | Cycle 3 Day 1 | xx.x<br>[xx.x, xx.x] | xx.<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |

XX.X

Programming notes: display all timepoints with at least five bser ations per group. Continue with the FACT-H&N HNS, Each of HNS individual symptom score, and the FACT-H&N FHNSI score

XX.X [XX.X, XX.X]

Notes: The mixed model includes treatment, timepoint, treatment x timepoint, and baseline as fixed effects and subject as random effect. If the interaction effect was not significant (p >0.10), the model was rerun without the interaction term and the overall LS mean differences and Cls were estimated. PRO assessments obtained at the end of treatment visit or at scheduled timepoints with fewer than 5 subjects in any treatment arm are not included. The final model [included] [did not include] an interaction term. The xxx covariance structure was used to estimate the interaction model. The xxx covariance structure was used to estimate the final model.

Programming note: Specify in footnote whether final model included an interaction term. Overall LS mean differences are not displayed if the interaction term is significant. Source Data: adam.adqs; Listing 16.2.9.1, 16.2.9.2

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Table 15.5.1.3: Summary of Actual Results and Change from Baseline in EQ-5D Index EQ-5D Analysis Set

HRG High

| PRO Measure<br>Visit | | Patritumab + cetuximab + cisplatin or carboplatin(N=xxx) | | |
|---|---|---|---|---|
| v ion | Result | Change | Result | cxxx)<br>Change |
| Baseline | | <u> </u> | | <u> </u> |
| n | XX | | XX | |
| Mean | XX.X | | XX.X | |
| SD | XX.XX | | xx.xx | |
| Minimum | XX | | XX | |
| Median | XX.X | | XX.X | |
| Maximum | XX | 10 | XX | |
| Cycle 2 Day 1 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | xx.xx | XX.XX | XX.XX |
| Minimum | XX | XX | XX | xx |
| Median | XX.X | XX.X | XX.X | XX.X |
| Maximum | xx | XX | XX | xx |
| Cycle 3 Day 1 | | | | |
| n | X | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | xx | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX |

Notes: The baseline value is defined as the last non-missing value before initial administration of study treatment.

PRO assessments obtained at the end of treatment visit or at scheduled timepoints with fewer than 5 subjects in any treatment arm are not included.

Source Data: adam.adqs; Listing 16.2.9.1, 16.2.9.2 Programming Note: continue for HRG Low and Overall on the next page

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

The following table follows Table 15.5.1.3:

Table 15.5.1.4 Summary of Actual Results and Change from Baseline in VAS Score EQ-5D Analysis Set




<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.1.1 CONSORT Diagram



Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.2.1.1 Kaplan-Meier Plot of Progression Free Survival (PFS) by Treatment Group Full Analysis Set

# HRG High



Source Data: adam.adtte; Listing 16.2.6.1 Programming Note: continue for HRG Low and Overall on the next page

## U31287-A-U203 Statistical Analysis Plan | VV-TMF-2768034 | 1.0

Daiichi Sankyo Pharma Development Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Programming note: Add the legend for different treatment arms in the plot.

Show the timepoint in the survival line when there is censored subject.

Replace the second sentence with "Medications taken on or after the first dose of study medication will be classified as concomitant medications".

The following figure follows Figure 15.2.1.1 and change the label for the y-axis accordingly.

Figure 15.2.1.3 Kaplan-Meier Plot of Progression Free Survival (PFS) for Different HRG Cutoffs by Treatment Group Full Analysis Set

Programming Note: Change the subtitle to "HRG Cutoff: XX; HRG High of Cutoff" and continue for HRG Cutoff: XX; HRG Low of Cutoff XX and HRG Cutoff: XX; Overall of Cutoff XX.

Continue for Different HRG cuteoffs.

Figure 15.2.2.1 Kaplan-Meier Plot of Overall Survival (OS) by Treatment Group Full Analysis Se

Figure 15.2.2.3 Kaplan-Meier Plot of Overall Surv val (O ) for Different HRG Cutoffs by Treatment Group F I Ana ysis Set

Programming Note: Change the subtitle to "HRG Cutoff: XX; HRG High of C toff" a d continue for HRG Cutoff: XX; HRG Low of Cutoff XX and HRG Cutoff: XX; Overall of Cutoff XX. Continue for Different HRG cuteoffs.

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.2.1.2 Forest Plot of Progression Free Survival (PFS) for Selected Subgroups Full Analysis Set



Figure 15.2.3: Waterfall Plot of Best (Minimum) Percent Change in Sum of Longest Diameters from Baseline in Target Lesions Full Analysis Set

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Page x of y <run date time>

# HRG High



Minimum Change (%)

| n | Mean | SD | Median | Minimum | M ximum | n | Mean | SD | Median | Minimum | Maximum |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: For each subject, the minimum percent change from baseline in the sum of Longest Diameters for all target lesions is represented by a vertical line.

Source Data: adam.adrs; Listing xxxx Programming Note: continue for HRG Low and Overall on the next page

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.2.4: Swimmer Plot of Tumor Response and Treatment Duration Full Analysis Set

HRG High

Treatment: Patritumab + cetuximab + cisplatin or carboplatin



<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Source Data: adam.adrs; Listing xxxx

Programming Note: continue for Placebo + cetuximab +cisplatin or carboplatin . Continue for HRG Low.

- 1. Please sort RS by date first then do the best response
- 2. Sort the plot by largest AVAL1. Each subject is a bar.
- 3. Add symbol of CR/PR start date of CR/PR subject (AVAL2).
- 4. Add symbol for status at the end of each bar (STATUS)



Daiichi Sankyo Pharma Development Page x of y Protocol U31287-A-U203 <run date time> 
<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.4.1.1 Mean Plasma Concentration of Patritumab by Time from Sparse PK Sampling Pharmacokinetic Analysis Set



-----Lower limit of quantification (<0.1)

Note: Mean Plasma Concentration data are plotted by C1D1 Pre-Infusion, C1D1 End of Infusion, C2D1 Pre-Infusion, C3D1 Pre-Infusion, C3D1 End of Infusion and End of Tr tment. CxDx = Cycle x Day x

If mean is BLQ, then these are plotted as zero on the linear scale and missing on the semi-log Scale.

Source Data: adam.adpk; Listing 16.2.5.2.1
Figure 15.4.1.2 Mean Plasma Concentration of Patritumab by Time from Intensive PK Sampling Pharamacokinetic Analysis Set



-----Lower limit of quantification (<0.1)

Note: Mean Plasma Concentration data are plotted by 0, 1(EOI), 3, 4, 5, 6, 24, 48, 168, 336 and 504 hours.

CxDx = Cycle x Day x

If mean is BLQ, then these are plotted as zero on the line r scale and missing on the semi-log scale.

Source Data: adam.adpk; Listing 16.2.5.2.1

The following figures follows Figure 15.4.1.2

Figure 15.4.1.3Mean Plasma Concentration of Cetuximab by Time from Intensive PK Sampling Pharmacokinetic Analysis Set

Similar as Table 15.4.1.3, will plot data by hours of 0, 3, 4, 5, 6, 7, 24, 48, and 168.

Figure 15.4.1.4Mean Plasma Concentration of Cisplatin by Time from Intensive PK Sampling Pharmacokinetic Analysis Set

Similar as Table 15.4.1.4, will plot data by hours of 0, 5, 6, 7, 24, and 48.

Figure 15.4.1.5Mean Plasma Concentration of Carboplatin by Time from Intensive PK Sampling Pharmacokinetic Analysis Set

Similar as Table 15.4.1.5, will plot data by hours of 0, 4.5, 5, 6, 7, 24, and 48.



<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.4.2.1 Boxplot of Patritumab PK Parameters at Cycle 1 Pharmacokinetic Analysis Set

HRG High



Source Data: adam.adpk; Listing 16.2.5.2.1

Programming Note: X-axis only presents one treatment group as Patritumab + cetuximab + cisplatin or carboplatin

Y-axis presents AUC<sub>last</sub> (ug.day/mL)
Programming Note: continue for HRG Low and Overall on the next page

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

The following figures follows Figure 15.4.2.1

- Figure 15.4.2.2 Boxplot of Cetuximab PK Parameters at Cycle 1 by Treatment Pharmacokinetic Analysis Set
- Boxplot of Cisplatin PK Parameters at Cyc e 1 by Treatment Figure 15.4.2.3 Pharmacokinetic Analysis Set
- Boxplot of Carboplatin PK Parameters at Cycle 1 by Treatment Figure 15.4.2.4 Pharmacokinetic Analys s Set

Downloaded

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Figure 15.5.1.1 Plot of Cumulative Distribution Function of Change from Baseline on FACT-H&N HNS Score FACT-H&N Analysis Set

**HRG** High



Source Data: adam.adqs; Listing 16.2.9.1, 16.2.9.2

Programming Note: x-axis will be displayed as follows: Cycle 2 Day 1 Change from Baseline; Cycle 3 Day 1 Change from Baseline; Cycle 5 Day

Programming Note: continue for HRG Low and Overall on the next page

Baseline and End-of-Treatment Change from Baseline. X-axis values will range from minimum change to maximum change depending on the data.

Display the legend for the two treatment groups: 

Patritumab + cetuximab + cisplatin or carboplatin

□ Placebo + cetuximab + cisplatin or carboplatin

Figure 15.6.1 Heregulin (HRG) Distribution


Downloaded on 07 Sep 2018

Protocol U31287-A-U203

<run date time>

Page x of y

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Full Analysis Set

**HRG** High

Treatment: Patritumab + cetuximab + cisplatin or carboplatin



Source Data: adam.adxx

Programming Note: X-axis presents heregulin

Y-axis presents frequency (number of people with the heregulin range)
Programming Note: continue for Placebo + cetuximab + cisplatin or carboplatin and continue for HRG Low and Overall on the next page

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

## Listing 16.2.1.1: Subject Disposition All Screen Subjects

| Subject ID/<br>Group/Age/<br>Gender | Screen Fail/<br>Reason | First Dose Date of<br>Patritumab/<br>Cetuximab/<br>Cisplatin/Capboplatin | Last Dose Date (Day) of<br>Patritumab/<br>Cetuximab/<br>Cisplatin/Capboplatin | Primary Reason for<br>Discontinuation<br>from Study<br>Treatment | Primary Reason for<br>Discontinuation<br>from Extension<br>Treatment | Follow-up<br>Contact<br>Date | Started New<br>Cancer<br>Treatment |
|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin /xx/M | No | yyyy-mm-dd/<br>yyyy-mm-dd/<br>yyyy-mm-dd | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | Completed | xxx xxxxxxx | yyyy-mm-dd (xx) | No |
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin /xx/M | No | yyyy-mm-dd/<br>yyyy-mm-dd/<br>yyyy-mm-dd | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | xxxxxxxxxx | Did not continue in Ext | yyyy-mm-dd (xx) | Yes – yyyy-mm-dd |
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin /xx/M | Yes – xxxxxxxx x | | 36.b | | | | |

Source: adam.adsl

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.1.2: Deaths Full Analysis Set

| HRG High | | | | |
|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | First Dose Date of<br>Patritumab/<br>Cetuximab/<br>Cisplatin/Capboplatin | Last Dose Date (Day) of<br>Patritumab/<br>Cetuximab/<br>Cisplatin/Capboplatin | Death Date<br>(Day) | Primary Cause of Death |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/M | yyyy-mm-dd/ | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/M | yyyy-mm-dd/<br>yyyy-mm-dd/<br>yyyy-mm-dd | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | 10 | |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/M | | | 0 | |
| | | NOB | | |

Source: adam.adsl

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.2.1: Inclusion/Exclusion Criteria All Screen Subjects

**HRG High** Subject ID/

Group/Age/ Gender

Inclusion/Exclusion

Assessment Date

Failed Inclusion/Exclusion If Yes, Specify Criteria [a]

1, 2, x

Criteria

xxxxxx/

No

Yes

yyyy-mm-dd

Patritumab+

cetuximab + cisplatin or carboplatin /xx/M

xxxxxx/

yyyy-mm-dd

Patritumab+ cetuximab + cisplatin

or carboplatin /xx/M

xxxxxx/

Patritumab+ cetuximab + cisplatin or carboplatin /xx/M

yyyy-mm-dd

Notes: [a] See appended pages of this listing for a complete list of the inclusion and exclusion criteria from Protocol Version 2.0.

Source: adam.adie, Protocol U31287-A-U203 Version 2.0 (27Aug2015)

Programming note: Append next 2 pages to end of this listing.

Programming Note: continue for HRG Low and Overall on the next page


Daiichi Sankyo Pharma Development Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.2.1: Inclusion Criteria

Subjects must satisfy all of the following criteria to be included in the study:

1

2

...



Source: adam.adie, Protocol U31287-A-U203 Version 2.0 (27Aug2015)

Programming note: list all inclusion criteria from the protocol.


Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.2.1: Exclusion Criteria

Subjects who meet any of the following criteria will not be included in the study:

'

2

...



Source: adam.adie, Protocol U31287-A-U203 Version 2.0 (27Aug2015)

Programming note: list all exclusion criteria from the protocol.


Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y font

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.2.2: Informed Consent Full Analysis Set

| HRG High<br>Subject ID/<br>Group/Age/<br>Gender | Study Informed<br>Consent Date (Day) | Consented to Pharmacogenomic Sampling | Sample Taken for<br>Pharmacogenomic/<br>Date (Day) | Consented to<br>Tumor Tissue Sampling | Sample Taken for<br>Tumor Tissue/<br>Date (Day) |
|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab<br>+ cisplatin or<br>carboplatin /xx/M | yyyy-mm-dd (xx) | Yes | Yes – yyyy-mm-dd (xx) | Yes | Yes – yyyy-mm-dd (xx) |
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin /xx/M xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin /xx/M | | No | 401 | 20 | |
| | | 52 | | | |

Source: adam.adsl, adam.adpg

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Source [a]

**ICOTRIAL** 

**CRF** 

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.2.3: Protocol Deviation Full Analysis Set

HRG High

| Group/Age/<br>Gender | Date of Deviation (Day) | Deviation Class | Deviation Text |
|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab | yyyy-mm-dd (xx) | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| + cisplatin or carboplatin /xx/M | | | |

XXXXXXXXXXXXXXXX

xxxxxx/ Patritumab+ cetuximab

+ cisplatin or carboplatin /xx/M

xxxxxx/

Patritumab+ cetuximab

+ cisplatin or carboplatin /xx/M

Note: [a] ICOTRIAL deviations are obtained from the clinical monitoring database. CRF deviations are derived using CRF data.

Source: adam.addv, ICOTRIAL

Need to confirm if programmed deviations from CRF data is needed.

Programming Note: continue for HRG Low and Overall on the next page

yyyy-mm-dd (xx)

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.3: Subject Inclusion in Analysis Sets Full Analysis Set

| HRG High<br>Subject ID/<br>Group/Age/<br>Gender | Safety Analysis Set | DLT Evaluable Set | Pharmacokinetic Analysis Set |
|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/M | Yes | No – Did not receive 80% of cetuximab | Yes |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/M | No – Not Dosed | No – Not Dosed | No No |

Source: adam.adsl

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.1: Demographic Data Full Analysis Set

HRG High

| Subject ID/Group | Date of<br>Birth | Study Informed<br>Consent Date (Day) | Age<br>(yrs) [a] | Gender | Ethnicity | Race | Height<br>(cm) | Baseline<br>Weight<br>(kg) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/Patritumab+<br>cetuximab + cisplatin or<br>carboplatin | yyyy-mm-dd | yyyy-mm-dd (xx) | xx | M | Hispanic/Latino | xxxxxxxxx | xxx.x | xxx.x |
| xxxxxx/Patritumab+<br>cetuximab + cisplatin or<br>carboplatin | yyyy-mm-dd | yyyy-mm-dd (xx) | xx | F | Non Hispanic/Non Latino | xxxxxxxx | xxx.x | xxx.x |
| xxxxxx/Patritumab+<br>cetuximab + cisplatin or<br>carboplatin | yyyy-mm-dd | yyyy-mm-dd (xx) | xx | М | Hispanic/Latino | Other: xxxxxxxxx | XXX.X | XXX.X |

Notes: [a] Age is calculated as the number of complete years between date of birth and date of informed consent.

Source: adam.adsl

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.2: Pregnancy Test Results Full Analysis Set

| HRG High | | | | | |
|---|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | Visit | Pregnancy<br>Test Done? | Date of Test<br>(Day) | Method | Result |
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin /xx/F | Screening | Yes | yyyy-mm-dd (xx) | Urine | Negative |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/F | Screening | No | | 018 | |

Source: adam.adlb

Daiichi Sankyo Pharma Development Protocol U31287-A-U203 Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.3: Medical/Surgical History
Full Analysis Set

| HRG High | | | |
|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | Event/Diagnosis | Onset Date<br>(Day) | Continuing |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/F | xxxxxxxxxxxxxxxx | yyyy-mm-dd (xxx) | Yes |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin<br>/xx/F | xxxxxxxxxxxxxxxx | yyyy-mm-dd (xxx) | No |

Source: adam.admh

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.4.1: Cancer History for SCCHN Full Analysis Set

**HRG** High

| Subject ID/<br>Group/Age/<br>Gender | Cancer<br>Type | Histology | Date of Initial<br>Histologic<br>Diagnosis | Time from<br>Initial Diagnosis to<br>Study Treatment<br>(Months) [a] | Tumor Staging<br>at Study<br>Entry | Grade | Date of<br>Biopsy | Anatomical<br>Location | Type of Biopsy |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin /<br>xx/F | xxxxx | xxxxxx | yyyy-mm-dd | xxx | IA | Well Differentiated | yyyy-mm-dd | xxxxxxxxx | FNAB |
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin/<br>xx/M | XXXXXXX | xxxxxxx | yyyy-mm-dd | xxx | IIB | Mod rat ly<br>Differentiated | yyyy-mm-dd | xxxxxxxxx | Core Needle |
| | | xxxxxxxx | yyyy-mm-dd | xxx | Oth r: xxx | Undifferentiated | yyyy-mm-dd | xxxxxxxxx | Surgery: xxx |
| | | xxxxxxxxxx | yyyy-mm-dd | xxx | V | Moderately<br>Differentiated | yyyy-mm-dd | xxxxxxxxx | Excisional |

Notes: [a] Time from initial diagnosis to study treatment = (date of initial administration of any study treatment – date of diagnosis + 1)/365.25x12.

Source: adam.admh

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.4.2: Prior Head and Neck Systemic Cancer Therapy
Full Analysis Set

HRG High

| Subject ID/<br>Group/Age/<br>Gender | Intended for | Best Response [a] | Agent Name | Start Date | Stop Date |
|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin /<br>xx/F | xxxxxxx | PR | xxxxx | yyyy-mm-dd | yyyy-mm-dd |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin /<br>xx/M | xxxxxxx | CR | xxxxxxxx | yyyy-mm-dd | yyyy-mm-dd |
| | | SD | xxxxxxx | yyyy-mm-dd | yyyy-mm-dd |
| | | PD | xxxxxx | yyyy-mm-dd | yyyy-mm-dd |

Note: [a] CR=Complete Response; PR=Partial Response; SD=Stable Disease; PD=Progressive Disease; NA=Not Applicable

Source: adam.adcm

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.4.4.3: Prior Radiation Therapy Full Analysis Set

|--|

| пко підп | | | | | |
|---|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | Any Prior Radiation<br>Therapy | Indication | Start Date | End Date | Location |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | Yes | xxxxxxxxxxxxx | yyyy-mm-dd | yyyy-mm-dd | xxxxxxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/M | Yes | xxxxxxxxxxxxx | yyyy-mm-dd | yyyy-mm-dd | xxxxxxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/M | No | | ~~~ | | |

Source: adam.adcm

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

# Listing 16.2.4.5: Prior/Concomitant Medication Safety Analysis Set

**HRG** High

| - 1 11 (O 1 11g) 1 | | | | | |
|---|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | C: Class<br>W: WHO Drug Term<br>V: Verbatim Name | S: Start Date (Day)<br>E: Stop Date (Day)<br>O: Ongoing | Dose (Units) | Frequency | Indication |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | C: xxxxxxxxxxxx<br>W: xxxxxxxxxxxx<br>V: xxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E:<br>O: Yes | xxxxxxx (Other/xxxx) | xxxxxxxxxx | xxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/M | C: xxxxxxxxxxxxx<br>W: xxxxxxxxxxxxx<br>V: xxxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E: yyyy-mm-dd (xxx)<br>O: No | xxxxxxx (xxxx) | xxxxxxxxx | xxxxxxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | C: xxxxxxxxxxxx<br>W: xxxxxxxxxxxx<br>V: xxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E: yyyy-mm-dd (xxx)<br>O: No | xxxx xx (xxxx) | xxxxxxx | xxxxxxxxxx |

Source: adam.adcm

Daiichi Sankyo Pharma Development Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

### Listing 16.2.4.6: Non-Drug Treatment/Procedures Safety Analysis Set

| HRG High | | | | |
|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | Treatment/Procedure | S: Start Date (Day)<br>E: End Date ( Day)<br>O: Ongoing | Duration | Indication |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | xxxxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E: yyyy-mm-dd (xxx)<br>O: No: | xxx | xxxxxxxxxx |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/M | xxxxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E:<br>O: Yes | XXX | xxxxxxxxxx |

Source: adam.adcm

Programming Note: continue for HRG Low and Overall on the next page


Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

#### Listing 16.2.5.1.1: Investigational Drug Patritumab Administration Safety Analysis Set

HRG High

| Subject ID/<br>Group/Age/<br>Gender | Visit | Date of Infusion<br>(Day) | Start Time/<br>Stop Time | Dose Level<br>(mg/kg) | Actual Total Dose<br>Administered<br>(mg/kg) | Was IV<br>Completed? | Reason for Change or<br>Interruption |
|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/xx/F | Cycle 1 Day 1 | yyyy-mm-dd (xx) | hh:mm/hh:mm | xx | xx | No | XXX |
| xxxxxx/<br>Patritumab+ cetuximab + | Cycle 1 Day 1 | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx | хх | Yes | xxx |
| cisplatin or carboplatin/xx/M | Cycle x Day 1 | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx | xx | Yes | xxx |

Source: adam.adex

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y fondate time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

# Listing 16.2.5.1.2: Cetuximab, Cisplatin, and Carboplatin Administration Safety Analysis Set

**HRG High** 

| Subject ID/ | | | | | | Actual Total Dose | | |
|---|---|---|---|---|---|---|---|---|
| Group/Age/<br>Gender | Visit | Study Drug | Date of Infusion (Day) | Start Time/<br>Stop Time | Dose Level (unit) | Administered (unit) | Was IV Completed? | Reason for Change or<br>Interruption |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/xx/F | Cycle 1 Day 1 | Cetuximab | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx (mg/m2) | xx (mg/m2) | No | xxx |
| carbopiatiri | | Cisplatin | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx (mg/m2) | xx (mg/m2) | Yes | XXX |
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/xx/M | Cycle 1 Day 1 | Cetuximab | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx (mg m2 | xx (mg/m2) | Yes | xxx |
| 33.23p.atii 1770 iii | | Carboplatin | yyyy-mm-dd (xx) | hh:mm/ hh:mm | xx (mg) | xx (mg) | Yes | xxx |

Source: adam.adex

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.5.1.3: Patritumab, Cetuximab, and Cisplatin/Carboplatin Exposure Safety Analysis Set

| HRG | Hiah |
|-----|------|

| Subject ID/<br>Group/Age/<br>Gender | Study Drug | Treatment Duration (Weeks) [a] | Treatment Duration (Cycles) [a] | Number of IV<br>Received | Cumulative Dose (unit) [b] |
|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/xx/F | Patritumab | xx.x | XX.X | xx | xxx (mg/kg) |
| al bopiati ii xuu i | Cetuximab<br>Cisplatin/Carboplatin | XX.X<br>XX.X | XX.X<br>XX.X | xx<br>xx | xxx (mg/m2)<br>xxx (mg/m2) / xxx (mg) |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/xx/M | | | 30 | | |

Notes: [a] Treatment duration (in weeks) for Patritumab and Cisplatin/Carboplatin is calculated as (date of the last dose – date of the first dose + 21)/7.

Treatment duration (in cycles) for Patritumab and Cisplatin/Carboplatin is calculated as (date of the last dose – date of the first dose + 21)/21.

Treatment duration (in weeks) for Cetuximab is calculated as (date of the last dose – date of the first dose + 7)/7.

Treatment duration (in cycles) for Cetuximab is calculated as (date of the last dose – date of the first dose + 7)/21.

[b] Total cumulative dose is the sum of doses taken by a subject across cycles.

Source: adam.adex

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.5.2.1: Patritumab Pharmacokinetic Sample Collection Time and Results
Pharmacokinetic Analysis Set

| Subject ID/<br>Group/Age/<br>Gender | Visit | Patritumab Infusion<br>Date Start Time/<br>Stop Time (Day) | Nominal<br>Time Point [a] | PK<br>Sample<br>Taken | Date/Time of Sample<br>Collection (Day) | Sample<br>Identification<br>Number | Result<br>(unit) | Excluded from<br>Analysis:<br>Reason if Y | AUC_0-21d<br>C_max |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/xx/F | C1D1 | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | Pre-Infusion | Yes | yyyy-mm-dd hh:mm (xx) | xxxxx | xxxxx | N | xxx.x/xxxx.x |
| | | | 1 h | Yes | yyyy-mm-dd hh:mm (xx) | xxxxx | xxxxxx | N | |
| | | | 3 h | Yes | yyyy-mm-dd hh:mm (xx) | xx xx | xxxxxx | Y:xxxxxxx | |
| | | | 4 h | No | yyyy-mm-dd hh:mm (xx) | XXXXX | XXXXXX | N | |
| | | | 5 h | | yyyy-mm-dd hh:mm (xx) | XXXXX | XXXXXX | N | |
| | C1D2 | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | 24 h | | yyyy-mm-dd h :mm (xx) | XXXXX | XXXXXX | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyyy mm-dd hh mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yy y-mm-dd hh:mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyy-mm-dd hh:mm (xx) | XXXXX | xxxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | N | yyyy-mm-dd hh:mm (xx) | XXXXX | xxxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | xx | O> | yyyy-mm-dd hh:mm (xx) | xxxxx | XXXXXX | N | |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or | | | | | | | | | |

Notes: [a] All nominal time points are relative to the end of infusion except for pre-infusion.

Source: adam.adpk

Programming Note: List scheduled times as shown in table 8.1 of the protocol. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.5.2.2: Cetuximab Pharmacokinetic Sample Collection Time and Results Pharmacokinetic Analysis Set

| Н | RG | Н | iα | r |
|---|----|---|----|---|

| Subject ID/<br>Group/Age/ | | Cetuximab Infusion<br>Date Start Time/ | Nominal | PK<br>Sample | Date/Time of Sample | Sample<br>Identification | Result | Excluded from<br>Analysis: | AUC_0-21d |
|---|---|---|---|---|---|---|---|---|---|
| Gender | Visit | Stop Time (Day) | Time Point [a] | Taken | Collection (Day) | Number | (unit) | Reason if Y | C_max |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/xx/F | C1D1 | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | Pre-Infusion | Yes | yyyy-mm-dd hh:mm (xx) | xxxxx | xxxxxx | N | xxx.x/xxxx.x |
| | | | 3 h | Yes | yyyy-mm-dd hh:mm (xx) | XXXX | XXXXXX | Y:xxxxxxx | |
| | | | 4 h | Yes | yyyy-mm-dd hh:mm (xx) | xx xx | XXXXXX | N | |
| | | | 5 h | No | yyyy-mm-dd hh:mm ( x) | XXXXX | XXXXXX | N | |
| | C1D2 | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | 24 h | | yyyy-mm-dd hh:mm (xx) | xxxxx | XXXXXX | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyyy-mm dd hh:mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyyy-mm dd hh:mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyyy mm-dd hh:mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | XX | | yyyy-mm-dd hh:mm (xx) | XXXXX | xxxxx | N | |
| | XX | yyyy-mm-dd<br>hh:mm/hh:mm (xx) | xx | JK | yyyy-mm-dd hh:mm (xx) | XXXXX | XXXXXX | N | |
| xxxxxx/<br>Placebo+<br>cetuximab +<br>cisplatin or | | | | | | | | | |

carboplatin/xx/F

Notes: [a] All nominal time points are relative to the end of infusion except for pre-infusion.

Source: adam.adpk

Programming Note: List scheduled times as shown in table 8.1 of the protocol. Programming Note: continue for HRG Low and Overall on the next page.

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

The following listings follow Table 16.2.5.2.2:

Listing 16.2.5.2.3: Patritumab Pharmacokinetic Sample Collection Time and Results

Listing 16.2.5.2.4: Cetuximab Pharmacokinetic Sample Collection Time and Results




Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

### Listing 16.2.6.1.1: Target Tumor Assessment Full Analysis Set

| HRG High | | | | | | |
|---|---|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | Lesion<br>Number | Location | Visit | Assessment Date (Day) | Assessment<br>Method | Longest Diameter<br>(mm) [a] |
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/ xx/F | 1 | xxxxxxxxx | Screening | yyyy-mm-dd (xxx) | Spiral CT Scan | xxx |
| *** | | | Cycle x | yyyy-mm-dd (xxx) | Spiral CT Scan | xxx |
| | 2 | Other (xxxxxxxxx) | Screening<br>Cycle x | yyyy-mm dd (xx )<br>yyyy-mm-dd (xxx) | Spiral CT Scan<br>Spiral CT Scan | xxx<br>xxx |
| | SUM LD | | Screening<br>Cycle x | yyyy-mm-dd (xxx)<br>yyyy mm-dd (xxx) | | xxx<br>xxx |
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/ xx/M | x | xxxxxxxxx | Screening | yyy-mm-dd (xxx) | xxxxxxxxxxx | xxx |
| AAIVI | x<br>x | xxxxxxxxxx | Cy le x<br>Cycle x | yyyy-mm-dd (xxx)<br>yyyy-mm-dd (xxx) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX<br>XXX |

Notes: [a] Shortest for lymph nodes. SUM LD = Sum of longest diameters.

Source: adam.adtm

Programming note: sort by subject ID, lesion number, and visit.

Daiichi Sankyo Pharma Development Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.6.1.2: Non-Target Tumor Assessment Full Analysis Set

HRG High

| Subject ID/<br>Group/Age/<br>Gender | Lesion<br>Number | Location | Visit | Assessment Date (Day) | Assessment<br>Method | Status |
|---|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/xx/F | 1 | xxxxxxxxx | Screening | yyyy-mm-dd (xxx) | Spiral CT Scan | Present |
| | | | Cycle x | yyyy-mm-dd (xxx | Spiral CT Scan | Absent |
| | 2 | Other (xxxxxxxx) | Screening<br>Cycle x | yyyy-mm-dd (xxx)<br>yyyy-mm-dd (xxx) | Spiral CT Scan<br>Spiral CT Scan | XXX<br>XXX |
| xxxxxx/ | x | xxxxxxxxx | Screening | yyyy-mm-dd (xxx) | xxxxxxxxxxx | XXX |
| Patritumab+ cetuximab + cisplatin or | | | Ü | | | |
| carboplatin/xx/M | Х | xxxxxxxxx | Cycle x | yyyy-mm-dd (xxx) | xxxxxxxxxxx | xxx |
| | X | XXXXXXXXX | Cycle x | yyy-mm-dd (xxx) | XXXXXXXXXXX | New |

Source: adam.adtm

Programming note: sort by subject ID, lesion number, and visit.

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.6.1.3: Overall Tumor Assessment Full Analysis Set

| HRG High Subject ID/ Group/Age/ Gender | Visit | Tumor Response<br>Assessment<br>Performed? | Date of Overall<br>Response<br>(Day) | Target Lesion<br>Overall Evaluation | Non-Target<br>Lesion Overall<br>Evaluation | Overall<br>Evaluation |
|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab + cisplatin or carboplatin/ | Cycle x | Yes | yyyy-mm-dd (xxx) | Partial Response | Non-CR/Non-PD | Partial Response |
| xx/F | Cycle x<br>Cycle x | Yes<br>No | yyyy-mm-dd (xxx) | Partial Response | Complete Response | Partial Response |
| | Cycle x | Yes | yyyy-mm-dd (xxx) | Stable Disease | Non-CR/Non-PD | Stable Disease |

Source: adam.adrs

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y fun date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.6.2: Progression-Free Survival and Overall Survival Full Analysis Set

**HRG High** 

| Subject ID/<br>Group/Age/<br>Gender | Randomization<br>Date (Day) | Date of<br>Last Tumor<br>Assessment<br>(Day) | Date of<br>Last Contact<br>When Alive<br>(Day) | Radiographic<br>Progression?/<br>Date of<br>Progression<br>(Day) | Death?/<br>Date of Death<br>(Day) | Progression<br>Free Survival<br>(Days) [a] | Overall<br>Survival<br>(Days) [b] | Time to Disease<br>Progression<br>(Days) [c] |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/ xx/F | YYYY-MM-DD<br>(xx) | YYYY-MM-DD<br>(xxx) | YYYY-MM-DD<br>(xxx) | No | Yes/YYYY-MM-DD<br>(xxx) | xxx | xxx | xxx |
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin/<br>xx/M | | | YYYY-MM-DD<br>(xxx) | No | No | 1 (C) | xxx (C) | 1 (C) |

Notes: (C) = censored observation

[a] PFS is defined as the time from the date of randomization the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1 as assessed by investigator) or death due to any cause. See the SAP for censoring rules.

Source: adam.adtte

<sup>[</sup>b] OS is defined as the time from the randomization date to the d te of death. If there is no death reported for a subject before the cut-off date for OS analysis, OS is censored at the last contact date at which the subject is known to be alive

<sup>[</sup>c] Time to disease progression is defined as the time from the randomization date to the date of first objective documentation of radiographic disease progression (per RECIST v1.1 as assessed by investigator). See the SAP for censoring rules

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.6.3: Subjects with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) Full Analysis Set

#### HRG High

| Subject ID/Group/Age/Gender | Best<br>Overall<br>Response | Date of Earliest<br>Response<br>(Day) | Radiographic<br>Progression?/<br>Date of<br>Progression<br>(Day) | Date of<br>Last Tumor<br>Assessment<br>(Day) | Duration of<br>Response<br>(Weeks) [a] | Time to<br>Response<br>(Weeks) [b] | Duration of<br>SD<br>(Weeks) [c] |
|---|---|---|---|---|---|---|---|
| xxxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/ xx/F | PR | YYYY-MM-DD<br>(xxx) | Yes/YYYY-MM-<br>DD (xxx) | YYYY-MM-DD<br>(xxx) | xxx | xxx | xxx |
| xxxxxx/<br>Patritumab+ cetuximab + cisplatin or<br>carboplatin/<br>xx/F | CR | YYYY-MM-DD<br>(xxx) | No | YYYY-MM-DD<br>(xxx) | xxx (C) | xxx | xxx (C) |
| xxxxxx/<br>Placebo + cetuximab + cisplatin or<br>carboplatin/<br>xx/M | SD | DDMMMYYYY<br>(xxx) | Yes/<br>DMMMYYYY<br>(xxx) | DDMMMYYYY<br>(xxx) | | | xxx |

Notes: (C) = censored observation

- [a] Duration of response is defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease (disease progression as assessed based upon tumor measurements and recorded on the CRF page "overall tumor assessment"). See the SAP for censoring rules. [b] Time to response is defined as the time from the randomization date to the date of the first documentation of objective response (CR or PR).
- [c] Duration of SD is defined for subjects whose best response is SD as the time from the date of randomization to the date of the first documentation of progressive disease (disease progression as assessed based upon tumor measurements and recorded on the CRF page "overall tumor assessment"). See the SAP for censoring rules.

Source: adam.adtte

#### Programming notes:

Sort by best overall response.

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.7.1: Adverse Events Safety Analysis Set

| HP | $\sim$ | ш | :~ ٢ |
|----|--------|---|------|

| HRG High | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID/<br>Group/Age/<br>Gender | TEAE? | S: Class<br>P: Preferred Term<br>V: Verbatim | S: Start Date (Day)<br>E: Stop Date (Day)<br>O: Ongoing | NCI<br>CTCAE<br>Grade | SAE? | DLT? | Causality Pa: Patritumab Ce: Cetuximab Ci: Cisplatin Ca: Carboplatin | Action [a] Pa: Patritumab Ce: Cetuximab Ci: Cisplatin Ca: Carboplatin | Outcome [b] | Other Action [c] |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/<br>xx/F | Yes | S: xxxxxxxxxxxx<br>P: xxxxxxxxxxxx<br>V: xxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E:<br>O: Yes | x | Yes | Yes | Related to Pa | Pa: xx<br>Ce: xx | xx | x |
| | Yes | S: xxxxxxxxxxxx<br>P: xxxxxxxxxxxx<br>V: xxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E:<br>O: Yes | x | Yes | Yes | Related to Ci | Pa: xx<br>Ce: xx | xx | х |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/<br>xx/M | Yes | S: xxxxxxxxxxxxxxxx P: xxxxxxxxxxxxxxxxx | S: yyyy-mm-dd (xxx)<br>E: yyyy-mm-dd (xxx)<br>O: No | x | No | es | Related to Pa and Ca | Pa: xx<br>Ce: xx | xx | 0 |

Notes: [a] Action Taken: N = Dose Not Changed, W = Drug Withdrawn, R = Dose Reduced, INT = Drug Interrupted

Source: adam.adae

<sup>[</sup>b] Outcome: R = Recovered/Resolved, RS = Recovered/Resolved with Sequelae, F = Fatal, NR = Not Recovered/Not Resolved, UNK = Unknown

<sup>[</sup>c] Other Action: N = None, M = Medication Required, H = Hospitalization or prolongation of hospitalization required, O = Other

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

These Appendices follow Listing 16.2.7.1:

Listing 16.2.7.2: Serious Adverse Events, Including Those Leading to Deaths Safety Analysis Set

Listing 16.2.7.3: Adverse Events Leading to Study Drug Discontinuation Safety Analysis Set

Listing 16.2.7.4: Adverse Event Leading to Study Drug Interrupti n or Dose Reduction Safety Analysis Set

Listing 16.2.7.5: Adverse Events o Interests Safety Analysi Set


Downloaded

on 07 Sep 2018

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.1.1: Laboratory Data – Hematology Safety Analysis Set

HRG High

| Subject ID/<br>Group/Age/<br>Gender | Lab Name | Parameter<br>(Standard Units) | Visit | Date/Time<br>of Sample<br>(Day) | Result<br>[a] | Normal<br>Limits | Change<br>from<br>Baseline | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin/<br>xx/F | xxxxxxxxx | Test #1 (xxxxx) | Screening | yyyy-mm-dd hh:mm (xx) | xxxx | XXXX-XXXX | | |
| 7001 | | | CxDx | yyyy-mm-dd hh:mm (xx) | xxxx (H) | xxxx-xxxx | xxxx | х |
| | | | CxDx | yyyy-mm-dd hh:mm (xx) | xxxx | XXXX-XXXX | XXXX | |
| | | | CxDx | yyyy-mm-dd hh:mm (xx) | XXXX | XXXX-XXXX | xxxx | |
| | | Test #2 (xxxxx) | Screening | yyyy-mm-dd hh:mm (xx) | XXXX | xxxx-xxxx | | |
| | | | CxDx | yyyy-m -dd hh:mm (xx) | XXXX | XXXX-XXXX | XXXX | |
| | | | CxDx | yyyy-mm-dd h:mm (xx) | XXXX | XXXX-XXXX | XXXX | |

Notes: [a] H = Abnormally High, L = Abnormally Low

Source: adam.adlb
Daiichi Sankyo Pharma Development Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

These Appendices follow Listing 16.2.8.1.1:

Listing 16.2.8.1.2: Laboratory Data – Chemistry Safety Analysis Set

Listing 16.2.8.1.3: Laboratory Data – Urinalysis Safety Analysis Set

Programming Notes: Remove Change from baseline and CTC grade columns for urinalysis.

Listing 16.2.8.1.4: Laboratory Data – Coagulat on Safety Analysis Set

Listing 16.2.8.2.1: Clinically Significant Laboratory Abnormalities or Abnormalities of CTCAE Grade 3 or 4 – Hematology Safety Analysis Set

Listing 16.2.8.2.2: Clinically Significant Laboratory Abnormalities or Abnormalities of CTCAE Grade 3 or 4 – Chemistry Safety Analysis Set


## U31287-A-U203 Statistical Analysis Plan | VV-TMF-2768034 | 1.0

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y fondate time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.2.3 Subjects with Liver Enzymes (ALT, AST) and Total Bilirubin (TBL) Elevation Safety Analysis Set

| Subject ID/<br>Group/Age/<br>Gender | Investigator/<br>Country/Site | Visit | Date/Time<br>of Sample<br>(Day) | AST<br>(xxx-xxx) [a] | ALT<br>(xxx-xxx) [a] | Total<br>Bilirubin<br>(xxx-xxx) [a] | ALP<br>(xxx-xxx) [a] |
|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+<br>cetuximab + cisplatin<br>or carboplatin/<br>xx/F | XXXXXXXXXX | Screening | yyyy-mm-dd hh:mm (xx) | xxxx | XXXX | xxxx-xxxx | xxxx |
| | | CxDx<br>CxDx | yyyy-mm-dd hh:mm (xx)<br>yyyy-mm-dd hh:mm (xx) | xxxx (H) | xxxx (H) | XXXX-XXXX<br>XXXX-XXXX | xxxx (H)<br>xxxx |
| | | CxDx | yyyy-mm-dd hh:mm (xx) | XXXX | xxxx | XXXX-XXXX | XXXX |

Notes: [a] H = Abnormally High, L = Abnormally Low

Source: adam.adlb

Programming Note: continue for HRG Low and Overall on the next page


Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.3.1: Vital Signs Safety Analysis Set

HRG High

| Subject ID/<br>Group/Age/<br>Gender | Visit | Time Point | Date of Vital Sign<br>Assessment<br>(Day) | Weight<br>(kg) | Pulse Rate<br>(beat/min) | Systolic BP (mmHg) | Diastolic BP<br>(mmHg) | Temperature (C) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/ xx/F | Screening | | yyyy-mm-dd (xx) | xxx.x | xxx | xxx | xxx | XXX.X |
| W.F | C1D1 | Pre-Infusion | yyyy-mm-dd (xx) | xxx.x | xxx | xxx | xxx | XXX.X |
| | C1D1<br>C1D8 | End of Infusion | yyyy-mm-dd (xx)<br>yyyy-mm-dd (xx) | XXX.X | XXX | XXX | XXX | XXX.X |
| | C1D15 | | yyyy-mm-dd (xx) | XXX.X | XXX | XXX | XXX | XXX.X |
| | CxDx | | yyyy-mm-dd (xx) | XXX.X | XXX | XXX | XXX | XXX.X |
| | EOT | | yyyy-mm-dd (xx) | XXX X | XX | XXX | XXX | XXX.X |

Source: adam.advs

Programming note: Time point will be missing for every visit except C1D1. Programming Note: continue for HRG Low and Overall on the next page

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.3.2: 12-Lead ECG Safety Analysis Set

HRG High

| HRG High | | | | | |
|---|---|---|---|---|---|
| Subject<br>ID/Group/Age/<br>Sex | Visit | Date of ECG Assessment (Day) | ECG<br>Interpretation | Heart Rate<br>(beats/min) | ECG Intervals (msec) |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/<br>xx/F | Screening | yyyy-mm-dd (xx) | Normal | xxx | PR: xx<br>RR: xx<br>QRS: xxx<br>QT: xxx<br>QTcB: xxx<br>QTcF: xxx |
| xxxxxx/<br>Patritumab+<br>cetuximab +<br>cisplatin or<br>carboplatin/<br>xx/M | Screening | yyyy-mm-dd (xx) | Abnormal, not clinically significant | XXX | PR: xx<br>RR: xx<br>QRS: xxx<br>QT: xxx<br>QTcB: xxx<br>QTcF: xxx |

QTcB = QTc by Bazett's Correction Formula (msec); QTcF = QTc by Fridericia's Correction Formula (msec)

Source: adam.adeg

Programming Note: continue for HRG Low and Overall on the next page


## U31287-A-U203 Statistical Analysis Plan | VV-TMF-2768034 | 1.0

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.3.3: Physical Examination Safety Analysis Set

#### HRG High

| Subject ID/<br>Group/Age/Gender | Visit | Physical Exam Status | Date of Exam<br>(Day) | Body System | Description of<br>Findings |
|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab | Screening | No clinically significant findings | yyyy-mm-dd (xx) | xxxxxxxxxxxx | xxxxxxxxxxxxxx |
| - cisplatin or<br>carboplatin/xx/F | | | | xxxxxxxxxxxx | xxxxxxxxxxxx |
| | | | | XXXXXXXX XXXXXX | XXXXXX |
| | | | | XXXXXXXXXX XXXX | xxxxxxxxxx |
| | | | | XXXXX XXXXXXXXX<br>XXXXXXXXXXXXXX | XXXXXXXXXX |
| | | | | XXXXXXXXXXXXX | XXXXXX |
| | CxDx | Clinically significant changes | yyyy-mm-dd (xx) | | |
| exxxxx/<br>Patritumab+ cetuximab<br>- cisplatin or | Screening | No clinically significant findings | yyyy-mm dd (xx) | xxxxxxxxxxxx | |
| carboplatin/xx/M | | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| | CxDx | Not Done | | *************************************** | |

Source: adam.adpe

Protocol U31287-A-U203

Page x of y cprogname> <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.3.4: Eastern Cooperative Oncology Group (ECOG) Performance Status Safety Analysis Set

| HRG High | | | | |
|---|---|---|---|---|
| Subject ID/<br>Group/Age/Gender | Visit | ECOG<br>Assessed? | Date of ECOG<br>Assessment (Day) | ECOG Score [a] |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/xx/F | Screening | Yes | yyyy-mm-dd (xxx) | x |
| xxxxxx/<br>Patritumab + cetuximab +<br>cisplatin or carboplatin<br>/xx/M | Screening | Yes | yyyy-mm-dd (xxx) | x |
| 7AATWI | CxDx | Yes | yyyy-mm-dd (xxx) | X |
| xxxxxx/ Patritumab + cetuximab + cisplatin or carboplatin/xx/F | Screening | Yes | yyyy-mm-dd (xxx) | х |
| Cispiani di Calbopani/XVI | CxDx | No | yyyy-mm-dd (xxx) | х |

Notes: [a] 0 = Fully active, able to carry on all pre-disease performance without restriction;

5 = Dead.

Source: adam.adgs

<sup>1=</sup> Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature;

<sup>2 =</sup> Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours;

<sup>3 =</sup> Capable of only limited self-care, confined to bed or chair more than 50% of waking hours;

<sup>4 =</sup> Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair;

## U31287-A-U203 Statistical Analysis Plan | VV-TMF-2768034 | 1.0

Daiichi Sankyo Pharma Development

Protocol U31287-A-U203

Page x of y fondate time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.3.5: Echocardiogram Safety Analysis Set

**HRG High** 

| Subject ID/<br>Group/Age/Gender | Visit | ECHO or MUGA<br>Scan Completed? | Date Procedure Performed (Day) | Type of Assessment | Left Ventricular Ejection Fraction (LVEF) (%) |
|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab<br>+ cisplatin or<br>carboplatin/<br>xx/F | Screening | Yes | yyyy-mm-dd (xx) | ЕСНО | XX.X |
| xxxxxx/<br>Patritumab+ cetuximab<br>+ cisplatin or<br>carboplatin/<br>xx/M | Screening | Yes | yyyy-mm-dd (xx) | MUGA | xx.x |
| | CxDx | No | yyyy-mm-dd (xx) | | |
| xxxxxx/<br>Patritumab+ cetuximab<br>+ cisplatin or<br>carboplatin/ | Screening | Yes | yyyy-mm-dd (xx) | | xx.x |
| xx/F | CxDx | Yes | yyyy mm-dd (xx) | | XX.X |

Source: adam.adeg

Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.8.4.1: Human Anti-Humanized Antibody (HAHA) Safety Analysis Set

**HRG High** 

| Subject ID/<br>Group/Age/Gender | Visit | Time Point | Date/Time of<br>Sample Collection (Day) | Assay Type | Screening<br>Results | Confirmatoy<br>Results | Titer<br>Results | Final<br>Results |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | C1D1 | xx | yyyy-mm-dd: hh:mm (xx) | xxxx | Negative | | | |
| | CxDx<br>CxDx | xx | yyyy-mm-dd: hh:mm (xx) | xxxx | Nega ive | | | |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | C1D1 | | yyyy-mm-dd: hh:mm (xx) | xxxx | Negative | <b>Y</b> | | |
| | CxDx | | yyyy-mm-dd: hh:mm (xx) | xxxx | Positive | | | |
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/<br>xx/F | C1D1 | | yyyy-mm-dd: hh:mm (xx) | xxxx | Negative | | | |
| | CxDx | | yyyy-mm-dd: hh:mm (xx) | xxxx | Negative | | | |
| | CxDx | | yyyy-mm-dd: hh:mm (xx) | xxxx | Negative | | | |

Note: CxDx = Cycle x Day x

Source: adam.adbi

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

# Listing 16.2.8.4.2: Tumor Tissue Sample Collection and Biomarker Results Safety Analysis Set

HRG High

| Subject ID/<br>Group/Age/Gender | Date of Collection (Day) | Sample ID | Sample Type | Biomarker Test<br>(Standard Unit) | Result |
|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or carboplatin/xx/F | yyyy-mm-dd (xxx) | xxxxxx | Fresh Tissue | Test #1 (xxx) | xxxx |
| xxxxxx/<br>Patritumab+ cetuximab + cisplatin<br>or carboplatin/xx/M | yyyy-mm-dd (xxx) | xxxxxx | Archived | Test #1 xxx) | xxxx |
| xxxxxx/<br>Patritumab+ cetuximab + cisplatin<br>or carboplatin/xx/F | yyyy-mm-dd (xxx) | XXXXXX | Archived | Tes #1 xxx) | |

Source: adam.adbi

Programming Note: continue for HRG Low and Overall on the next page


Protocol U31287-A-U203

Page x of y <run date time>

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

#### Listing 16.2.9.1.1: FACT-H&N Item Scores FACT-H&N Analysis Set

HRG High

| Subject ID/Group/<br>Age/Gender | Visit | Date of<br>Assessment<br>(Study Day) | Scale | Item | Raw Score | Imputed Score [a] |
|---|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab + | C1D1 | YYYY-MM-DD<br>(xxx) | HNS | H&N <sub>i</sub> | x | |
| cisplatin or carboplatin/xx/F | | | | (i=112) | x | Х |
| | | | EWB | GE1 | x | |
| | | | | GE2 | X | X |
| | | | FWB | GF1 | X | X |
| | | | | GF2 | X | |
| | | | PWB | GP1 | X | X |
| | | | | GP2 | X | |
| | | | SWB | GS1 | X | X |
| | | | | GS2 | X | X |
| | C1D1 | YYYY-MM-DD<br>(xxx) | HNS | H&N <sub>i</sub> | X | |
| | | , , | | H&N2 | X | |
| | | | EWB | GE1 | X | |
| | | | | GE2 | X | |
| | | | FWB | GF1 | X | x |
| | | | | GF2 | х | X |

Notes: EWB=Emotional Well-Being; FWB=Functional Well-Being; PWB=Physical Well-Being; SWB=Social/Family Well-Being; HNS = Head and Neck Additional Concerns Subscale.

[a] If fewer than 50% of the raw score are missing on the subscale the raw score is imputed using the mean of the non-missing items. Source: adam.adqs

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.9.1.2: FACT-H&N Total and Subscale Scores FACT-H&N Analysis Set

HRG High

| Subject<br>ID/Group/Age/Gender | Visit | Date of<br>Assessment<br>(Study Day) | PWB<br>(# Missing) | SWB<br>(# Missing) | EWB<br>(# Missing) | FWB<br>(# Missing) | HNS Score<br>(# Missing) | FHNSI Score<br>(# Missing) | FACT-H&N |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx/ Patritumab+ cetuximab + cisplatin or | C1D1 | YYYY-MM-DD<br>(xxx) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| carboplatin/xx/F | CxD1 | YYYY-MM-DD<br>(xxx) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| xxxxxx/<br>Patritumab + cetuximab +<br>cisplatin or carboplatin<br>/xx/M | C1D1 | YYYY-MM-DD<br>(xxx) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| /AA/WI | C2D1 | YYYY-MM-DD<br>(xxx) | xx (x) | x (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| xxxxxx/<br>Patritumab + cetuximab +<br>cisplatin or | C1D1 | YYYY-MM-DD<br>(xxx) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| carboplatin/xx/F | C2D1 | YYYY-MM-D<br>(xxx) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx (x) | xx |
| | CxD1 | | 7 7 | | | | | | |

Notes: EWB=Emotional Well-Being; FWB=Functional Well-Being; PWB=Physical Well-Being; SWB=Social Well-Being; HNS = Head and Neck Additional Concerns Subscale; FHNSI = Head & Neck Symptom Index; FACT-H&N total score = PWB + SWB + EWB + FWB + HNS

Source: adam.adqs

Protocol U31287-A-U203

<Run Type> (Data Cut Date: DDMMMYYYY; Data Extraction Date: DDMMMYYY)

Listing 16.2.9.2: EQ-5D Scale Scores EQ-5D Analysis Set

**HRG High** 

| Subject ID/Group/<br>Age/Gender | Visit | Date of<br>Assessment<br>(Study Day) | Item | Response | Change from Baseline |
|---|---|---|---|---|---|
| xxxxxx/<br>Patritumab+ cetuximab +<br>cisplatin or carboplatin/xx/F | C1D1 | YYYY-MM-DD<br>(xxx) | Self-care Susual Activities A.Pain/Discomfort Anxiety/Depression VAS Score Index Score | Not a problem A modera e problem | x<br>x<br>x |
| | C1D1 | YYYY-MM-DD<br>(xxx) | OPIC | | |

Notes: EQ-5D descriptive system is coded 1 - 5, with higher core indicating more severe result.

The VAS score is numbered from 0 to 100, which 100 means the best health you can imagine, 0 means the worst health you can imagine.

Based on the patient's response to each of the 5 dimensions, a 1-digit number expressing the level selected for that dimension will be recorded and combined in a 5-digit number describing the respondent's health state. Each of the 5-digit combinations will be converted to a country-specific index value defining the health state of the patient.

Source: adam.adqs